CLINICAL TRIAL: NCT02732145
Title: Diagnostic Accuracy of "Three Rings Vulvoscopy" for Detection of Vulvar Dermatosis
Acronym: DATRIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ginekološka Poliklinika Dr. Vesna Harni (Other)
Collaborators: Klinički Bolnički Centar Zagreb (Other); University of Zagreb (Other)
Responsible Party: Principal Investigator, Vesna Harni, Dr. med. Vesna Harni, Ginekološka Poliklinika Dr. Vesna Harni
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PH20111201001
Record Dates: First submitted 2016-03-15; First posted 2016-04-08 (Estimated); Results first posted 2019-10-30 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Lichen Sclerosus; Lichen Planus; Lichen Simplex Chronicus; Vulvodynia
Keywords: Three-Vulvar-Rings; Three-Rings-Vulvoscopy; N-S-P scheme; Vulvoscopy Index; Vulvar Dermatosis; Vulvar Lichen Sclerosus; Lichen Planus; Lichen Simplex Chronicus; Vulvodynia; Provoked Vestibulodynia; Vulvar Vestibulitis; Vulvar Diseases
MeSH Terms: conditions — Lichen Sclerosus et Atrophicus; Lichen Planus; Neurodermatitis; Vulvodynia; Vulvar Lichen Sclerosus; Vulvar Vestibulitis; Vulvar Diseases

STUDY DESIGN:
Intervention Model Description: We performed the same interventions: Three Rings Vulvoscopy, Vulvar Biopsy and Histopathologically Evaluation in four groups of patients with and without vulvar discomfort, with the aim to detect vulvar dermatosis.
Oversight: Data Monitoring Committee: No

ARMS (4):
- Normal vulva (Placebo Comparator): The "Normal vulva" group consisted of patients without vulvar discomfort (ISSVD Questionnaire), and without any vulvar lesion (Clinical examination) undergoing planned labioplasty. For each patient with vulvar dermatosis, the first consecutive patient with normal vulva was taken for comparison.
  Interventions: Three Rings Vulvoscopy, Vulvar Biopsy, and Histopathology.
  Interventions: Diagnostic Test: "Three Rings Vulvoscopy" (TRIV); Procedure: Histopathology
- Impaired vulvar skin (Placebo Comparator): The group of "Impaired vulvar skin" was formed by the patients without vulvar symptoms (ISSVD Questionnaire), but with some non-specific vulvar lesions (Clinical examination) undergoing planned labioplasty, before surgery. For each patient with vulvar dermatosis, the first consecutive patient with impaired vulvar skin was taken for comparison.
  Interventions: Three Rings Vulvoscopy, Vulvar Biopsy, and Histopathology.
  Interventions: Diagnostic Test: "Three Rings Vulvoscopy" (TRIV); Procedure: Histopathology
- Vulvodynia (Placebo Comparator): The "Vulvodynia" group consisted of patients with vulvar discomfort (ISSVD Questionnaire), who fulfilled Friedrich's criteria (Clinical examination). Non-specific lesions found with TRIV were not relevant for the diagnosis of vulvodynia. For each patient with vulvar dermatosis, the first consecutive patient with vulvodynia was taken for comparison.
  Interventions: Three Rings Vulvoscopy, Vulvar Biopsy, and Histopathology.
  Interventions: Diagnostic Test: "Three Rings Vulvoscopy" (TRIV); Procedure: Histopathology
- Vulvar dermatosis (Active Comparator): The group of "Vulvar Dermatosis" was formed by the patients with vulvar discomfort (ISSVD Questionnaire) and vulvar lesion specific for dermatosis (Clinical examination).
  Interventions: Three Rings Vulvoscopy, Vulvar Biopsy, and Histopathology.
  Interventions: Diagnostic Test: "Three Rings Vulvoscopy" (TRIV); Procedure: Histopathology

INTERVENTIONS:
Diagnostic Test: "Three Rings Vulvoscopy" (TRIV) — Mapping of the vulvar lesions according to the three vulvar rings and specificity of the lesions during "Three Rings Vulvoscopy" technique (TRIV Form Data). Assessing of the data by the "Vulvoscopy Index" and the "N-S-P Scheme".
  Other Names: Colposcopy of the Vulva
Procedure: Histopathology — Biopsy of the vulva in symptomatic patients, vulvar samples after labiaplasty in asymptomatic patients.
  Other Names: Biopsy of the Vulva

SUMMARY:
The objective of the study was to determine sensitivity, specificity and diagnostic accuracy of "Three Rings Vulvoscopy" for detection of vulvar dermatosis using histopathology as the reference standard.

DETAILED DESCRIPTION:
"Three Rings Vulvoscopy" (TRIV) is a new, and original technique for performing colposcopy of the vulva, taking into account three different skin types and zones as well as morphological evaluation of vulvar lesions according to their specificity (non-specific and lesions specific for dermatosis). To evaluate the clinical value of TRIV, we designed two index tests, a quantitative test called "Vulvoscopy Index" and a semi-quantitative test marked as "N-S-P scheme." The sensitivity, specificity and diagnostic accuracy of both index tests were estimated in comparison with histopathology as the reference test in two groups of 164 consecutive patients with vulvar discomfort (82 patients with vulvar dermatosis and 82 patients with vulvodynia ) and 164 consecutive patients without vulvar discomfort (82 patients with "normal vulva" and 82 patients with "impaired vulvar skin").

The study was performed stratified, on three levels, whereby the first two levels were pre-assignments.

The first level of the study was an evaluation of vulvar discomfort during the routine gynecological care in the clinic "Poliklinika Harni" Zagreb, Croatia, where we searched for symptomatic patients; and in the esthetic gynecological unit of the same clinic, where we searched for asymptomatic patients. Vulvar discomfort was evaluated anamnestically by the "International Society for the Study of Vulvovaginal Disease (ISSVD) Vulvodynia Pattern Questionnaire." On the second level, we performed detailed clinical examination (inspection and Cotton-Swab test), searching for non-specific and lesions specific for skin (vulvar) dermatosis, and patients with vulvodynia who fulfilled Friedrich's criteria. Patients with vulvar infection or pre/malignancy were excluded from the study. Vulvar lesions in patients with vulvodynia were not relevant to the diagnosis of vulvodynia.

Among women without vulvar discomfort, we described those without any clinical findings ("normal vulva") and those with some non-specific findings on the vulva. We called this group "impaired vulvar skin." The results of the clinical examination were collected using "TRIV Form Data." On this way, we identified four groups of patients during the recruitment: vulvar dermatosis, vulvodynia, impaired vulvar skin, and normal vulva. For each patient with vulvar dermatosis (82 patients), the first consecutive patient with vulvodynia (82), impaired vulvar skin (82) and normal vulva (82) were taken for comparison.

The third level of the study presents the investigation and included diagnostic interventions "Three Rings Vulvoscopy" and vulvar biopsy with histopathology. The results of vulvoscopy were collected using "TRIV Form Data" and then assessed by "Vulvoscopy Index" and the "N-S-P Scheme." Biopsy of the vulva from the symptomatic patients was taken to confirm/exclude vulvar dermatosis. Asymptomatic patients, who were recruited from patients undergoing planned labiaplasty, granted vulvar samples to further investigation.

The statistical tests were made on a personal computer (PC) in the Statistical Package 12.0. All qualitative variables are shown in the tables with the absolute number and percentage. Quantitative variables are presented with arithmetic mean and standard deviation (if normal distribution), and by the median and range (if not a normal distribution).

A chi-squared test was used to test the difference between qualitative variables among the two groups. A chi-squared test with Yates correction was used for 2x2 size tables, and Fisher's exact test was used for small values. T-test proportions were used for the evaluation of the differences between the two percentages. Variance analysis (ANOVA) and post hoc Tukey HSD were used to test quantitative variables with normal distribution between multiple groups. Differences between the arithmetic mean of the two groups were tested by t-test.

Variables that did not have normal distribution were tested by nonparametric tests. The differences between several groups were tested by Kruskal-Wallis ANOVA and the differences between the two groups Mann-Whitney U test.

ELIGIBILITY:
Inclusion Criteria:

"Three Rings Vulvoscopy" performed at Poliklinika Harni, during the period from December 2011 - December 2016.

Ability to provide Informed Consent and complete Questionnaire.

Exclusion Criteria:

Incomplete medical records. Lack of histopathology. Vulvo-vaginal infection. Benign tumors of the vulva. Pre-/malignant conditions of the vulva.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 328 (Actual)
Dates: Start 2011-12; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vesna Harni, MD, Principal Investigator — Poliklinika Harni, Bukovacka 1, HR-10000 Zagreb, Croatia
Locations (1):
- Poliklinika Harni, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moyal-Barracco M, Wendling J. Vulvar dermatosis. Best Pract Res Clin Obstet Gynaecol. 2014 Oct;28(7):946-58. doi: 10.1016/j.bpobgyn.2014.07.005. Epub 2014 Jul 18. PMID 25132276
- [Background] Doyen J, Demoulin S, Delbecque K, Goffin F, Kridelka F, Delvenne P. Vulvar skin disorders throughout lifetime: about some representative dermatoses. Biomed Res Int. 2014;2014:595286. doi: 10.1155/2014/595286. Epub 2014 Jan 8. PMID 24511539
- [Background] Ball SB, Wojnarowska F. Vulvar dermatoses: lichen sclerosus, lichen planus, and vulval dermatitis/lichen simplex chronicus. Semin Cutan Med Surg. 1998 Sep;17(3):182-8. doi: 10.1016/s1085-5629(98)80012-6. PMID 9759675
- [Background] McKay M. Vulvar dermatoses: common problems in dermatological and gynaecological practice. Br J Clin Pract Suppl. 1990 Sep;71:5-10. PMID 2091734
- [Background] O'Keefe RJ, Scurry JP, Dennerstein G, Sfameni S, Brenan J. Audit of 114 non-neoplastic vulvar biopsies. Br J Obstet Gynaecol. 1995 Oct;102(10):780-6. doi: 10.1111/j.1471-0528.1995.tb10842.x. PMID 7547733
- [Background] Cooper SM, Ali I, Baldo M, Wojnarowska F. The association of lichen sclerosus and erosive lichen planus of the vulva with autoimmune disease: a case-control study. Arch Dermatol. 2008 Nov;144(11):1432-5. doi: 10.1001/archderm.144.11.1432. PMID 19015417
- [Background] Raspollini MR, Asirelli G, Moncini D, Taddei GL. A comparative analysis of lichen sclerosus of the vulva and lichen sclerosus that evolves to vulvar squamous cell carcinoma. Am J Obstet Gynecol. 2007 Dec;197(6):592.e1-5. doi: 10.1016/j.ajog.2007.04.003. Epub 2007 Aug 21. PMID 17714682
- [Background] Shier M, El-Khatib S. Vulvar lichen sclerosus. J Obstet Gynaecol Can. 2010 Oct;32(10):929-30. doi: 10.1016/s1701-2163(16)34676-x. No abstract available. English, French. PMID 21176300
- [Background] Petersen CD, Kristensen E, Lundvall L, Giraldi A. A retrospective study of relevant diagnostic procedures in vulvodynia. J Reprod Med. 2009 May;54(5):281-7. PMID 19517691
- Available data/document: Chapter/Commentary: ISBN:978-1-63484-507-6 — https://novapublishers.com/shop/cryosurgery-and-colposcopy-practices-outcomes-and-potential-complications/ — Harni V, Babic D, Barisic D. "Three Rings Vulvoscopy" - A New Approach to the Vulva. In: Cryosurgery and Colposcopy: Practices, Outcomes and Potential Complications, Editor: Lillian Watson. Publisher: Nova Science Publishers Inc, NewYork, USA, 2016.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at "Poliklinika Harni," Zagreb, Croatia, during routine gynecological care, and from esthetic unit to obtain vulvar specimens from patients with the normal vulva.
  For each patient with vulvar dermatosis, the first consecutive patient with vulvodynia, impaired vulvar skin, and normal vulva was taken for comparison.
Pre-assignment Details: Vulvar discomfort was evaluated with the ISSVD Vulvodynia Pattern Questionnaire (1. level of the investigation/pre-assignment), and vulvar lesions were assessed by clinical examination and Cotton-Swab test (2. level of the study/pre-assignment).
  Patients with vulvar infection and pre/malignancy were excluded from further investigation.
Groups:
- Normal Vulva: Patients without vulvar discomfort (ISSVD Vulvodynia Pattern Questionnaire) and finding any vulvar lesion (Clinical Examination and Cotton-Swab Test); undergoing planned labioplasty, who granted vulvar specimens for further investigation.
- Impaired Vulvar Skin: Patients without vulvar symptoms (ISSVD Vulvodynia Pattern Questionnaire), but with some non-specific vulvar lesions (Clinical Examination and Cotton-Swab Test); undergoing planned labioplasty, who granted vulvar specimens for further investigation.
- Vulvodynia: Patients with vulvar discomfort (ISSVD Vulvodynia Pattern Questionnaire), who clinically fulfilled Friedrich's criteria (Clinical Examination and Cotton-Swab Test). Non-specific lesions found with TRIV were not relevant for the diagnosis of vulvodynia.
- Vulvar Dermatosis: Patients with vulvar discomfort (ISSVD Vulvodynia Pattern Questionnaire) and vulvar lesions specific for dermatosis (Clinical Examination and Cotton-Swab Test).
Period: Overall Study
Arm/Group | Normal Vulva | Impaired Vulvar Skin | Vulvodynia | Vulvar Dermatosis
Started | 82 | 82 | 82 | 82
Completed | 82 | 82 | 82 | 82
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Vulva | Impaired Vulvar Skin | Vulvodynia | Vulvar Dermatosis | Total
Number analyzed (Participants) | 82 | 82 | 82 | 82 | 328
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 2 | 0 | 1 | 4
  Between 18 and 65 years | 81 | 79 | 82 | 66 | 308
  >=65 years | 0 | 1 | 0 | 15 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.21 (10.01) | 34.44 (9.37) | 35.71 (7.97) | 51.11 (16.21) | 38.87 (10.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 82 | 82 | 82 | 328
  Male | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 82 | 82 | 82 | 82 | 328
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Croatia | 82 | 82 | 82 | 82 | 328

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Accuracy of "Three Rings Vulvoscopy" by the "Vulvoscopy Index" for Detection of Vulvar Dermatosis
Description: The table shows the distribution of patients with and without vulvar dermatosis diagnosed by "Three Rings Vulvoscopy" (TRIV) using the "Vulvoscopy Index" and histopathology as a reference test.
  The Vulvoscopy Index as an outcome measure of TRIV is designed as a quantitative test based on five characteristics: vulvar complaints, Marinoff index, Cotton-Swab test, vulvar lesions according to the three vulvar rings and specificity of lesions; with following results: "Normal Vulva" (0-2 points), "Impaired Vulvar Skin" (3-11 points), "Vulvodynia" (12-18 points), and "Vulvar Dermatosis" (19-32 points).
  Since histopathology distinguishes only patients with and without vulvar dermatosis, the clinical value the Vulvoscopy Index had been estimated according to these two groups of patients. Patients with vulvoscopy diagnoses: "Normal Vulva," "Impaired Vulvar Skin" and "Vulvodynia" were classified into the group "Absent Vulvar Dermatosis."
Time Frame: ISSVD Questionnaire and TRIV, up to 75 minutes for each participant.
Population: Vulvar dermatosis was diagnosed in 82 patients by vulvoscopy and 72 patients by histopathology. Absent vulvar dermatosis was found in 246 patients by vulvoscopy and 256 patients by histopathology. The likelihood of vulvar dermatosis was higher as the value of the Vulvoscopy index was higher.
Measure: Count of Participants; unit: Participants
Groups:
- Vulvoscopy: Vulvar Dermatosis: Patients with vulvoscopy diagnosis "Vulvar Dermatosis" according to the "Vulvoscopy Index" (19-32 points).
- Vulvoscopy: Absent Vulvar Dermatosis: Patients with vulvoscopy diagnoses "Normal Vulva" (0-2 points), "Impaired Vulvar Skin" (3-11 points) and "Vulvodynia" (12-18 points) according to the "Vulvoscopy Index", who were classified into one group labeled by the term" Absent Vulvar Dermatosis".
Arm/Group | Vulvoscopy: Vulvar Dermatosis | Vulvoscopy: Absent Vulvar Dermatosis
Number analyzed (Participants) | 82 | 246
Participants
  Histopathology: Vulvar Dermatosis | 72 | 0
  Histopathology: Absent Vulvar Dermatosis | 10 | 246
Statistical Analysis 1: Comparison: Vulvoscopy: Vulvar Dermatosis vs Vulvoscopy: Absent Vulvar Dermatosis; Parameter: Sensitivity of "Three Rings Vulvoscopy" for detection of vulvar dermatosis; Test type: Other — Question: Determination of sensitivity of the "Vulvoscopy Index" as a measure of the sensitivity of "Three Rings Vulvoscopy" in comparison to the histopathological diagnosis of vulvar dermatosis; Sensitivity (2x2 Table) = 1.0000, 95% CI 2-sided [1.0000 to 1.0000] — The Sensitivity of the "Vulvoscopy Index" for Detection of Vulvar Dermatosis was 1.000 (Range: 1.0000 - 1.0000)
Statistical Analysis 2: Comparison: Vulvoscopy: Vulvar Dermatosis vs Vulvoscopy: Absent Vulvar Dermatosis; Parameter: Specificity of "Three Rings Vulvoscopy" for detection of vulvar dermatosis; Test type: Other — Question: Determination of specificity of the "Vulvoscopy index" as a measure of the specificity of "Three Rings Vulvoscopy" in comparison to the histopathological diagnosis of vulvar dermatosis; Specificity (2x2 Table) = 0.9609, 95% CI 2-sided [0.5794 to 1.0000] — The Specificity of the "Vulvoscopy Index" for Detection of Vulvar Dermatosis was 0.9609 (Range: 0.5794 - 1.0000)
Statistical Analysis 3: Comparison: Vulvoscopy: Vulvar Dermatosis vs Vulvoscopy: Absent Vulvar Dermatosis; Parameter: Diagnostic accuracy of "Three Rings Vulvoscopy" for detection of vulvar dermatosis; Test type: Other — Question: Determination of diagnostic accuracy of the "Vulvoscopy index" as a measure of the diagnostic value of "Three Rings Vulvoscopy" in comparison to the histopathological diagnosis of vulvar dermatosis; Diagnostic Accuracy (2x2 Table) = 0.9695, 95% CI 2-sided [0.6313 to 1.0000] — The Diagnostic accuracy of the "Vulvoscopy Index" for Detection of Vulvar Dermatosis was 0.9695 (Range: 0.6313 - 1.0000)
Statistical Analysis 4: Comparison: Vulvoscopy: Vulvar Dermatosis vs Vulvoscopy: Absent Vulvar Dermatosis; Parameter: Positive predictive value of "Three Rings Vulvoscopy" for detection of vulvar dermatosis; Test type: Superiority — Question: Determination of positive predictive value of the "Vulvoscopy index" for detection of vulvar dermatosis in comparison to the histopathology results; PPV (2x2 Table) = 0.8780, 95% CI 2-sided [0.2270 to 1.0000] — Positive predictive value of the "Vulvoscopy Index" for Detection of Vulvar Dermatosis was 0.8780 (Range: 0.2270 - 1.0000)
Statistical Analysis 5: Comparison: Vulvoscopy: Vulvar Dermatosis vs Vulvoscopy: Absent Vulvar Dermatosis; Parameter: Negative predictive value of "Three Rings Vulvoscopy" for detection of vulvar dermatosis; Test type: Other — Question: Determination of negative predictive value of the "Vulvoscopy index" for detection of vulvar dermatosis in comparison to the histopathology results; NPV (2x2 Table) = 1.0000, 95% CI 2-sided [1.0000 to 1.0000] — Negative predictive value of the "Vulvoscopy Index" for Detection of Vulvar Dermatosis was 1.0000 (Range: 1.0000 - 1.0000)
Statistical Analysis 6: Comparison: Vulvoscopy: Vulvar Dermatosis vs Vulvoscopy: Absent Vulvar Dermatosis; Parameter: The difference in the diagnostic accuracy between TRIV using the "Vulvoscopy Index" and histopathology for detection of vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the diagnostic accuracy of the "Vulvoscopy Index" as an outcome measure of the diagnostic value of "Three Rings Vulvoscopy," and histopathology?; p = 0.6108, t-test proportion

2. Primary Outcome: Distribution of Patients With Vulvar Dermatosis Diagnosed by Vulvoscopy (TRIV) and Histopathology According to Single Categories of the "Vulvoscopy Index"
Description: The table shows the distribution of patients with "Vulvar Dermatosis" diagnosed by "Three Rings Vulvoscopy" and histopathology according to single categories of the "Vulvoscopy Index."
  We described five categories within the Vulvoscopy Index:
  1. Vulvar complaints (present vs. absent),
  2. Marinoff index (positive vs. negative),
  3. Cotton-Swab test (positive vs. negative),
  4. Vulvar lesions according to the vulvar rings (Outer, Middle, and Inner Vulvar Ring Lesion) and
  5. Specificity of lesions (Non-specific and Specific Lesions).
Time Frame: ISSVD Questionnaire and TRIV, up to 75 minutes for each participant.
Population: Vulvar dermatosis was diagnosed in 82 patients by vulvoscopy and 72 patients by histopathology. The likelihood of vulvar dermatosis was higher as the value of the Vulvoscopy index was higher.
Measure: Count of Participants; unit: Participants
Groups:
- Histopathology: Vulvar Dermatosis: Histopathological diagnosis "Vulvar Dermatosis" from the vulvar specimens of 328 women was set in 72 patients.
Arm/Group | Vulvoscopy: Vulvar Dermatosis | Histopathology: Vulvar Dermatosis
Number analyzed (Participants) | 82 | 72
Participants
  Vulvar Complaints | 82 | 72
  Positive Marinoff Index | 35 | 31
  Positive Cotton-Swab | 28 | 24
  Lesions In Any Vulvar Ring | 82 | 72
  Outer Vulvar Ring Lesions | 77 | 68
  Middle Vulvar Ring Lesions | 82 | 72
  Inner Vulvar Ring Lesions | 74 | 68
  Non-Specific Lesions | 71 | 63
  Specific Lesions | 82 | 72
Statistical Analysis 1: Comparison: Vulvoscopy: Vulvar Dermatosis vs Histopathology: Vulvar Dermatosis; Parameter: The difference in the frequency of vulvar complaints in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Superiority — Question: Is there a difference in the frequency of vulvar complaints among the patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 1.0000, t-test proportion
Statistical Analysis 2: Comparison: Vulvoscopy: Vulvar Dermatosis vs Histopathology: Vulvar Dermatosis; Parameter: The difference in the frequency of positive Marinoff Index in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Superiority — Question: Is there a difference in the frequency of positive Marinoff Index among the patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.9628, t-test proportion
Statistical Analysis 3: Comparison: Vulvoscopy: Vulvar Dermatosis vs Histopathology: Vulvar Dermatosis; Parameter: The difference in the frequency of the positive Cotton-Swab test in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Superiority — Question: Is there a difference in the frequency of the positive Cotton-Swab test among the patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.9152, t-test proportion
Statistical Analysis 4: Comparison: Vulvoscopy: Vulvar Dermatosis vs Histopathology: Vulvar Dermatosis; Parameter: The difference in the frequency of any lesion in any vulvar ring in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Superiority — Question: Is there a difference in the frequency of any lesion in any vulvar ring in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 1.0000, t-test proportion
Statistical Analysis 5: Comparison: Vulvoscopy: Vulvar Dermatosis vs Histopathology: Vulvar Dermatosis; Parameter: The difference in the frequency of any vulvar lesion of the Outer Vulvar Ring in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Superiority — Question: Is there a difference in the frequency of any vulvar lesion of the Outer Vulvar Ring among the patients with vulvar dermatosis diagnosed with vulvoscopy and histopathology?; p = 0.8862, t-test proportion
Statistical Analysis 6: Comparison: Vulvoscopy: Vulvar Dermatosis vs Histopathology: Vulvar Dermatosis; Parameter: The difference in the frequency of any vulvar lesion of the Middle Vulvar Ring in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Superiority — Question: Is there a difference in the frequency of any vulvar lesion of the Middle Vulvar Ring among the patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 1.0000, t-test proportion
Statistical Analysis 7: Comparison: Vulvoscopy: Vulvar Dermatosis vs Histopathology: Vulvar Dermatosis; Parameter: The difference in the frequency of any vulvar lesion of the Inner Vulvar Ring in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Superiority — Question: Is there a difference in the frequency of any vulvar lesion of the Inner Vulvar Ring among the patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.3319, t-test proportion
Statistical Analysis 8: Comparison: Vulvoscopy: Vulvar Dermatosis vs Histopathology: Vulvar Dermatosis; Parameter: The difference in the frequency of non-specific vulvar lesions in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Superiority — Question: Is there a difference in the frequency of non-specific vulvar lesions among the patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.8662, t-test proportion
Statistical Analysis 9: Comparison: Vulvoscopy: Vulvar Dermatosis vs Histopathology: Vulvar Dermatosis; Parameter: The difference in the frequency of vulvar lesions specific for dermatosis in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Superiority — Question: Is there a difference in the frequency of specific vulvar lesions among the patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 1.0000, t-test proportion

3. Primary Outcome: Distribution of Patients With "Absent Vulvar Dermatosis" Diagnosed by Vulvoscopy (TRIV) and Histopathology According to Single Categories of the "Vulvoscopy Index"
Description: The table shows the distribution of patients with "Absent Vulvar Dermatosis" diagnosed by "Three Rings Vulvoscopy" (patients with vulvoscopical diagnoses "Normal Vulva," Impaired Vulvar Skin "and" Vulvodynia") and histopathology, according to single categories of the "Vulvoscopy Index."
  The five categories within the Vulvoscopy Index are:
  1. Vulvar complaints (present vs. absent),
  2. Marinoff index (positive vs. negative),
  3. Cotton-Swab test (positive vs. negative),
  4. Vulvar lesions according to the vulvar rings (Outer, Middle, and Inner Vulvar Ring Lesion) and
  5. Specificity of lesions (Non-specific and Specific Lesions).
Time Frame: ISSVD Questionnaire and TRIV, up to 75 minutes for each participant.
Population: "Absent Vulvar Dermatosis" was diagnosed in 246 patients by vulvoscopy and 256 patients by histopathology. The likelihood of absent vulvar dermatosis was higher as the value of the Vulvoscopy index was lower.
Measure: Count of Participants; unit: Participants
Groups:
- Histopathology: Absent Vulvar Dermatosis: Histopathological diagnosis "Normal Vulva" or absent vulvar dermatosis.
Arm/Group | Vulvoscopy: Absent Vulvar Dermatosis | Histopathology: Absent Vulvar Dermatosis
Number analyzed (Participants) | 246 | 256
Participants
  Vulvar Complaints | 82 | 92
  Positive Marinoff Index | 74 | 78
  Positive Cotton-Swab | 104 | 108
  Any Vulvar Ring Lesions | 163 | 173
  Outer Vulvar Ring Lesions | 18 | 27
  Middle Vulvar Ring Lesions | 115 | 125
  Inner Vulvar Ring Lesions | 156 | 162
  Non-Specific Lesions | 163 | 171
  Specific Lesions | 0 | 10
Statistical Analysis 1: Comparison: Vulvoscopy: Absent Vulvar Dermatosis vs Histopathology: Absent Vulvar Dermatosis; Parameter: The difference in the frequency of vulvar complaints in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Superiority — Question: Is there a difference in the frequency of vulvar complaints among the patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.5399, t-test proportion
Statistical Analysis 2: Comparison: Vulvoscopy: Absent Vulvar Dermatosis vs Histopathology: Absent Vulvar Dermatosis; Parameter: The difference in the frequency of positive Marinoff Index in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Superiority — Question: Is there a difference in the frequency of positive Marinoff Index among the patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.9248, t-test proportion
Statistical Analysis 3: Comparison: Vulvoscopy: Absent Vulvar Dermatosis vs Histopathology: Absent Vulvar Dermatosis; Parameter: The difference in the frequency of the positive Cotton-Swab test in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Superiority — Question: Is there a difference in the frequency of the positive Cotton-Swab test among the patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.9839, t-test proportion
Statistical Analysis 4: Comparison: Vulvoscopy: Absent Vulvar Dermatosis vs Histopathology: Absent Vulvar Dermatosis; Parameter: The difference in the frequency of any lesion in any vulvar ring in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Superiority — Question: Is there a difference in the frequency of any lesion in any vulvar ring among the patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.7537, t
Statistical Analysis 5: Comparison: Vulvoscopy: Absent Vulvar Dermatosis vs Histopathology: Absent Vulvar Dermatosis; Parameter: The difference in the frequency of any vulvar lesion of the Outer Vulvar Ring in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Superiority — Question: Is there a difference in the frequency of any vulvar lesion of the Outer Vulvar Ring among the patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.2054, t-test proportion
Statistical Analysis 6: Comparison: Vulvoscopy: Absent Vulvar Dermatosis vs Histopathology: Absent Vulvar Dermatosis; Parameter: The difference in the frequency of any vulvar lesion of the Middle Vulvar Ring in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Superiority — Question: Is there a difference in the frequency of any vulvar lesion of the Middle Vulvar Ring among the patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.6409, t-test proportion
Statistical Analysis 7: Comparison: Vulvoscopy: Absent Vulvar Dermatosis vs Histopathology: Absent Vulvar Dermatosis; Parameter: The difference in the frequency of any vulvar lesion of the Inner Vulvar Ring in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Superiority — Question: Is there a difference in the frequency of any vulvar lesion of the Inner Vulvar Ring among the patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.9753, t-test proportion
Statistical Analysis 8: Comparison: Vulvoscopy: Absent Vulvar Dermatosis vs Histopathology: Absent Vulvar Dermatosis; Parameter: The difference in the frequency of non-specific vulvar lesions in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Superiority — Question: Is there a difference in the frequency of non-specific vulvar lesions among the patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.8986, t-test proportion
Statistical Analysis 9: Comparison: Vulvoscopy: Absent Vulvar Dermatosis vs Histopathology: Absent Vulvar Dermatosis; Parameter: The difference in the frequency of vulvar lesions specific for dermatosis in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology (first biopsy); Test type: Superiority — Question: Is there a difference in the frequency of specific vulvar lesions among the patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology (first biopsy)?; p = 0.0017, t-test proportion

4. Primary Outcome: "Vulvoscopy Index" (Mean ± SD) in Patients With "Vulvar Dermatosis" Diagnosed by Vulvoscopy (TRIV) and Histopathology
Description: The table shows the results of "Three Rings Vulvoscopy" (TRIV) by single categories of the "Vulvoscopy Index" (mean ± SD) in patients with "Vulvar Dermatosis" diagnosed by TRIV and histopathology.
  The Vulvoscopy Index is based on five characteristics:
  1. Vulvar complaints (negative=0; positive=4 points),
  2. Marinoff index (negative=0; positive=3 points),
  3. Cotton-Swab test (negative=0; positive=2 points),
  4. Vulvar lesions according to the vulvar rings (Outer Vulvar Ring Lesions=4 points; Middle Vulvar Ring Lesions=2 points and Inner Vulvar Ring Lesions=1 point) and
  5. Specificity of lesions (Non-Specific Lesions=2 points; Specific Lesions=14 points).
  According to the Vulvoscopy Index, we have set the diagnoses: "Normal Vulva" (0-2 points), "Impaired Vulvar Skin" (3-11 points), "Vulvodynia" (12-18 points), and "Vulvar Dermatosis" (19-32 points).
  The likelihood of the diagnosis of "Vulvar Dermatosis" was higher as the value of the Vulvoscopy index was higher.
Time Frame: ISSVD Questionnaire and TRIV, up to 75 minutes for each participant.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vulvoscopy: Vulvar Dermatosis | Histopathology: Vulvar Dermatosis
Number analyzed (Participants) | 82 | 72
units on a scale
  Vulvar Complaints (0-4 Points) | 4.0 (0.0) | 4.0 (0.0)
  Marinoff Index (0-3 Points) | 1.28 (1.49) | 1.29 (1.50)
  Cotton-Swab (0-2 Points) | 0.68 (0.95) | 0.67 (0.95)
  Any Vulvar Ring Lesions (0-7 Points) | 6.66 (1.08) | 6.72 (1.00)
  Outer Vulvar Ring Lesions (0-4 Points) | 3.76 (0.96) | 3.78 (0.92)
  Middle Vulvar Ring Lesions (0-2 Points) | 2.0 (0.0) | 2.0 (0.0)
  Inner Vulvar Ring Lesions (0-1 Point) | 0.90 (0.30) | 0.94 (0.23)
  Specificity of Lesions (0-16) | 15.73 (0.69) | 15.75 (0.67)
  Non-Specific Lesions (0-2 Points) | 1.73 (0.69) | 1.75 (0.67)
  Specific Lesions (0-14 Points) | 14.0 (0.0) | 14.0 (0.0)
  Sum (0-32 Points) | 28.35 (2.46) | 28.43 (2.47)
Statistical Analysis 1: Comparison: Vulvoscopy: Vulvar Dermatosis vs Histopathology: Vulvar Dermatosis; Parameter: The difference in the score for vulvar complaints (mean) in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Equivalence — Question: Is there a difference in the score for vulvar complaints (mean) among the patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 1.0000, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Vulvoscopy: Vulvar Dermatosis vs Histopathology: Vulvar Dermatosis; Parameter: The difference in the score for Marinoff Index (mean) in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Equivalence — Question: Is there a difference in the score for Marinoff Index (mean) among patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.9899, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Vulvoscopy: Vulvar Dermatosis vs Histopathology: Vulvar Dermatosis; Parameter: The difference in the score for the Cotton-Swab test (mean) in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Equivalence — Question: Is there a difference in the score for the Cotton-Swab test (mean) among the patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.9686, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Vulvoscopy: Vulvar Dermatosis vs Histopathology: Vulvar Dermatosis; Parameter: The difference in the score for any lesion in any vulvar ring (mean) in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Equivalence — Question: Is there a difference in the score for any lesion in any vulvar ring (mean) among the patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.7055, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Vulvoscopy: Vulvar Dermatosis vs Histopathology: Vulvar Dermatosis; Parameter: The difference in the score for any vulvar lesion of the Outer Vulvar Ring (mean) in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Equivalence — Question: Is there a difference in the score for any vulvar lesion of the Outer Vulvar Ring (mean) among the patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.8852, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Vulvoscopy: Vulvar Dermatosis vs Histopathology: Vulvar Dermatosis; Parameter: The difference in the score for any vulvar lesion of the Middle Vulvar Ring (mean) in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Equivalence — Question: Is there a difference in the score for any vulvar lesion of the Middle Vulvar Ring (mean) among the patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 1.0000, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Vulvoscopy: Vulvar Dermatosis vs Histopathology: Vulvar Dermatosis; Parameter: The difference in the score for any vulvar lesion of the Inner Vulvar Ring (mean) in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Equivalence — Question: Is there a difference in the score for any vulvar lesion of the Inner Vulvar Ring (mean) among the patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.3351, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Vulvoscopy: Vulvar Dermatosis vs Histopathology: Vulvar Dermatosis; Parameter: The difference in the score for the specificity of vulvar lesions (mean) in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Equivalence — Question: Is there a difference in the score for the specificity of vulvar lesions (mean) among the patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.8673, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: Vulvoscopy: Vulvar Dermatosis vs Histopathology: Vulvar Dermatosis; Parameter: The difference in the score for non-specific vulvar lesions (mean) in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Equivalence — Question: Is there a difference in the score for non-specific vulvar lesions (mean) among the patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.8673, Wilcoxon (Mann-Whitney)
Statistical Analysis 10: Comparison: Vulvoscopy: Vulvar Dermatosis vs Histopathology: Vulvar Dermatosis; Parameter: The difference in the score for specific vulvar lesions (mean) with vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Equivalence — Question: Is there a difference in the score for specific vulvar lesions (mean) among the patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 1.0000, Wilcoxon (Mann-Whitney)
Statistical Analysis 11: Comparison: Vulvoscopy: Vulvar Dermatosis vs Histopathology: Vulvar Dermatosis; Parameter: The difference in the overall sum of points for the "Vulvoscopy Index" (mean) in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Equivalence — Question: Is there a difference in the overall sum of points for the "Vulvoscopy Index" (mean) among the patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.8472, Wilcoxon (Mann-Whitney)

5. Primary Outcome: "Vulvoscopy Index" (Mean ± SD) in Patients With "Absent Vulvar Dermatosis" Diagnosed by Vulvoscopy (TRIV) and Histopathology
Description: The table shows the results of "Three Rings Vulvoscopy" (TRIV) by single categories of the "Vulvoscopy Index" (mean± SD) in patients with "Absent Vulvar Dermatosis" diagnosed by TRIV and histopathology.
  According to the Vulvoscopy Index, we have set the diagnoses: "Normal Vulva" (0-2 points), "Impaired Vulvar Skin" (3-11 points), "Vulvodynia" (12-18 points), and "Vulvar Dermatosis" (19-32 points).
  Since histopathology can distinguish only patients with and without vulvar dermatosis, the distribution was estimated according to these two groups of patients. Hence, patients with vulvoscopical diagnoses "Normal Vulva," Impaired Vulvar Skin "and" Vulvodynia" were classified into the one group called "Absent Vulvar Dermatosis." The likelihood of the diagnosis of "Absent Vulvar Dermatosis" was higher as the value of the Vulvoscopy index was lower.
Time Frame: ISSVD Questionnaire and TRIV, up to 75 minutes for each participant.
Population: "Absent Vulvar Dermatosis" was diagnosed in 246 patients by vulvoscopy and 256 patients by histopathology.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Histopathology: Absent Vulvar Dermatosis: Histopathological diagnosis: "Normal Vulva" or absent vulvar dermatosis.
Arm/Group | Vulvoscopy: Absent Vulvar Dermatosis | Histopathology: Absent Vulvar Dermatosis
Number analyzed (Participants) | 246 | 256
units on a scale
  Vulvar Complaints (0-4 Points) | 1.33 (1.89) | 1.44 (1.92)
  Marinoff Index (0-3 Points) | 0.90 (1.38) | 0.91 (1.38)
  Cotton-Swab (0-2 Points) | 0.85 (0.99) | 0.84 (0.99)
  Any Vulvar Ring Lesions (0-7 Points) | 1.86 (1.92) | 2.03 (2.09)
  Outer Vulvar Ring Lesions (0-4 Points) | 0.29 (1.04) | 0.49 (1.23)
  Middle Vulvar Ring Lesions (0-2 Points) | 0.93 (1.00) | 0.98 (1.00)
  Inner Vulvar Ring Lesions (0-1 Point) | 0.63 (0.48) | 0.63 (0.48)
  Specificity of Lesions (0-16 Points) | 1.33 (0.95) | 1.88 (2.93)
  Non-Specific Lesions (0-2 Points) | 1.33 (0.95) | 1.34 (094)
  Specific Lesions (0-14 Points) | 0.0 (0.0) | 0.55 (2.72)
  Sum (0-32 Points) | 6.27 (5.89) | 7.11 (7.15)

6. Primary Outcome: "Vulvoscopy Index" (Median | Range) in Patients With "Vulvar Dermatosis" Diagnosed by Vulvoscopy (TRIV) and Histopathology
Description: The table shows the results of "Three Rings Vulvoscopy" (TRIV) by single categories of the "Vulvoscopy Index" (median ± SD) in patients with "Vulvar Dermatosis" diagnosed by TRIV and histopathology.
  The Vulvoscopy Index is based on five characteristics:
  1. Vulvar complaints (negative=0; positive=4 points),
  2. Marinoff index (negative=0; positive=3 points),
  3. Cotton-Swab test (negative=0; positive=2 points),
  4. Vulvar lesions according to the vulvar rings (Outer Vulvar Ring Lesions=4 points; Middle Vulvar Ring Lesions=2 points and Inner Vulvar Ring Lesions=1 point) and
  5. Specificity of lesions (Non-specific Lesions=2 points; Specific Lesions=14 points).
  According to the Vulvoscopy Index, we have set the diagnoses: "Normal Vulva" (0-2 points), "Impaired Vulvar Skin" (3-11 points), "Vulvodynia" (12-18 points), and "Vulvar Dermatosis" (19-32 points).
  The likelihood of the diagnosis of "Vulvar Dermatosis" was higher as the value of the Vulvoscopy index was higher.
Time Frame: ISSVD Questionnaire and TRIV, up to 75 minutes for each participant.
Population: Vulvar dermatosis was diagnosed in 82 patients by vulvoscopy and 72 patients by histopathology.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Vulvoscopy: Vulvar Dermatosis | Histopathology: Vulvar Dermatosis
Number analyzed (Participants) | 82 | 72
units on a scale
  Vulvar Complaints (0-4 Points) | 4 [4 to 4] | 4 [4 to 4]
  Marinoff Index (0-3 Points) | 0 [0 to 3] | 0 [0 to 3]
  Cotton-Swab (0-2 Points) | 0 [0 to 2] | 0 [0 to 2]
  Any Vulvar Ring Lesions (0-7 Points) | 7 [2 to 7] | 7 [2 to 7]
  Outer Vulvar Ring Lesions (0-4 Points) | 4 [0 to 4] | 4 [0 to 4]
  Middle Vulvar Ring Lesions (0-2 Points) | 2 [2 to 2] | 2 [2 to 2]
  Inner Vulvar Ring Lesions (0-1 Point) | 1 [0 to 1] | 1 [0 to 1]
  Specificity of Lesions, in total (0-16 Points) | 16 [14 to 16] | 16 [14 to 16]
  Non-Specific Lesions (0-2 Points) | 2 [0 to 2] | 2 [0 to 2]
  Specific Lesions (0-14 Points) | 14 [14 to 14] | 14 [14 to 14]
  Sum (0-32 Points) | 28.5 [21 to 32] | 28.5 [21 to 32]
Statistical Analysis 1: Comparison: Vulvoscopy: Vulvar Dermatosis vs Histopathology: Vulvar Dermatosis; Parameter: The difference in the score for vulvar complaints (median) in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Equivalence — Question: Is there a difference in the score for vulvar complaints (median) among the patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 1.0000, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Vulvoscopy: Vulvar Dermatosis vs Histopathology: Vulvar Dermatosis; Parameter: The difference in the score for Marinoff Index (median) in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Equivalence — Question: Is there a difference in the score for Marinoff Index (median) among the patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.9629, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Vulvoscopy: Vulvar Dermatosis vs Histopathology: Vulvar Dermatosis; Parameter: The difference in the score for the Cotton-Swab test (median) in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Equivalence — Question: Is there a difference in the score for the Cotton-Swab test (median) among the patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.9155, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Vulvoscopy: Vulvar Dermatosis vs Histopathology: Vulvar Dermatosis; Parameter: The difference in the score for any lesion in any vulvar ring (median) in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Equivalence — Question: Is there a difference in the score for any lesion in any vulvar ring (median) among the patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.4913, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Vulvoscopy: Vulvar Dermatosis vs Histopathology: Vulvar Dermatosis; Parameter: The difference in the score for any vulvar lesion of the Outer Vulvar Ring (median) in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Equivalence — Question: Is there a difference in the score for any vulvar lesion of the Outer Vulvar Ring (median) among the patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.8866, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Vulvoscopy: Vulvar Dermatosis vs Histopathology: Vulvar Dermatosis; Parameter: The difference in the score for any vulvar lesion of the Middle Vulvar Ring (median) in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Equivalence — Question: Is there a difference in the score for any vulvar lesion of the Middle Vulvar Ring (median) among the patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 1.0000, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Vulvoscopy: Vulvar Dermatosis vs Histopathology: Vulvar Dermatosis; Parameter: The difference in the score for any vulvar lesion of the Inner Vulvar Ring (median) in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Equivalence — Question: Is there a difference in the score for any vulvar lesion of the Inner Vulvar Ring (median) among the patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.3335, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Vulvoscopy: Vulvar Dermatosis vs Histopathology: Vulvar Dermatosis; Parameter: The difference in the score for the specificity of vulvar lesions (median) in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Equivalence — Question: Is there a difference in the score for the specificity of vulvar lesions (median) among the patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.8666, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: Vulvoscopy: Vulvar Dermatosis vs Histopathology: Vulvar Dermatosis; Parameter: The difference in the score for non-specific vulvar lesions (median) in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Equivalence — Question: Is there a difference in the score for non-specific vulvar lesions (median) among the patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.8666, Wilcoxon (Mann-Whitney)
Statistical Analysis 10: Comparison: Vulvoscopy: Vulvar Dermatosis vs Histopathology: Vulvar Dermatosis; Parameter: The difference in the score for specific vulvar lesions (median) with vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Equivalence — Question: Is there a difference in the score for specific vulvar lesions (median) among the patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 1.0000, Wilcoxon (Mann-Whitney)
Statistical Analysis 11: Comparison: Vulvoscopy: Vulvar Dermatosis vs Histopathology: Vulvar Dermatosis; Parameter: The difference in the overall sum of points for the "Vulvoscopy Index" (median) in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Equivalence — Question: Is there a difference in the overall sum of points for the "Vulvoscopy Index" (median) among the patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.8144, Wilcoxon (Mann-Whitney)

7. Primary Outcome: "Vulvoscopy Index" (Median | Range) in Patients With "Absent Vulvar Dermatosis" Diagnosed by Vulvoscopy (TRIV) and Histopathology
Description: The table shows the results of "Three Rings Vulvoscopy" (TRIV) by single categories of the "Vulvoscopy Index" (median ± SD) in patients with "Absent Vulvar Dermatosis" diagnosed by TRIV (patients with vulvoscopical diagnoses "Normal Vulva," Impaired Vulvar Skin "and" Vulvodynia") and histopathology.
  According to the Vulvoscopy Index, we have set the diagnoses: "Normal Vulva" (0-2 points), "Impaired Vulvar Skin" (3-11 points), "Vulvodynia" (12-18 points), and "Vulvar Dermatosis" (19-32 points).
  The likelihood of the diagnosis of "Absent Vulvar Dermatosis" was higher as the value of the Vulvoscopy index was lower.
Time Frame: ISSVD Questionnaire and TRIV, up to 75 minutes for each participant.
Population: "Absent Vulvar Dermatosis" was diagnosed in 246 patients by vulvoscopy and 256 patients by histopathology.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Vulvoscopy: Absent Vulvar Dermatosis | Histopathology: Absent Vulvar Dermatosis
Number analyzed (Participants) | 246 | 256
units on a scale
  Vulvar Complaints (0-4 Points) | 0 [0 to 4] | 0 [0 to 4]
  Marinoff Index (0-3 Points) | 0 [0 to 3] | 0 [0 to 3]
  Cotton-Swab (0-2 Points) | 0 [0 to 2] | 0 [0 to 2]
  Any Vulvar Ring Lesions (0-7 Points) | 1 [0 to 7] | 1 [0 to 7]
  Outer Vulvar Ring Lesions (0-4 Points) | 0 [0 to 4] | 0 [0 to 4]
  Middle Vulvar Ring Lesions (0-2 Points) | 0 [0 to 2] | 0 [0 to 2]
  Inner Vulvar Ring Lesions (0-1 Point) | 1 [0 to 1] | 1 [0 to 1]
  Specificity of Lesions, in total (0-16 Points) | 2 [0 to 2] | 2 [0 to 16]
  Non-Specific Lesions (0-2 Points) | 2 [0 to 2] | 2 [0 to 2]
  Specific Lesions (0-14 Points) | 0 [0 to 0] | 0 [0 to 14]
  Sum (0-32 Points) | 5 [0 to 18] | 5 [0 to 32]
Statistical Analysis 1: Comparison: Vulvoscopy: Absent Vulvar Dermatosis vs Histopathology: Absent Vulvar Dermatosis; Parameter: The difference in the score for vulvar complaints (median) in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Equivalence — Question: Is there a difference in the score for vulvar complaints in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.5403, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Vulvoscopy: Absent Vulvar Dermatosis vs Histopathology: Absent Vulvar Dermatosis; Parameter: The difference in the score for Marinoff Index (median) in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Equivalence — Question: Is there a difference in the score for Marinoff Index in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.9248, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Vulvoscopy: Absent Vulvar Dermatosis vs Histopathology: Absent Vulvar Dermatosis; Parameter: The difference in the score for the Cotton-Swab test (median) in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Equivalence — Question: Is there a difference in the score for the Cotton-Swab test in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.9839, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Vulvoscopy: Absent Vulvar Dermatosis vs Histopathology: Absent Vulvar Dermatosis; Parameter: The difference in the score for any lesion in any vulvar ring (median) in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Equivalence — Question: Is there a difference in the score for any lesion in any vulvar ring (median) in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.5124, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Vulvoscopy: Absent Vulvar Dermatosis vs Histopathology: Absent Vulvar Dermatosis; Parameter: The difference in the score for any vulvar lesion of the Outer Vulvar Ring (median) in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Equivalence — Question: Is there a difference in the score for any vulvar lesion of the Outer Vulvar Ring in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.2058, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Vulvoscopy: Absent Vulvar Dermatosis vs Histopathology: Absent Vulvar Dermatosis; Parameter: The difference in the score for any vulvar lesion of the Middle Vulvar Ring (median) in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Equivalence — Question: Is there a difference in the score for any vulvar lesion of the Middle Vulvar Ring in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.6412, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Vulvoscopy: Absent Vulvar Dermatosis vs Histopathology: Absent Vulvar Dermatosis; Parameter: The difference in the score for any vulvar lesion of the Inner Vulvar Ring (median) in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Equivalence — Question: Is there a difference in the score for any vulvar lesion of the Inner Vulvar Ring in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.9753, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Vulvoscopy: Absent Vulvar Dermatosis vs Histopathology: Absent Vulvar Dermatosis; Parameter: The difference in the score for the specificity of vulvar lesions (median) in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Equivalence — Question: Is there a difference in the score for the specificity of vulvar lesions in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.3621, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: Vulvoscopy: Absent Vulvar Dermatosis vs Histopathology: Absent Vulvar Dermatosis; Parameter: The difference in the score for non-specific vulvar lesions (median) in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Equivalence — Question: Is there a difference in the score for non-specific vulvar lesions in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.8987, Wilcoxon (Mann-Whitney)
Statistical Analysis 10: Comparison: Vulvoscopy: Absent Vulvar Dermatosis vs Histopathology: Absent Vulvar Dermatosis; Parameter: The difference in the score for vulvar lesions specific for dermatosis (median) in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology (first biopsy); Test type: Equivalence — Question: Is there a difference in the score for specific vulvar lesions in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology (first biopsy)?; p = 0.0018, Wilcoxon (Mann-Whitney)
Statistical Analysis 11: Comparison: Vulvoscopy: Absent Vulvar Dermatosis vs Histopathology: Absent Vulvar Dermatosis; Parameter: The difference in the overall sum of points for the "Vulvoscopy Index" (median) in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Equivalence — Question: Is there a difference in the overall sum of points for the "Vulvoscopy Index" in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.4409, Wilcoxon (Mann-Whitney)

8. Primary Outcome: Diagnostic Accuracy of "Three Rings Vulvoscopy" by the "N-S-P Scheme" for Detection of Vulvar Dermatosis
Description: The distribution of patients with and without vulvar dermatosis diagnosed by vulvoscopy ("N-S-P Scheme") and histopathology.
  According to the specificity of lesions, vulvoscopy results were classified as normal "N" (absence of any lesion), suspect "S" (non-specific lesions) and pathologic "P" results (lesion specific to dermatosis); and each of the three vulvar rings is represented by a single result.
  The final vulvoscopy result is presented in the form of a three-letter formula, where the first letter indicates the vulvoscopy result in the Outer Vulvar Ring, the mean initial indicates the vulvoscopy result of the Middle Vulvar Ring and the last letter denotes the vulvoscopy result of the Inner Vulvar Ring.
  "N-S-P Scheme" divides the results of the vulvoscopy into three groups: "Normal Vulvoscopy," "Suspect Vulvoscopy" and "Pathological Vulvoscopy." Diagnosis of vulvar dermatosis was established if one or more vulvar rings showed pathological results ("Pathological Vulvoscopy").
Time Frame: ISSVD Questionnaire and TRIV, up to 75 minutes for each participant.
Population: Histopathology distinguishes two groups of patients with and without vulvar dermatosis. Therefore the accuracy of the "N-S-P Scheme" had been estimated according to these two groups of patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Vulvoscopy: Vulvar Dermatosis | Vulvoscopy: Absent Vulvar Dermatosis
Number analyzed (Participants) | 82 | 246
Participants
  Histopathology: Vulvar Dermatosis | 72 | 0
  Histopathology: Absent Vulvar Dermatosis | 10 | 246
Statistical Analysis 1: Comparison: Vulvoscopy: Vulvar Dermatosis vs Vulvoscopy: Absent Vulvar Dermatosis; Parameter: Sensitivity of "Three Rings Vulvoscopy" for detection of vulvar dermatosis; Test type: Other — Question: Determination of sensitivity of the "N-S-P Scheme" as a measure of the sensitivity of "Three Rings Vulvoscopy", in comparison to the histopathological diagnosis of vulvar dermatosis; Sensitivity (2x2 Table) = 1.0000, 95% CI 2-sided [1.0000 to 1.0000] — The Sensitivity of the "N-S-P Scheme" for Detection of Vulvar Dermatosis was 1.0000 (Range: 1.0000 - 1.0000)
Statistical Analysis 2: Comparison: Vulvoscopy: Vulvar Dermatosis vs Vulvoscopy: Absent Vulvar Dermatosis; Parameter: Specificity of "Three Rings Vulvoscopy" for detection of vulvar dermatosis; Test type: Other — Question: Determination of specificity of the "N-S-P Scheme" as a measure of the specificity of "Three Rings Vulvoscopy", in comparison to the histopathological diagnosis of vulvar dermatosis; Specificity (2x2 Table) = 0.9609, 95% CI 2-sided [0.5794 to 1.0000] — The Specificity of the "N-S-P Scheme" for Detection of Vulvar Dermatosis was 0.9609 (Range: 0.5794 - 1.0000)
Statistical Analysis 3: Comparison: Vulvoscopy: Vulvar Dermatosis vs Vulvoscopy: Absent Vulvar Dermatosis; Parameter: Diagnostic accuracy of "Three Rings Vulvoscopy" for detection of vulvar dermatosis; Test type: Other — Question: Determination of diagnostic accuracy of the "N-S-P Scheme" as a measure of the diagnostic value of the "Three Rings Vulvoscopy", in relation to the histopathological diagnosis of vulvar dermatosis; Diagnostic Accuracy (2x2 Table) = 0.9695, 95% CI 2-sided [0.6313 to 1.0000] — The Diagnostic accuracy of the "N-S-P Scheme" for Detection of Vulvar Dermatosis was 0.9695 (Range: 0.6313 - 1.0000)
Statistical Analysis 4: Comparison: Vulvoscopy: Vulvar Dermatosis vs Vulvoscopy: Absent Vulvar Dermatosis; Parameter: Positive predictive value of "Three Rings Vulvoscopy" for detection of vulvar dermatosis; Test type: Other — Question: Determination of positive predictive value of the "N-S-P Scheme" for detection of vulvar dermatosis in comparison to the histopathology results; PPV (2x2 Table) = 0.8780, 95% CI 2-sided [0.2270 to 1.0000] — Positive predictive value of the "N-S-P Scheme" for Detection of Vulvar Dermatosis was 0.8780 (Range: 0.2270 - 1.0000)
Statistical Analysis 5: Comparison: Vulvoscopy: Vulvar Dermatosis vs Vulvoscopy: Absent Vulvar Dermatosis; Parameter: Negative predictive value of "Three Rings Vulvoscopy" for detection of vulvar dermatosis; Test type: Other — Question: Determination of negative predictive value of the "N-S-P Scheme" for detection of vulvar dermatosis in comparison to the histopathology results; NPV (2x2 Table) = 1.0000, 95% CI 2-sided [1.0000 to 1.0000] — Negative predictive value of the "N-S-P Scheme" for Detection of Vulvar Dermatosis was 1.0000 (Range: 1.0000 - 1.0000)
Statistical Analysis 6: Comparison: Vulvoscopy: Vulvar Dermatosis vs Vulvoscopy: Absent Vulvar Dermatosis; Parameter: The difference in the diagnostic accuracy between TRIV using the "N-S-P Scheme" and histopathology for detection of vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the diagnostic accuracy of the "N-S-P Scheme" as an outcome measure of the diagnostic value of "Three Rings Vulvoscopy," and histopathology?; p = 0.6108, t-test proportion

9. Primary Outcome: Distribution of Vulvar Lesions According to the "N-S-P Scheme" in Patients With Vulvar Dermatosis Diagnosed by Vulvoscopy (TRIV) and Histopathology
Description: The table shows the distribution of vulvoscopy lesions in relation to the vulvar rings and their specificity according to the "N-S-P Scheme," in patients with vulvar dermatosis diagnosed by vulvoscopy (TRIV) and histopathology.
  Vulvoscopy findings of each of the three vulvar rings: Outer (first letter in the formula), Middle (second letter), and Inner Vulvar Ring (third letter) were evaluated as normal "N" (absence of any lesions), suspect "S" (non-specific lesions), or pathological "P" (lesions specific for dermatosis).
  "Normal vulvoscopy" indicated the absence of any lesion in all three vulvar rings ("N-N-N").
  "Suspect vulvoscopy" was used to mark findings of non-specific lesions ("S-#*-#"; "S-S-#"; "S-S-S"; "S-N-S" etc.).
  "Pathological vulvoscopy" spelled out the finding of lesions specific for dermatosis in any of the three vulvar rings ("P-#-#"; "P-P-"; "P-P-P"; "P-N-S" etc.).
  * is the label for any of the three possibilities: N or S or P.
Time Frame: ISSVD Questionnaire and TRIV, up to 75 minutes for each participant.
Population: Vulvar dermatosis was diagnosed in 82 patients by vulvoscopy and 72 patients by histopathology. The likelihood of vulvar dermatosis was higher as one or more of the vulvar rings were assessed as "P."
Measure: Count of Participants; unit: Participants
Arm/Group | Vulvoscopy: Vulvar Dermatosis | Histopathology: Vulvar Dermatosis
Number analyzed (Participants) | 82 | 72
Participants
  Outer Vulvar Ring: No Lesion | N-#-# | 6 | 5
  Outer Vulvar Ring: Non-Specific Lesions | S-#-# | 24 | 22
  Outer Vulvar Ring: Specific Lesions | P-#-# | 73 | 64
  Middle Vulvar Ring: No Lesion | #-N-# | 0 | 0
  Middle Vulvar Ring: Non-Specific Lesions | #-S-# | 41 | 35
  Middle Vulvar Ring: Specific Lesions | #-P-# | 73 | 65
  Inner Vulvar Ring: No Lesion | #-#-N | 9 | 5
  Inner Vulvar Ring: Non-Specific Lesions | #-#-S | 55 | 51
  Inner Vulvar Ring: Specific Lesions | #-#-P | 49 | 46
  All Three Vulvar Rings: No Lesion N-N-N | 0 | 0
  Any Vulvar Ring: Non-Specific Lesions | 67 | 60
  Any Vulvar Ring: Specific Lesions | 82 | 72
Statistical Analysis 1: Comparison: Vulvoscopy: Vulvar Dermatosis vs Histopathology: Vulvar Dermatosis; Parameter: The difference in the frequency of "N-#-#" result (no lesions) of the Outer Vulvar Ring in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Superiority — Question: Is there a difference in the frequency of "N-#-#" result (no lesions) of the Outer Vulvar Ring in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.9286, t-test proportion
Statistical Analysis 2: Comparison: Vulvoscopy: Vulvar Dermatosis vs Histopathology: Vulvar Dermatosis; Parameter: The difference in the frequency of "S-#-#" result (non-specific lesions) of the Outer Vulvar Ring in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Superiority — Question: Is there a difference in the frequency of "S-#-#" result (non-specific lesions) of the Outer Vulvar Ring in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.8618, t-test proportion
Statistical Analysis 3: Comparison: Vulvoscopy: Vulvar Dermatosis vs Histopathology: Vulvar Dermatosis; Parameter: The difference in the frequency of "P-#-#" result (specific lesions) of the Outer Vulvar Ring in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Superiority — Question: Is there a difference in the frequency of "P-#-#" result (specific lesions) of the Outer Vulvar Ring in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.9786, t-test proportion
Statistical Analysis 4: Comparison: Vulvoscopy: Vulvar Dermatosis vs Histopathology: Vulvar Dermatosis; Parameter: The difference in the frequency of "#-N-#" result (no lesions) of the Middle Vulvar Ring in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Superiority — Question: Is there a difference in the frequency of "#-N-#" result (no lesions) of the Middle Vulvar Ring in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 1.0000, t-test proportion
Statistical Analysis 5: Comparison: Vulvoscopy: Vulvar Dermatosis vs Histopathology: Vulvar Dermatosis; Parameter: The difference in the frequency of "#-S-#" result (non-specific lesions) of the Middle Vulvar Ring in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Superiority — Question: Is there a difference in the frequency of "#-S-#" result (non-specific lesions) of the Middle Vulvar Ring in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.8634, t-test proportion
Statistical Analysis 6: Comparison: Vulvoscopy: Vulvar Dermatosis vs Histopathology: Vulvar Dermatosis; Parameter: The difference in the frequency of "#-P-#" result (specific lesions) of the Middle Vulvar Ring in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Superiority — Question: Is there a difference in the frequency of "#-P-#" result (specific lesions) of the Middle Vulvar Ring in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.7992, t-test proportion
Statistical Analysis 7: Comparison: Vulvoscopy: Vulvar Dermatosis vs Histopathology: Vulvar Dermatosis; Parameter: The difference in the frequency of "#-#-N" result (no lesions) of the Inner Vulvar Ring in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Superiority — Question: Is there a difference in the frequency of "#-#-N" result (no lesions) of the Inner Vulvar Ring in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.3912, t-test proportion
Statistical Analysis 8: Comparison: Vulvoscopy: Vulvar Dermatosis vs Histopathology: Vulvar Dermatosis; Parameter: The difference in the frequency of "#-#-S" result (non-specific lesions) of the Inner Vulvar Ring in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Superiority — Question: Is there a difference in the frequency of "#-#-S" result (non-specific lesions) of the Inner Vulvar Ring in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.6152, t-test proportion
Statistical Analysis 9: Comparison: Vulvoscopy: Vulvar Dermatosis vs Histopathology: Vulvar Dermatosis; Parameter: The difference in the frequency of "#-#-P" result (specific lesions) of the Inner Vulvar Ring in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Superiority — Question: Is there a difference in the frequency of "#-#-P" result (specific lesions) of the Inner Vulvar Ring in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.6108, t-test proportion
Statistical Analysis 10: Comparison: Vulvoscopy: Vulvar Dermatosis vs Histopathology: Vulvar Dermatosis; Parameter: The difference in the frequency of "N-N-N" result (no lesions) in any of the Three Vulvar Rings in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Superiority — Question: Is there a difference in the frequency of "N-N-N" result (no lesions) in any of the Three Vulvar Rings in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 1.0000, t-test proportion
Statistical Analysis 11: Comparison: Vulvoscopy: Vulvar Dermatosis vs Histopathology: Vulvar Dermatosis; Parameter: The difference in the frequency of "S" result (non-specific lesions) in any of the Three Vulvar Rings ("S-#-#"; "S-S-#"; "S-S-S"; "S-N-S" etc.) in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Superiority — Question: Is there a difference in the frequency of "S" result (non-specific lesions) in any of the Three Vulvar Rings ("S-#-#"; "S-S-#"; "S-S-S"; "S-N-S" etc.) in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.7912, t-test proportion
Statistical Analysis 12: Comparison: Vulvoscopy: Vulvar Dermatosis vs Histopathology: Vulvar Dermatosis; Parameter: The difference in the frequency of "P" result (specific lesions) in any of the Three Vulvar Rings ("P-#-#"; "P-P-"; "P-P-P"; "P-N-S" etc.) in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Superiority — Question: Is there a difference in the frequency of "P" result (specific lesions) in any of the Three Vulvar Rings ("P-#-#"; "P-P-"; "P-P-P"; "P-N-S" etc.) in patients with vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 1.0000, t-test proportion

10. Primary Outcome: Distribution of Vulvar Lesions According to the "N-S-P Scheme" in Patients With Absent Vulvar Dermatosis Diagnosed by Vulvoscopy (TRIV) and Histopathology
Description: The table shows the distribution of lesions according to their specificity and vulvar rings in patients without vulvar dermatosis diagnosed by vulvoscopy (TRIV) and histopathology, as a reference test.
  According to the "N-S-P scheme," we have set the diagnoses: "Normal result" (no lesion), "Suspect result" (non-specific lesion in any of the vulvar rings), and "Pathological result" (specific for dermatosis in any of the vulvar rings).
  Since histopathology can distinguish only patients with and without dermatosis, the distribution was estimated according to these two groups of patients. Hence, patients with normal and suspect vulvoscopic results were classified into one group called "Absent Vulvar Dermatosis."
Time Frame: ISSVD Questionnaire and TRIV, up to 75 minutes for each participant.
Population: "Absent Vulvar Dermatosis" was diagnosed in 246 patients by vulvoscopy and 256 patients by histopathology. The likelihood of absent vulvar dermatosis was higher as none of the vulvar rings were assessed as "P."
Measure: Count of Participants; unit: Participants
Groups:
- Vulvoscopy: Absent Vulvar Dermatosis: Patients with vulvoscopy diagnoses: "Normal Vulva", "Impaired Vulvar Skin" and "Vulvodynia" according to the "N-S-P Scheme", who were classified into one group marked by the term" Absent Vulvar Dermatosis".
Arm/Group | Vulvoscopy: Absent Vulvar Dermatosis | Histopathology: Absent Vulvar Dermatosis
Number analyzed (Participants) | 246 | 256
Participants
  Outer Vulvar Ring: No Lesion | N-#-# | 227 | 228
  Outer Vulvar Ring: Non-Specific Lesions | S-#-# | 18 | 20
  Outer Vulvar Ring: Specific Lesions | P-#-# | 0 | 9
  Middle Vulvar Ring: No Lesion | #-N-# | 131 | 131
  Middle Vulvar Ring: Non-Specific Lesions | #-S-# | 115 | 121
  Middle Vulvar Ring: Specific Lesions | #-P-# | 0 | 8
  Inner Vulvar Ring: No Lesion | #-#-N | 89 | 93
  Inner Vulvar Ring: Non-Specific Lesions | #-#-S | 157 | 161
  Inner Vulvar Ring: Specific Lesions | #-#-P | 0 | 3
  All Three Vulvar Rings: No Lesion N-N-N | 83 | 83
  Any Vulvar Ring: Non-Specific Lesions | 163 | 170
  Any Vulvar Ring: Specific Lesions | 0 | 10
Statistical Analysis 1: Comparison: Vulvoscopy: Absent Vulvar Dermatosis vs Histopathology: Absent Vulvar Dermatosis; Parameter: The difference in the frequency of "N-#-#" result (no lesions) of the Outer Vulvar Ring in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Superiority — Question: Is there a difference in the frequency of "N-#-#" result (no lesions) of the Outer Vulvar Ring in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.2530, t-test proportion
Statistical Analysis 2: Comparison: Vulvoscopy: Absent Vulvar Dermatosis vs Histopathology: Absent Vulvar Dermatosis; Parameter: The difference in the frequency of "S-#-#" result (non-specific lesions) of the Outer Vulvar Ring in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Superiority — Question: Is there a difference in the frequency of "S-#-#" result (non-specific lesions) of the Outer Vulvar Ring in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.8338, t-test proportion
Statistical Analysis 3: Comparison: Vulvoscopy: Absent Vulvar Dermatosis vs Histopathology: Absent Vulvar Dermatosis; Parameter: The difference in the frequency of "P-#-#" result (specific lesions) of the Outer Vulvar Ring in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Superiority — Question: Is there a difference in the frequency of "P-#-#" result (specific lesions) of the Outer Vulvar Ring in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.0019, t-test proportion
Statistical Analysis 4: Comparison: Vulvoscopy: Absent Vulvar Dermatosis vs Histopathology: Absent Vulvar Dermatosis; Parameter: The difference in the frequency of "#-N-#" result (no lesions) of the Middle Vulvar Ring in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Superiority — Question: Is there a difference in the frequency of "#-N-#" result (no lesions) of the Middle Vulvar Ring in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.6541, t-test proportion
Statistical Analysis 5: Comparison: Vulvoscopy: Absent Vulvar Dermatosis vs Histopathology: Absent Vulvar Dermatosis; Parameter: The difference in the frequency of "#-S-#" result (non-specific lesions) of the Middle Vulvar Ring in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Superiority — Question: Is there a difference in the frequency of "#-S-#" result (non-specific lesions) of the Middle Vulvar Ring in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.8224, t-test proportion
Statistical Analysis 6: Comparison: Vulvoscopy: Absent Vulvar Dermatosis vs Histopathology: Absent Vulvar Dermatosis; Parameter: The difference in the frequency of "#-P-#" result (specific lesions) of the Middle Vulvar Ring in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Superiority — Question: Is there a difference in the frequency of "#-P-#" result (specific lesions) of the Middle Vulvar Ring in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.0064, t-test proportion
Statistical Analysis 7: Comparison: Vulvoscopy: Absent Vulvar Dermatosis vs Histopathology: Absent Vulvar Dermatosis; Parameter: The difference in the frequency of "#-#-N" result (no lesions) of the Inner Vulvar Ring in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Superiority — Question: Is there a difference in the frequency of "#-#-N" result (no lesions) of the Inner Vulvar Ring in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.9723, t-test proportion
Statistical Analysis 8: Comparison: Vulvoscopy: Absent Vulvar Dermatosis vs Histopathology: Absent Vulvar Dermatosis; Parameter: The difference in the frequency of "#-#-S" result (non-specific lesions) of the Inner Vulvar Ring in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Superiority — Question: Is there a difference in the frequency of "#-#-S" result (non-specific lesions) of the Inner Vulvar Ring in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.8161, t-test proportion
Statistical Analysis 9: Comparison: Vulvoscopy: Absent Vulvar Dermatosis vs Histopathology: Absent Vulvar Dermatosis; Parameter: The difference in the frequency of "#-#-P" result (specific lesions) of the Inner Vulvar Ring in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Superiority — Question: Is there a difference in the frequency of "#-#-P" result (specific lesions) of the Inner Vulvar Ring in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.1165, t-test proportion
Statistical Analysis 10: Comparison: Vulvoscopy: Absent Vulvar Dermatosis vs Histopathology: Absent Vulvar Dermatosis; Parameter: The difference in the frequency of "N-N-N" result (no lesions) in any of the Three Vulvar Rings in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Superiority — Question: Is there a difference in the frequency of "N-N-N" result (no lesions) in any of the Three Vulvar Rings in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.6339, t-test proportion
Statistical Analysis 11: Comparison: Vulvoscopy: Absent Vulvar Dermatosis vs Histopathology: Absent Vulvar Dermatosis; Parameter: The difference in the frequency of "S" result (non-specific lesions) in any of the Three Vulvar Rings ("S-#-#"; "S-S-#"; "S-S-S"; "S-N-S" etc.) in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Superiority — Question: Is there a difference in the frequency of "S" result (non-specific lesions) in any of the Three Vulvar Rings ("S-#-#"; "S-S-#"; "S-S-S"; "S-N-S" etc.) in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.9724, t-test proportion
Statistical Analysis 12: Comparison: Vulvoscopy: Absent Vulvar Dermatosis vs Histopathology: Absent Vulvar Dermatosis; Parameter: The difference in the frequency of "P" result (specific lesions) in any of the Three Vulvar Rings ("P-#-#"; "P-P-"; "P-P-P"; "P-N-S" etc.) in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology; Test type: Superiority — Question: Is there a difference in the frequency of "P" result (specific lesions) in any of the Three Vulvar Rings ("P-#-#"; "P-P-"; "P-P-P"; "P-N-S" etc.) in patients with absent vulvar dermatosis diagnosed by vulvoscopy and histopathology?; p = 0.0016, t-test proportion

11. Secondary Outcome: Baseline Characteristics: Age
Description: The table shows the age in four groups of patients with and without vulvar discomfort.
Time Frame: ISSVD Questionnaire, up to 30 minutes for each participant.
Population: Baseline characteristics were assessed by anamnestic data (ISSVD Vulvodynia Pattern Questionnaire) and clinical examination.
Measure: Mean (Standard Deviation); unit: years
Groups:
- Normal Vulva: Patients without vulvar discomfort (ISSVD Vulvodynia Pattern Questionnaire) and without finding any clinical and colposcopy vulvar lesion.
- Impaired Vulvar Skin: Patients without vulvar symptoms (ISSVD Vulvodynia Pattern Questionnaire) but with some non-specific vulvar lesions found clinically and with TRIV.
- Vulvodynia: Patients with vulvar discomfort (ISSVD Vulvodynia Pattern Questionnaire), who clinically fulfilled Friedrich's criteria. Non-specific lesions found with TRIV were not relevant for diagnosis of vulvodynia.
- Vulvar Dermatosis: Patients with vulvar discomfort (ISSVD Vulvodynia Pattern Questionnaire), clinical and vulvoscopy (TRIV) finding of lesions specific for dermatosis.
Arm/Group | Normal Vulva | Impaired Vulvar Skin | Vulvodynia | Vulvar Dermatosis
Number analyzed (Participants) | 82 | 82 | 82 | 82
years | 34.2 (10.0) | 34.4 (9.4) | 34.2 (10.0) | 51.1 (16.2)
Statistical Analysis 1: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the age of patients from different groups; Test type: Equivalence — Question: Is there a difference in the age of patients from different groups?; p = 0.0000, ANOVA

12. Secondary Outcome: Baseline Characteristics: Weight
Description: The table shows the weight in four groups of patients with and without vulvar discomfort.
Time Frame: ISSVD Questionnaire, up to 30 minutes for each participant.
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Normal Vulva | Impaired Vulvar Skin | Vulvodynia | Vulvar Dermatosis
Number analyzed (Participants) | 82 | 82 | 82 | 82
kg | 61.9 (8.3) | 63.3 (10.9) | 61.1 (9.2) | 71.3 (12.0)
Statistical Analysis 1: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; The difference in the weight of patients from different groups; Test type: Equivalence — Is there a difference in the weight of patients from different groups?; p = 0.0000, ANOVA

13. Secondary Outcome: Baseline Characteristics: Height
Description: The table shows the height in four groups of patients with and without vulvar discomfort.
Time Frame: ISSVD Questionnaire, up to 30 minutes for each participant.
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Normal Vulva | Impaired Vulvar Skin | Vulvodynia | Vulvar Dermatosis
Number analyzed (Participants) | 82 | 82 | 82 | 82
cm | 169.1 (6.0) | 168.7 (6.3) | 166.7 (6.7) | 167.5 (5.7)
Statistical Analysis 1: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; The difference in the height of patients from different groups; Test type: Equivalence — Is there a difference in the height of patients from different groups; p = 0.0557, ANOVA

14. Secondary Outcome: Baseline Characteristics: BMI
Description: The table shows the body mass index (Mean ± SD) in four groups of patients with and without vulvar discomfort.
Time Frame: ISSVD Questionnaire, up to 30 minutes for each participant.
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Normal Vulva | Impaired Vulvar Skin | Vulvodynia | Vulvar Dermatosis
Number analyzed (Participants) | 82 | 82 | 82 | 82
kg/m^2 | 21.6 (2.5) | 22.3 (3.6) | 22.0 (2.9) | 25.4 (4.1)
Statistical Analysis 1: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; The difference in the body mass index of patients from different groups; Test type: Equivalence — Is there a difference in the body mass index of patients from different groups; p = 0.0000, ANOVA

15. Secondary Outcome: Demographic Data in Patients With and Without Vulvar Discomfort
Description: The table shows demographic data - age: more or less than 65 years, reproductive age, menopause, domicile country as a country of birth, the degree of education (more and less than 12 years), marital status, births, abortions, and using of contraception among four groups of patient.
Time Frame: ISSVD Questionnaire, up to 30 minutes for each participant.
Population: We assesses demographic data by ISSVD Vulvodynia Pattern Questionnaire (anamnestic).
Measure: Count of Participants; unit: Participants
Groups:
- Normal Vulva: Patients without vulvar discomfort (ISSVD Vulvodynia Pattern Questionnaire) and without finding of any clinical and colposcopy vulvar lesion.
Arm/Group | Normal Vulva | Impaired Vulvar Skin | Vulvodynia | Vulvar Dermatosis
Number analyzed (Participants) | 82 | 82 | 82 | 82
Participants
  Age: ≥ 65 years | 0 | 1 | 0 | 15
  Age: < 65 years | 82 | 81 | 82 | 67
  Reproductive Age | 77 | 79 | 76 | 36
  Menopausal age | 5 | 3 | 6 | 46
  Domicile country (Croatia) as a Country of Birth | 68 | 62 | 68 | 61
  Education: >12 Years | 52 | 58 | 52 | 42
  Education: ≤12 Years | 30 | 24 | 30 | 40
  Married | 44 | 39 | 44 | 69
  Nuliparious | 49 | 52 | 44 | 17
  Multiparous (3 and more births) | 6 | 4 | 6 | 12
  Abortion | 8 | 7 | 15 | 29
  Contraception | 21 | 16 | 20 | 10
Statistical Analysis 1: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of patients older than 65 years between different groups; Test type: Equivalence — Question: Is there a difference in the incidence of patients older than 65 years in different groups?; p = 0.0000, Chi-squared
Statistical Analysis 2: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of menopausal patients among different groups; Test type: Equivalence — Question: Is there a difference in the incidence of menopausal patients among different groups?; p = 0.0000, Chi-squared
Statistical Analysis 3: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of domicile country (Croatia) as a country of birth among patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of domicile country (Croatia) as a country of birth among patients from different groups; p = 0.3708, Chi-squared
Statistical Analysis 4: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of patients educated equally or less than 12 years among different groups; Test type: Equivalence — Question: Is there a difference in the incidence of patients educated equally or less than 12 years among different groups?; p = 0.0180, Chi-squared
Statistical Analysis 5: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of marital status among patients from different groups; Test type: Equivalence — Question: Is there a difference in marital status among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 6: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the nulliparity among patients from different groups; Test type: Equivalence — Question: Is there a difference in the nulliparity among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 7: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the multiparity among patients from different groups; Test type: Equivalence — Question: Is there a difference in the multiparity among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 8: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the number of abortions among patients from different groups; Test type: Equivalence — Question: Is there a difference in the number of abortions among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 9: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the using of contraception among patients from different groups; Test type: Equivalence — Question: Is there a difference in the using of contraception among patients from different groups?; p = 0.1323, Chi-squared

16. Secondary Outcome: Various Characteristics and Duration of Vulvar Discomfort in Patients With Vulvar Dermatosis and Vulvodynia
Description: The table shows various characteristics of vulvar pain (complaints) in patients with vulvar dermatosis or vulvodynia.
  Generally, we can differentiate between two categories of pain - the dull pain vs. the sharp pain depending on the nerve fibers in the skin, which are involved in the provocation of the pain.
  The symptoms of the dull pain are burning, stinging, soreness, irritation, itching, feeling of inflammation and aching.
  The symptoms of the sharp pain are a knife-like pain, paper-cuts pain, stabbing and sticking. We do not know, are there some symptoms characteristic for vulvar dermatosis or vulvodynia.
Time Frame: ISSVD Questionnaire, up to 30 minutes for each participant.
Population: Vulvar discomfort was evaluated anamnestically by the "ISSVD Vulvodynia Pattern Questionnaire".
Measure: Count of Participants; unit: Participants
Groups:
- Vulvodynia: Patients with vulvar discomfort (ISSVD Vulvodynia Pattern Questionnaire) who clinically fulfilled Friedrich's criteria. Non-specific lesions found with TRIV were not relevant for diagnosis of vulvodynia.
Arm/Group | Vulvar Dermatosis | Vulvodynia
Number analyzed (Participants) | 82 | 82
Participants
  Dull / Slow Pain | 82 | 81
  Burning | 22 | 37
  Stinging | 65 | 66
  Soreness | 37 | 54
  Irritation | 35 | 48
  Itching | 79 | 63
  Inflammation | 38 | 49
  Aching | 21 | 45
  Sharp / Fast Pain | 12 | 31
  Knife-Like Pain | 5 | 13
  Paper-Cuts Pain | 3 | 10
  Stabbing | 6 | 17
  Sticking | 9 | 18
  Association Of Symptoms | 24 | 64
  Duration Of Discomfort >24 month | 58 | 53
  Duration Of Discomfort >12 monts | 11 | 16
  Duration Of Discomfort >6 months | 9 | 8
Statistical Analysis 1: Comparison: Vulvar Dermatosis vs Vulvodynia; Parameter: The difference in the incidence of symptoms of the dull pain of the vulva (burning, stinging, soreness, irritation, itching, inflammation, aching) among patients with vulvar discomfort; Test type: Equivalence — Question: Is there a difference in the incidence of symptoms of the dull pain of the vulva among patients with vulvar discomfort?; p = 0.3158, Chi-squared
Statistical Analysis 2: Comparison: Vulvar Dermatosis vs Vulvodynia; Parameter: The difference in the incidence of symptoms of the sharp pain in the vulva (stabbing, sticking, knife-like pain, paper-cuts pain) among patients with vulvar discomfort; Test type: Equivalence — Question: Is there a difference in the incidence of symptoms of the sharp pain of the vulva among patients with vulvar discomfort?; p = 0.0007, Chi-squared
Statistical Analysis 3: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of symptoms of the dull pain versus the sharp pain of the vulva in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of the dull pain versus the sharp pain of the vulva in the patients with vulvar dermatosis?; p = 0.0000, Chi-squared
Statistical Analysis 4: Comparison: Vulvodynia; Parameter: The difference in the incidence of symptoms of the dull pain versus the sharp pain of the vulva in patients with vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of the dull pain versus the sharp pain of the vulva in the patients with vulvodynia?; p = 0.0000, Chi-squared
Statistical Analysis 5: Comparison: Vulvar Dermatosis vs Vulvodynia; Parameter: The difference in the incidence of vulvar burning among patients with vulvar discomfort; Test type: Equivalence — Question: Is there a difference in the incidence of vulvar burning among patients with vulvar discomfort?; p = 0.0147, Chi-squared
Statistical Analysis 6: Comparison: Vulvar Dermatosis vs Vulvodynia; Parameter: The difference in the incidence of vulvar stinging among patients with vulvar discomfort; Test type: Equivalence — Question: Is there a difference in the incidence of vulvar stinging among patients with vulvar discomfort?; p = 0.8456, Chi-squared
Statistical Analysis 7: Comparison: Vulvar Dermatosis vs Vulvodynia; Parameter: The difference in the incidence of vulvar soreness among patients with vulvar discomfort; Test type: Equivalence — Question: Is there a difference in the incidence of vulvar soreness among patients with vulvar discomfort?; p = 0.0076, Chi-squared
Statistical Analysis 8: Comparison: Vulvar Dermatosis vs Vulvodynia; Parameter: The difference in the incidence of irritation of the vulva among patients with vulvar discomfort; Test type: Equivalence — Question: Is there a difference in the incidence of irritation of the vulva among the patients with vulvar discomfort?; p = 0.0423, Chi-squared
Statistical Analysis 9: Comparison: Vulvar Dermatosis vs Vulvodynia; Parameter: The difference in the incidence of the knife-like pain in the vulva among patients with vulvar discomfort; Test type: Equivalence — Question: Is there a difference in the incidence of the knife-like pain in the vulva among the patients with vulvar discomfort?; p = 0.0457, Chi-squared
Statistical Analysis 10: Comparison: Vulvar Dermatosis vs Vulvodynia; Parameter: The difference in the incidence of the paper-cuts pain of the vulva among patients with vulvar discomfort; Test type: Equivalence — Question: Is there a difference in the incidence of the paper-cuts pain of the vulva among the patients with vulvar discomfort?; p = 0.0430, Chi-squared
Statistical Analysis 11: Comparison: Vulvar Dermatosis vs Vulvodynia; Parameter: The difference in the incidence of the stabbing of the vulva among patients with vulvar discomfort; Test type: Equivalence — Question: Is there a difference in the incidence of the stabbing of the vulva among the patients with vulvar discomfort?; p = 0.0134, Chi-squared
Statistical Analysis 12: Comparison: Vulvar Dermatosis vs Vulvodynia; Parameter: The difference in the incidence of sticking of the vulva among patients with vulvar discomfort; Test type: Equivalence — Question: Is there a difference in the incidence of sticking of the vulva among the patients with vulvar discomfort?; p = 0.0581, Chi-squared
Statistical Analysis 13: Comparison: Vulvar Dermatosis vs Vulvodynia; Parameter: The difference in the incidence of itching of the vulva among patients with vulvar discomfort; Test type: Equivalence — Question: Is there a difference in the incidence of itching of the vulva among the patients with vulvar discomfort?; p = 0.0002, Chi-squared
Statistical Analysis 14: Comparison: Vulvar Dermatosis vs Vulvodynia; Parameter: The difference in the incidence of the feeling of inflammation of the vulva among patients with vulvar discomfort; Test type: Equivalence — Question: Is there a difference in the incidence of the feeling of inflammation of the vulva among the patients with vulvar discomfort?; p = 0.0852, Chi-squared; t-test proportion = 0.0000
Statistical Analysis 15: Comparison: Vulvar Dermatosis vs Vulvodynia; Parameter: The difference in the incidence of aching of the vulva among patients with vulvar discomfort; Test type: Equivalence — Question: Is there a difference in the incidence of aching of the vulva among the patients with vulvar discomfort?; p = 0.0001, Chi-squared
Statistical Analysis 16: Comparison: Vulvar Dermatosis vs Vulvodynia; Parameter: The difference in the incidence of association of different vulvar symptoms among patients with vulvar discomfort; Test type: Equivalence — Question: Is there a difference in the association of different symptoms of the vulva among the patients with vulvar discomfort?; p = 0.0000, Chi-squared
Statistical Analysis 17: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of vulvar itching versus burning in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of vulvar itching versus burning in the patients with vulvar dermatosis?; p = 0.0000, t-test proportion
Statistical Analysis 18: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of vulvar itching versus stinging in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of vulvar itching versus stinging in the patients with vulvar dermatosis?; p = 0.0008, t-test proportion
Statistical Analysis 19: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of vulvar itching versus soreness in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of vulvar itching versus soreness in the patients with vulvar dermatosis?; p = 0.0000, t-test proportion
Statistical Analysis 20: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of vulvar itching versus irritation in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of vulvar itching versus irritation in the patients with vulvar dermatosis?; p = 0.0000, t-test proportion
Statistical Analysis 21: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of vulvar itching versus the feeling of inflammation in patients with vulvar dermatosis; Test type: Superiority; p = 0.0000, t-test proportion — There was a statistically significant difference at p<0.001. Patients with vulvar dermatosis had significantly more often itching than the feeling of inflammation of the vulva
Statistical Analysis 22: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of vulvar itching versus aching in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of vulvar itching versus aching in the patients with vulvar dermatosis?; p = 0.0000, t-test proportion
Statistical Analysis 23: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of vulvar stinging versus burning in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of vulvar stinging versus burning in the patients with vulvar dermatosis?; p = 0.0000, t-test proportion
Statistical Analysis 24: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of vulvar stinging versus soreness in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of vulvar stinging versus soreness in the patients with vulvar dermatosis?; p = 0.0000, t-test proportion
Statistical Analysis 25: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of vulvar stinging versus irritation in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of vulvar stinging versus irritation in the patients with vulvar dermatosis?; p = 0.0000, t-test proportion
Statistical Analysis 26: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of vulvar stinging versus the feeling of inflammation in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of vulvar stinging versus the feeling of inflammation in the patients with vulvar dermatosis?; p = 0.0000, t-test proportion
Statistical Analysis 27: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of vulvar stinging versus aching in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of vulvar stinging versus aching in the patients with vulvar dermatosis?; p = 0.0000, t-test proportion
Statistical Analysis 28: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of vulvar aching versus burning in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of vulvar aching versus burning in the patients with vulvar dermatosis?; p = 0.8591, t-test proportion
Statistical Analysis 29: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of vulvar aching versus soreness in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of vulvar aching versus soreness in the patients with vulvar dermatosis?; p = 0.0090, t-test proportion
Statistical Analysis 30: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of vulvar aching versus irritation in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of vulvar aching versus irritation in the patients with vulvar dermatosis?; p = 0.0212, t-test proportion
Statistical Analysis 31: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of vulvar aching versus the feeling of inflammation in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of vulvar aching versus the feeling of inflammation in the patients with vulvar dermatosis?; p = 0.0057, t-test proportion
Statistical Analysis 32: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of vulvar sticking versus knife-like pain in patients with vulvar dermatosis who had sharp vulvar pain; Test type: Superiority — Question: Is there a difference in the incidence of vulvar sticking versus knife-like pain in the patients with vulvar dermatosis who had sharp pain?; p = 0.0977, t-test proportion
Statistical Analysis 33: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of vulvar sticking versus paper-cuts pain in patients with vulvar dermatosis who had sharp vulvar pain; Test type: Superiority — Question: Is there a difference in the incidence of vulvar sticking versus paper-cuts pain in the patients with vulvar dermatosis who had sharp pain?; p = 0.0143, t-test proportion
Statistical Analysis 34: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of vulvar sticking versus stabbing in patients with vulvar dermatosis who had sharp vulvar pain; Test type: Superiority — Question: Is there a difference in the incidence of vulvar sticking versus stabbing in the patients with vulvar dermatosis who had sharp pain?; p = 0.2059, t-test proportion
Statistical Analysis 35: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of vulvar stabbing versus knife-like pain in patients with vulvar dermatosis who had sharp vulvar pain; Test type: Superiority — Question: Is there a difference in the incidence of vulvar stabbing versus knife-like pain in the patients with vulvar dermatosis who had sharp pain?; p = 0.6820, t-test proportion
Statistical Analysis 36: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of vulvar stabbing versus paper-cuts pain in patients with vulvar dermatosis who had sharp vulvar pain; Test type: Superiority — Question: Is there a difference in the incidence of vulvar stabbing versus paper-cuts pain in the patients with vulvar dermatosis who had sharp pain?; p = 0.2059, t-test proportion
Statistical Analysis 37: Comparison: Vulvodynia; Parameter: The difference in the incidence of vulvar stinging versus burning in patients with vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of vulvar stinging versus burning in the patients with vulvodynia?; p = 0.0000, t-test proportion
Statistical Analysis 38: Comparison: Vulvodynia; Parameter: The difference in the incidence of vulvar stinging versus soreness in patients with vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of vulvar stinging versus soreness in the patients with vulvodynia?; p = 0.0344, t-test proportion
Statistical Analysis 39: Comparison: Vulvodynia; Parameter: The difference in the incidence of vulvar stinging versus irritation in patients with vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of vulvar stinging versus irritation in the patients with vulvodynia?; p = 0.0023, t-test proportion
Statistical Analysis 40: Comparison: Vulvodynia; Parameter: The difference in the incidence of vulvar stinging versus itching in patients with vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of vulvar stinging versus itching in the patients with vulvodynia?; p = 0.5675, t-test proportion
Statistical Analysis 41: Comparison: Vulvodynia; Parameter: The difference in the incidence of vulvar stinging versus the feeling of inflammation in patients with vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of vulvar stinging versus the feeling of inflammation in the patients with vulvodynia?; p = 0.0037, t-test proportion
Statistical Analysis 42: Comparison: Vulvodynia; Parameter: The difference in the incidence of vulvar stinging versus aching in patients with vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of vulvar stinging versus aching in the patients with vulvodynia?; p = 0.0005, t-test proportion
Statistical Analysis 43: Comparison: Vulvodynia; Parameter: The difference in the incidence of vulvar itching versus burning in patients with vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of vulvar itching versus burning in the patients with vulvodynia?; p = 0.0000, t-test proportion
Statistical Analysis 44: Comparison: Vulvodynia; Parameter: The difference in the incidence of vulvar itching versus soreness in patients with vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of vulvar itching versus soreness in the patients with vulvodynia?; p = 0.1201, t-test proportion
Statistical Analysis 45: Comparison: Vulvodynia; Parameter: The difference in the incidence of vulvar itching versus irritation in patients with vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of vulvar itching versus irritation in the patients with vulvodynia?; p = 0.0123, t-test proportion
Statistical Analysis 46: Comparison: Vulvodynia; Parameter: The difference in the incidence of vulvar itching versus the feeling of inflammation in patients with vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of vulvar itching versus the feeling of inflammation in the patients with vulvodynia?; p = 0.0188, t-test proportion
Statistical Analysis 47: Comparison: Vulvodynia; Parameter: The difference in the incidence of vulvar itching versus aching in patients with vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of vulvar itching versus aching in the patients with vulvodynia?; p = 0.0030, t-test proportion
Statistical Analysis 48: Comparison: Vulvodynia; Parameter: The difference in the incidence of vulvar aching versus burning in patients with vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of vulvar aching versus burning in the patients with vulvodynia?; p = 0.2155, t-test proportion
Statistical Analysis 49: Comparison: Vulvodynia; Parameter: The difference in the incidence of vulvar aching versus soreness in patients with vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of vulvar aching versus soreness in the patients with vulvodynia?; p = 0.1508, t-test proportion
Statistical Analysis 50: Comparison: Vulvodynia; Parameter: The difference in the incidence of vulvar aching versus irritation in patients with vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of vulvar aching versus irritation in the patients with vulvodynia?; p = 0.6364, t-test proportion
Statistical Analysis 51: Comparison: Vulvodynia; Parameter: The difference in the incidence of vulvar aching versus the feeling of inflammation in patients with vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of vulvar aching versus the feeling of inflammation in the patients with vulvodynia?; p = 0.5277, t-test proportion
Statistical Analysis 52: Comparison: Vulvodynia; Parameter: The difference in the incidence of vulvar sticking versus knife-like pain in patients with vulvodynia who had sharp vulvar pain; Test type: Superiority — Question: Is there a difference in the incidence of vulvar sticking versus knife-like pain in the patients with vulvodynia who had sharp vulvar pain?; p = 0.2041, t-test proportion
Statistical Analysis 53: Comparison: Vulvodynia; Parameter: The difference in the incidence of vulvar sticking versus paper-cuts pain in patients with vulvodynia who had sharp vulvar pain; Test type: Superiority — Question: Is there a difference in the incidence of vulvar sticking versus paper-cuts pain in the patients with vulvodynia who had sharp vulvar pain?; p = 0.0412, t-test proportion
Statistical Analysis 54: Comparison: Vulvodynia; Parameter: The difference in the incidence of vulvar sticking versus stabbing in patients with vulvodynia who had sharp vulvar pain; Test type: Superiority — Question: Is there a difference in the incidence of vulvar sticking versus stabbing in the patients with vulvodynia who had sharp vulvar pain?; p = 0.7978, t-test proportion
Statistical Analysis 55: Comparison: Vulvodynia; Parameter: The difference in the incidence of vulvar stabbing versus knife-like pain in patients with vulvodynia who had sharp vulvar pain; Test type: Superiority — Question: Is there a difference in the incidence of vulvar stabbing versus knife-like pain in the patients with vulvodynia who had sharp vulvar pain?; p = 0.3094, t-test proportion
Statistical Analysis 56: Comparison: Vulvodynia; Parameter: The difference in the incidence of vulvar stabbing versus paper-cuts pain in patients with vulvodynia who had sharp vulvar pain; Test type: Superiority — Question: Is there a difference in the incidence of vulvar stabbing versus paper-cuts pain in the patients with vulvodynia who had sharp vulvar pain?; p = 0.0730, t-test proportion
Statistical Analysis 57: Comparison: Vulvar Dermatosis vs Vulvodynia; Parameter: The difference in the duration of vulvar complaints for more than 24 months among patients with vulvar dermatosis or vulvodynia; Test type: Equivalence — Question: Is there a difference in the duration of vulvar complaints for more than 24 months among patients with vulvar dermatosis and vulvodynia?; p = 0.4038, Chi-squared
Statistical Analysis 58: Comparison: Vulvar Dermatosis vs Vulvodynia; Parameter: The difference in the duration of vulvar complaints for more than 12 months among patients with vulvar dermatosis or vulvodynia; Test type: Equivalence — Question: Is there a difference in the duration of vulvar complaints for more than 12 months among patients with vulvar dermatosis and vulvodynia?; p = 0.7299, Chi-squared
Statistical Analysis 59: Comparison: Vulvar Dermatosis vs Vulvodynia; Parameter: The difference in the duration of vulvar complaints for more than six months among patients with vulvar dermatosis or vulvodynia; Test type: Equivalence — Question: Is there a difference in the duration of vulvar complaints for more than six months among patients with vulvar dermatosis and vulvodynia?; p = 0.7241, Chi-squared

17. Secondary Outcome: Sexual Activity and Abstinence in Patients With and Without Vulvar Discomfort
Description: The table shows sexual activity and sexual abstinence due to dyspareunia or lack of a sexual partner in four groups of patients.
Time Frame: ISSVD Questionnaire, up to 30 minutes for each participant.
Population: Sexual activity was evaluated anamnestically by the "ISSVD Vulvodynia Pattern Questionnaire."
Measure: Count of Participants; unit: Participants
Groups:
- Vulvodynia: Patients with vulvar discomfort (ISSVD Vulvodynia Pattern Questionnaire), who clinically fulfilled Friedrich's criteria. Non-specific lesions found with TRIV (some non-specific lesions of the vulva) were not relevant for diagnosis of vulvodynia.
Arm/Group | Normal Vulva | Impaired Vulvar Skin | Vulvodynia | Vulvar Dermatosis
Number analyzed (Participants) | 82 | 82 | 82 | 82
Participants
  Sexually Active Patients | 81 | 77 | 73 | 49
  No sexual activity | 1 | 5 | 9 | 33
  Sexual Abstinence Due To Dyspareunia | 1 | 1 | 8 | 1
  Dyspareunia And Lack Of Partner | 0 | 0 | 9 | 32
Statistical Analysis 1: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the sexual activity among patients from different groups; Test type: Equivalence — Question: Is there a difference in the sexual activity among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 2: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the frequency of dyspareunia as a cause of sexual inactivity among patients from different groups; Test type: Equivalence — Question: Is there a difference in the frequency of dyspareunia as a cause of sexual inactivity among patients from different groups?; p = 0.0006, Chi-squared
Statistical Analysis 3: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the frequency of sexual inactivity due to dyspareunia and lack of a sexual partner among patients from different groups; Test type: Equivalence — Question: Is there a difference in the frequency of sexual inactivity due to dyspareunia and lack of a sexual partner among patients from different groups?; p = 0.0000, Chi-squared

18. Secondary Outcome: Dyspareunia and Marinoff Index in Patients With and Without Vulvar Discomfort
Description: The table shows the degree of dyspareunia in sexually active patients with and without vulvar discomfort. We used Marinoff Index as a measure of the degree of dyspareunia.
  Negative Marinoff Index (0) is a sign of the absence of dyspareunia.
  Four grades of Marionoff Index are:
  Marinoff Index 0 = no dyspareunia; Marinoff Index 1= discomfort/pain with intercourse that doesn't interfere with the frequency of sex; Marinoff Index 2= pain with intercourse which sometimes prevents intercourse and Marinoff Index 3= pain with intercourse preventing any intercourse.
Time Frame: ISSVD Questionnaire, up to 30 minutes for each participant.
Population: Dyspareunia and Marinoff Index were evaluated anamnestically by the "ISSVD Vulvodynia Pattern Questionnaire". We assessed the degree of dyspareunia only in sexually active patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Vulva | Impaired Vulvar Skin | Vulvodynia | Vulvar Dermatosis
Number analyzed (Participants) | 81 | 77 | 73 | 34
Participants
  Dyspareunia | 1 | 1 | 73 | 34
  Marinoff Index 0 | 80 | 76 | 0 | 0
  Marinoff Index 1 | 1 | 0 | 22 | 7
  Marinoff Index 2 | 0 | 1 | 40 | 18
  Marinoff Index 3 | 0 | 0 | 11 | 9
Statistical Analysis 1: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the frequency of dyspareunia among patients from different groups; Test type: Equivalence — Question: Is there a difference in the frequency of dyspareunia among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 2: Comparison: Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the degree of dyspareunia (Marinoff Index) among sexually active patients with vulvodynia or vulvar dermatosis who had dyspareunia; Test type: Equivalence — Parameter: The difference in the degree of dyspareunia (Marinoff Index) among sexually active patients with vulvodynia or vulvar dermatosis who had dyspareunia; p = 0.2999, Chi-squared

19. Secondary Outcome: Aggravation Of Vulvar Complaints Depending On Sexual Intercourse In Patients With Vulvar Dermatosis And Vulvodynia
Description: The relationship between sexual vulvar discomfort and sexual intercourse (provocation and aggravation) in patients with vulvar dermatosis and vulvodynia, as recommended in the ISSVD Questionnaire.
Time Frame: ISSVD Questionnaire, up to 30 minutes for each participant.
Population: Provocation and aggravation of vulvar discomfort depending on sexual intercourse were evaluated anamnestically by the "ISSVD Vulvodynia Pattern Questionnaire."
Measure: Count of Participants; unit: Participants
Arm/Group | Vulvar Dermatosis | Vulvodynia
Number analyzed (Participants) | 82 | 82
Participants
  Sexually active patients | 49 | 73
  Intercourse aggravates vulvar discomfort | 0 | 27
  Penetration aggravates vulvar complaints | 16 | 39
  Vulvar complaints during intercourse | 15 | 21
  Vulvar complaints after intercourse | 14 | 42
Statistical Analysis 1: Comparison: Vulvar Dermatosis vs Vulvodynia; Parameter: The difference in the frequency of vulvar discomfort provoked through the intercourse in patients with vulvodynia and vulvar dermatosis; Test type: Equivalence — Question: Is there a difference in the incidence of the frequency of vulvar discomfort provoked through the intercourse in patients with vulvodynia and vulvar dermatosis?; p = 0.0000, Chi-squared
Statistical Analysis 2: Comparison: Vulvar Dermatosis vs Vulvodynia; Parameter: The difference in the frequency of vulvar discomfort provoked through the penetration in patients with vulvodynia and vulvar dermatosis; Test type: Equivalence — Question: Is there a difference in the frequency of vulvar discomfort provoked through the penetration in patients with vulvodynia and vulvar dermatosis?; p = 0.0347, Chi-squared
Statistical Analysis 3: Comparison: Vulvar Dermatosis vs Vulvodynia; Parameter: The difference in the frequency of vulvar discomfort aggravated through sexual intercourse in patients with vulvodynia and vulvar dermatosis; Test type: Equivalence — Question: Is there a difference in the frequency of vulvar discomfort aggravated through sexual intercourse in patients with vulvodynia and vulvar dermatosis?; p = 0.7068, Chi-squared
Statistical Analysis 4: Comparison: Vulvar Dermatosis vs Vulvodynia; Parameter: The difference in the frequency of vulvar discomfort aggravated after sexual intercourse in patients with vulvodynia and vulvar dermatosis; Test type: Equivalence — Question: Is there a difference in the frequency of vulvar discomfort aggravated after sexual intercourse in patients with vulvodynia and vulvar dermatosis?; p = 0.0025, Chi-squared

20. Secondary Outcome: Aggravation of Vulvar Discomfort Through Various Triggers in Patients With Vulvar Dermatosis and Vulvodynia
Description: The table shows the relationship among worsening of vulvar discomfort by using tampons, cycling, wearing tight clothes, menstruation, and urination in patients with vulvar dermatosis and vulvodynia.
Time Frame: ISSVD Questionnaire, up to 30 minutes for each participant.
Population: Worsening of vulvar discomfort by the using of tampons, cycling, wearing tight clothes, menstruation and urination in symptomatic patients were evaluated anamnestically by the "ISSVD Vulvodynia Pattern Questionnaire".
Measure: Count of Participants; unit: Participants
Arm/Group | Vulvar Dermatosis | Vulvodynia
Number analyzed (Participants) | 82 | 82
Participants
  Using of tampons | 21 | 54
  Tampon aggravates vulvar complaints | 7 | 21
  Cycling | 19 | 42
  Cycling aggravates vulvar complaints | 9 | 26
  Wearing tight clothes | 44 | 70
  Tight clothes aggravates vulvar complaints | 26 | 46
  Menstrual cycle | 36 | 76
  Influence of menstrual cycle on symptoms | 15 | 44
  Worsening before menstrual bleeding | 5 | 27
  Worsening during menstrual bleeding | 4 | 6
  Worsening after menstrual bleeding | 7 | 18
  Worsening between menstrual bleeding | 3 | 4
  Worsening during urination | 30 | 39
  Worsening during urination after intercourse | 7 | 14
Statistical Analysis 1: Comparison: Vulvar Dermatosis vs Vulvodynia; Parameter: The difference in the frequency of use of vaginal tampon among patients with vulvodynia and vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the frequency of use of vaginal tampon among patients with vulvodynia and vulvar dermatosis?; p = 0.0000, Chi-squared
Statistical Analysis 2: Comparison: Vulvar Dermatosis vs Vulvodynia; Parameter: The difference in the frequency of worsening of vulvar discomfort due to the use of vaginal tampon in symptomatic patients, who use vaginal tampons; Test type: Superiority — Question: Is there a difference in the frequency of worsening of vulvar discomfort due to the use of vaginal tampon in symptomatic patients, who use vaginal tampons?; p = 0.6552, Chi-squared
Statistical Analysis 3: Comparison: Vulvar Dermatosis vs Vulvodynia; Parameter: The difference in the frequency of cycling among patients with vulvodynia and vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the frequency of cycling among patients with vulvodynia and vulvar dermatosis?; p = 0.0002, Chi-squared
Statistical Analysis 4: Comparison: Vulvar Dermatosis vs Vulvodynia; Parameter: The difference in the frequency of worsening of vulvar discomfort due to the cycling in symptomatic patients, who ride a bicycle; Test type: Superiority — Question: Is there a difference in the frequency of worsening of vulvar discomfort due to the cycling in symptomatic patients, who ride a bicycle?; p = 0.2877, Chi-squared
Statistical Analysis 5: Comparison: Vulvar Dermatosis vs Vulvodynia; Parameter: The difference in the frequency of wearing tight clothes among patients with vulvar dermatosis and vulvodynia; Test type: Superiority — Question: Is there a difference in the frequency of wearing tight clothes among patients with vulvar dermatosis and vulvodynia?; p = 0.0001, Chi-squared
Statistical Analysis 6: Comparison: Vulvar Dermatosis vs Vulvodynia; Parameter: The difference in the frequency of worsening of vulvar discomfort due to wearing of tight clothes in symptomatic patients, who wear tight clothes; Test type: Superiority — Question: Is there a difference in the frequency of worsening of vulvar discomfort due to wearing of tight clothes in symptomatic patients, who wear tight clothes?; p = 0.4754, Chi-squared
Statistical Analysis 7: Comparison: Vulvar Dermatosis vs Vulvodynia; Parameter: The difference in the frequency of worsening of vulvar discomfort depending on the menstrual cycle in symptomatic patients of reproductive age; Test type: Superiority — Question: Is there a difference in the frequency of worsening of vulvar discomfort depending on the menstrual cycle in symptomatic patients of reproductive age?; p = 0.1082, Chi-squared
Statistical Analysis 8: Comparison: Vulvar Dermatosis vs Vulvodynia; Parameter: The difference in the frequency of worsening of vulvar discomfort before starting menstrual bleeding in symptomatic patients of reproductive age; Test type: Superiority — Question: Is there a difference in the frequency of worsening of vulvar discomfort before starting menstrual bleeding in symptomatic patients of reproductive age?; p = 0.0179, Chi-squared
Statistical Analysis 9: Comparison: Vulvar Dermatosis vs Vulvodynia; Parameter: The difference in the frequency of worsening of vulvar discomfort during menstrual bleeding in symptomatic patients of reproductive age; Test type: Superiority — Question: Is there a difference in the frequency of worsening of vulvar discomfort during menstrual bleeding in symptomatic patients of reproductive age?; p = 0.5722, Chi-squared
Statistical Analysis 10: Comparison: Vulvar Dermatosis vs Vulvodynia; Parameter: The difference in the frequency of worsening of vulvar discomfort after menstrual bleeding in symptomatic patients of reproductive age; Test type: Superiority — Question: Is there a difference in the frequency of worsening of vulvar discomfort after menstrual bleeding in symptomatic patients of reproductive age?; p = 0.6148, Chi-squared
Statistical Analysis 11: Comparison: Vulvar Dermatosis vs Vulvodynia; Parameter: The difference in the frequency of worsening of vulvar discomfort between two menstrual bleeding in symptomatic patients of reproductive age; Test type: Superiority — Question: Is there a difference in the frequency of worsening of vulvar discomfort between two menstrual bleeding in symptomatic patients of reproductive age?; p = 0.5307, Chi-squared
Statistical Analysis 12: Comparison: Vulvar Dermatosis vs Vulvodynia; Parameter: The difference in the frequency of worsening of vulvar discomfort during urination; Test type: Superiority — Question: Is there a difference in the frequency of worsening of vulvar discomfort during urination?; p = 0.1546, Chi-squared
Statistical Analysis 13: Comparison: Vulvar Dermatosis vs Vulvodynia; Parameter: The difference in the frequency of worsening of vulvar complaints during urination after sexual intercourse in symptomatic patients, who are sexually active; Test type: Superiority — Question: Is there a difference in the frequency of worsening of vulvar complaints during urination after sexual intercourse in symptomatic patients, who are sexually active?; p = 0.1019, Chi-squared

21. Secondary Outcome: Problems Associated With Urination and Defecation in Patients With and Without Vulvar Discomfort
Description: The table shows the incidence of the problems with urination and defecation in four groups of patients with and without vulvar discomfort.
Time Frame: ISSVD Questionnaire, up to 30 minutes for each participant.
Population: Problems with urination and defecation were evaluated anamnestically by the "ISSVD Vulvodynia Pattern Questionnaire".
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Vulva | Impaired Vulvar Skin | Vulvodynia | Vulvar Dermatosis
Number analyzed (Participants) | 82 | 82 | 82 | 82
Participants
  Any Problem With Urinating and Defecation | 54 | 47 | 74 | 72
  Dysuria | 7 | 7 | 36 | 33
  Intermittent Dysuria | 7 | 7 | 26 | 26
  Frequent Dysuria | 0 | 0 | 10 | 7
  Urinary Incontinence | 16 | 11 | 19 | 32
  Intermittent Urinary Incontinence | 16 | 10 | 17 | 21
  Frequent Urinary Incontinence | 0 | 1 | 2 | 11
  Difficulties At Starting Urination | 2 | 1 | 12 | 9
  Intermittent Diff. At Starting Urination | 2 | 0 | 11 | 7
  Frequent Diff. At Starting Urination | 0 | 1 | 1 | 2
  Urgency | 11 | 11 | 24 | 24
  Intermittent Urgency | 11 | 11 | 22 | 15
  Frequent Urgency | 0 | 0 | 2 | 9
  Nocturia | 30 | 22 | 40 | 56
  Intermittent Nocturia | 25 | 20 | 31 | 30
  Frequent Nocturia | 5 | 2 | 9 | 26
  Recurrent Cystitis | 8 | 4 | 15 | 10
  Constipation | 12 | 16 | 27 | 20
  Intermittent Constipation | 9 | 13 | 20 | 14
  Frequent Constipation | 3 | 3 | 7 | 6
  Diarrhea | 3 | 2 | 9 | 12
  Intermittent Diarrhea | 3 | 1 | 7 | 10
  Frequent Diarrhea | 0 | 1 | 2 | 2
  Irritable Colon | 0 | 2 | 7 | 9
Statistical Analysis 1: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of problems associated with urination and defecation between patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of problems associated with urination and defecation between patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 2: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of dysuria between patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of dysuria between patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 3: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of intermittent dysuria between patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of intermittent dysuria between patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 4: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of frequent dysuria between patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of frequent dysuria between patients from different groups?; p = 0.0003, Chi-squared
Statistical Analysis 5: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of urinary incontinence between patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of urinary incontinence between patients from different groups?; p = 0.0010, Chi-squared
Statistical Analysis 6: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of intermittent urinary incontinence between patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of intermittent urinary incontinence between patients from different groups?; p = 0.1859, Chi-squared
Statistical Analysis 7: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of frequent urinary incontinence between patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of frequent urinary incontinence between patients from different groups?; p = 0.0003, Chi-squared
Statistical Analysis 8: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of difficulties at starting urination between patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of difficulties at starting urination between patients from different groups?; p = 0.0015, Chi-squared
Statistical Analysis 9: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of intermittent difficulties at starting urination between patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of intermittent difficulties at starting urination between patients from different groups?; p = 0.0013, Chi-squared
Statistical Analysis 10: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of frequent difficulties at starting urination between patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of frequent difficulties at starting urination between patients from different groups?; p = 0.5673, Chi-squared
Statistical Analysis 11: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of urgency between patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of urgency between patients from different groups?; p = 0.0065, Chi-squared
Statistical Analysis 12: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of intermittent urgency between patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of intermittent urgency between patients from different groups?; p = 0.0830, Chi-squared
Statistical Analysis 13: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of frequent urgency between patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of frequent urgency between patients from different groups?; p = 0.0001, Chi-squared
Statistical Analysis 14: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of nocturia between patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of nocturia between patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 15: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of intermittent nocturia between patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of intermittent nocturia between patients from different groups?; p = 0.2315, Chi-squared
Statistical Analysis 16: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of frequent nocturia between patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of frequent nocturia between patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 17: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of recurrent cystitis between patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of recurrent cystitis between patients from different groups?; p = 0.0539, Chi-squared
Statistical Analysis 18: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of constipation between patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of constipation between patients from different groups?; p = 0.0379, Chi-squared
Statistical Analysis 19: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of intermittent constipation between patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of intermittent constipation between patients from different groups?; p = 0.1485, Chi-squared
Statistical Analysis 20: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of frequent constipation between patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of frequent constipation between patients from different groups?; p = 0.4155, Chi-squared
Statistical Analysis 21: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of diarrhea between patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of diarrhea between patients from different groups?; p = 0.0092, Chi-squared
Statistical Analysis 22: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of intermittent diarrhea between patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of intermittent diarrhea between patients from different groups?; p = 0.0192, Chi-squared
Statistical Analysis 23: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of frequent diarrhea between patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of frequent diarrhea between patients from different groups?; p = 0.5253, Chi-squared
Statistical Analysis 24: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of the irritable colon between patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of the irritable colon between patients from different groups?; p = 0.0060, Chi-squared

22. Secondary Outcome: Other Associated Symptoms and Diseases in Patients With and Without Vulvar Discomfort
Description: The table shows the incidence of the other associated symptoms and diseases in four groups of patients, as recommended in the ISSVD Questionnaire.
Time Frame: ISSVD Questionnaire, up to 30 minutes for each participant.
Population: Other associated symptoms and diseases were evaluated anamnestically by the "ISSVD Vulvodynia Pattern Questionnaire".
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Vulva | Impaired Vulvar Skin | Vulvodynia | Vulvar Dermatosis
Number analyzed (Participants) | 82 | 82 | 82 | 82
Participants
  Other Symptoms and Diseases | 52 | 58 | 79 | 75
  Recurrent Headache | 13 | 17 | 21 | 14
  Chronic Fatigue | 4 | 10 | 28 | 25
  Lumbar Pain | 14 | 24 | 40 | 34
  Fibromyalgia | 3 | 13 | 31 | 23
  Energy Loss | 11 | 22 | 50 | 43
  Sleep Disorders | 9 | 14 | 23 | 35
  Pelvic Pain | 2 | 7 | 28 | 17
  Unintended Weight Loss | 7 | 1 | 6 | 4
  Endometriosis | 1 | 4 | 6 | 4
  "D-D-D Triad" | 0 | 1 | 7 | 1
  Hypertension | 2 | 0 | 2 | 22
  Angina pectoris | 0 | 0 | 0 | 2
  Diabetes mellitus | 0 | 0 | 0 | 2
  Genital Herpes | 2 | 1 | 2 | 2
  Thyroid Disease | 11 | 8 | 24 | 24
  Drug Allergy | 9 | 8 | 15 | 8
  Recurrent Attacs of Sinusitis | 10 | 26 | 23 | 15
  HPV Testing | 29 | 36 | 45 | 19
  Positive Human Papillomavirus (HPV) test | 9 | 20 | 19 | 10
  Abnormal Papanicolaou (PAP) Smear | 8 | 19 | 25 | 10
  Genital Warts | 1 | 3 | 6 | 3
  Conization | LETZ (Loop Excis. of the Trans. Zone) | 4 | 11 | 10 | 7
Statistical Analysis 1: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of any associated symptom or disease among patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of any associated symptom or disease among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 2: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of a frequent headache among patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of a frequent headache among patients from different groups?; p = 0.3957, Chi-squared
Statistical Analysis 3: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of chronic fatigue among patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of chronic fatigue among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 4: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of lumbar pain among patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of lumbar pain among patients from different groups?; p = 0.0001, Chi-squared
Statistical Analysis 5: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of fibromyalgia among patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of fibromyalgia among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 6: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of energy loss among patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of energy loss among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 7: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of sleep disorders among patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of sleep disorders among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 8: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of pelvic pain among patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of pelvic pain among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 9: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of unintended weight loss among patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of unintended weight loss among patients from different groups?; p = 0.1764, Chi-squared
Statistical Analysis 10: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of endometriosis among patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of endometriosis among patients from different groups?; p = 0.3127, Chi-squared
Statistical Analysis 11: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the difference in the incidence of "D-D-D Triad" (Dysmenorrhoea-Dyspareunia-Dysuria) among patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of "D-D-D Triad" among patients from different groups?; p = 0.0028, Chi-squared
Statistical Analysis 12: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of hypertension among patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of hypertension among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 13: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of genital herpes among patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of genital herpes among patients from different groups?; p = 0.9323, Chi-squared
Statistical Analysis 14: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of thyroid disease among patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of thyroid disease among patients from different groups?; p = 0.0011, Chi-squared
Statistical Analysis 15: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of drug allergy among patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of drug allergy among patients from different groups?; p = 0.2756, Chi-squared
Statistical Analysis 16: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of recurrent attacks of sinusitis among patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of recurrent attacks of sinusitis among patients from different groups?; p = 0.0105, Chi-squared
Statistical Analysis 17: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of HPV infection among patients from different groups, who were tested for HPV; Test type: Equivalence — Question: Is there a difference in the incidence of HPV infection among patients from different groups, who were tested for HPV?; p = 0.2128, Chi-squared
Statistical Analysis 18: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of abnormal PAP smear among patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of abnormal PAP smear among patients from different groups?; p = 0.0018, Chi-squared
Statistical Analysis 19: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of genital warts among patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of genital warts among patients from different groups?; p = 0.2524, Chi-squared
Statistical Analysis 20: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of conization or LETZ among patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of conization or LETZ among patients from different groups?; p = 0.2452, Chi-squared

23. Secondary Outcome: Previous Treatment of Patients With Vulvar Dermatosis and Vulvodynia
Description: The table shows the incidence of the previous treatment in patients with vulvar dermatosis and vulvodynia.
Time Frame: ISSVD Questionnaire, up to 30 minutes for each participant.
Population: Previous treatment was evaluated anamnestically by the "ISSVD Vulvodynia Pattern Questionnaire".
Measure: Count of Participants; unit: Participants
Arm/Group | Vulvar Dermatosis | Vulvodynia
Number analyzed (Participants) | 82 | 82
Participants
  Any prior treatment | 33 | 42
  Antifungals Local | 26 | 39
  Antifungals Systemic | 10 | 12
  Antibiotics Local | 18 | 22
  Antibiotics Systemic | 11 | 17
  Corticosteroids Local | 25 | 5
  Corticosteroids Systemic | 1 | 0
  Antidepressants | 1 | 5
Statistical Analysis 1: Comparison: Vulvar Dermatosis vs Vulvodynia; Parameter: The difference in the frequency of any previous treatment between patients with vulvar dermatosis and vulvodynia; Test type: Superiority — Question: Is there a difference in the frequency of any previous treatment between patients with vulvar dermatosis and vulvodynia?; p = 0.1583, Chi-squared
Statistical Analysis 2: Comparison: Vulvar Dermatosis vs Vulvodynia; Parameter: The difference in the frequency of previous local treatment with antifungals among patients with vulvar dermatosis and vulvodynia; Test type: Superiority — Question: Is there a difference in the frequency of previous local treatment with antifungals between the patients with vulvar dermatosis and vulvodynia?; p = 0.0380, Chi-squared
Statistical Analysis 3: Comparison: Vulvar Dermatosis vs Vulvodynia; Parameter: The difference in the frequency of previous systemic treatment with antifungals among patients with vulvar dermatosis and vulvodynia; Test type: Superiority — Question: Is there a difference in the frequency of previous systemic treatment with antifungals between the patients with vulvar dermatosis and vulvodynia?; p = 0.6468, Chi-squared
Statistical Analysis 4: Comparison: Vulvar Dermatosis vs Vulvodynia; Parameter: The difference in the frequency of previous local treatment with antibiotics among patients with vulvar dermatosis and vulvodynia; Test type: Superiority — Question: Is there a difference in the frequency of previous local treatment with antibiotics between the patients with vulvar dermatosis and vulvodynia?; p = 0.4670, Chi-squared
Statistical Analysis 5: Comparison: Vulvar Dermatosis vs Vulvodynia; Parameter: The difference in the frequency of previous systemic treatment with antibiotics among patients with vulvar dermatosis and vulvodynia; Test type: Superiority — Question: Is there a difference in the frequency of previous systemic treatment with antibiotics between the patients with vulvar dermatosis and vulvodynia?; p = 0.2131, Chi-squared
Statistical Analysis 6: Comparison: Vulvar Dermatosis vs Vulvodynia; Parameter: The difference in the frequency of previous local treatment with corticoids among patients with vulvar dermatosis and vulvodynia; Test type: Superiority — Question: Is there a difference in the frequency of previous local treatment with corticosteroids between the patients with vulvar dermatosis and vulvodynia?; p = 0.0000, Chi-squared
Statistical Analysis 7: Comparison: Vulvar Dermatosis vs Vulvodynia; Parameter: The difference in the frequency of previous systemic treatment with antidepressant among patients with vulvar dermatosis and vulvodynia; Test type: Superiority — Question: Is there a difference in the frequency of previous systemic treatment with antidepressant between the patients with vulvar dermatosis and vulvodynia?; p = 0.0962, Chi-squared

24. Secondary Outcome: Cotton Swab Test (Q-Tip) in Patients With and Without Vulvar Discomfort
Description: The table shows the results of Cotton-Swab Test in four groups of patients. Cotton-Swab Test or Q-Tip Testing is part of a multidisciplinary approach to the assessment of sexual pain, especially, vulvodynia or vestibulodynia, in women. ISSVD recommended the Cotton-Swab test for the differential diagnosis of vulvodynia.
  The test consists of using a cotton-swab to palpate multiple vulvar and vestibular site while recording the woman's pain.
  We performed Cotton-Swab Test by touching the vulva at 6 points (each vulvar ring), organized into locations based on a clock face and marked like the hours on the clock: 2h, 4h, 6h, 8h, 10h, and 12 h.
Time Frame: Cotton Swab Test, up to 10 minutes for each participant.
Population: Cotton-Swab test was evaluated by clinical examination of the Inner Vulvar Ring ("TRIV Data Form").
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Vulva | Impaired Vulvar Skin | Vulvodynia | Vulvar Dermatosis
Number analyzed (Participants) | 82 | 82 | 82 | 82
Participants
  Positive Cotton Swab Test, generally (any point) | 10 | 11 | 73 | 28
  Positive Cotton Swab at the point of 2h | 2 | 4 | 34 | 9
  Positive Cotton Swab at the point of 4h | 6 | 9 | 58 | 17
  Positive Cotton Swab at the point of 6h | 7 | 11 | 62 | 21
  Positive Cotton Swab at the point of 8h | 6 | 11 | 59 | 18
  Positive Cotton Swab at the point of 10h | 4 | 9 | 42 | 11
  Positive Cotton Swab at the point of 12h | 3 | 8 | 38 | 9
Statistical Analysis 1: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of a positive Cotton-Swab test of the vulva among patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of a positive Cotton-Swab test of the vulva among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 2: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of a positive Cotton-Swab test at the point marked as 2h among patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of a positive Cotton-Swab test at the point marked as 2h among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 3: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of a positive Cotton-Swab test at the point marked as 4h among patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of a positive Cotton-Swab test at the point marked as 4h among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 4: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of a positive Cotton-Swab test at the point marked as 6h among patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of a positive Cotton-Swab test at the point marked as 6h among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 5: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of a positive Cotton-Swab test at the point marked as 8h among patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of a positive Cotton-Swab test at the point marked as 8h among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 6: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of a positive Cotton-Swab test at the point marked as 10h among patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of a positive Cotton-Swab test at the point marked as 10h among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 7: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of a positive Cotton-Swab test at the point marked as 12h among patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of a positive Cotton-Swab test at the point marked as 12h among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 8: Comparison: Normal Vulva vs Vulvar Dermatosis; Parameter: The difference in the incidence of a positive Cotton-Swab test of the vulva in patients with vulvar dermatosis versus normal vulva; Test type: Superiority — Question: Is there a difference in the incidence of a positive Cotton-Swab test of the vulva in patients with vulvar dermatosis versus normal vulva?; p = 0.0009, Chi-squared
Statistical Analysis 9: Comparison: Normal Vulva vs Vulvar Dermatosis; Parameter: The difference in the incidence of a positive Cotton-Swab test at the point marked as 2h in patients with vulvar dermatosis versus normal vulva; Test type: Superiority — Question: Is there a difference in the incidence of a positive Cotton-Swab test at the point marked as 2h in patients with vulvar dermatosis versus normal vulva?; p = 0.0289, Chi-squared
Statistical Analysis 10: Comparison: Normal Vulva vs Vulvar Dermatosis; Parameter: The difference in the incidence of a positive Cotton-Swab test at the point marked as 4h in patients with vulvar dermatosis and normal vulva; Test type: Superiority — Question: Is there a difference in the incidence of a positive Cotton-Swab test at the point marked as 4h in patients with vulvar dermatosis versus normal vulva?; p = 0.0134, Chi-squared
Statistical Analysis 11: Comparison: Normal Vulva vs Vulvar Dermatosis; Parameter: The difference in the incidence of a positive Cotton-Swab test at the point marked as 6h in patients with vulvar dermatosis and normal vulva; Test type: Superiority — Question: Is there a difference in the incidence of a positive Cotton-Swab test at the point marked as 6h in patients with vulvar dermatosis versus normal vulva?; p = 0.0037, Chi-squared
Statistical Analysis 12: Comparison: Normal Vulva vs Vulvar Dermatosis; Parameter: The difference in the incidence of a positive Cotton-Swab test at the point marked as 8h in patients with vulvar dermatosis and normal vulva; Test type: Superiority — Question: Is there a difference in the incidence of a positive Cotton-Swab test at the point marked as 8h in patients with vulvar dermatosis and normal vulva?; p = 0.0080, Chi-squared
Statistical Analysis 13: Comparison: Normal Vulva vs Vulvar Dermatosis; Parameter: The difference in the incidence of a positive Cotton-Swab test at the point marked as 10h in patients with vulvar dermatosis and normal vulva; Test type: Superiority — Question: Is there a difference in the incidence of a positive Cotton-Swab test at the point marked as 10h in patients with vulvar dermatosis versus normal vulva?; p = 0.0579, Chi-squared
Statistical Analysis 14: Comparison: Normal Vulva vs Vulvar Dermatosis; Parameter: The difference in the incidence of a positive Cotton-Swab test at the point marked as 12h in patients with vulvar dermatosis and normal vulva; Test type: Superiority — Question: Is there a difference in the incidence of a positive Cotton-Swab test at the point marked as 12h in patients with vulvar dermatosis versus normal vulva?; p = 0.0720, Chi-squared

25. Secondary Outcome: Distribution of Non-Specific and Specific Vulvar Lesions in Relation to The Three Vulvar Rings (TRIV)
Description: The table shows the distribution of non-specific and specific vulvar lesions in relation to the three vulvar rings (TRIV).
  The "OUTER Vulvar Ring" includes vulvar skin, the "MIDDLE Vulvar Ring" encompasses the modified mucosa, and the "INNER Vulvar Ring" is presented with glicogenized mucosa.
  "Non-Specific Lesions" include non-specific erythema, punctuations, papillae, paleness and smoothness, fissures or sores in the absence of infection and pre/malignancy in any part of the vulva.
  "Specific Lesions" comprise eczematous inflammation with thickened, excoriated skin within chronic lichen simplex; hypopigmented or white lesions, fusion or resorption of the labia minora and clitoral hood, loss of vulvar architecture and sclerotic changes in lichen sclerosis; white reticular pattern to extensive erosion with agglutination or resorption of the labia within lichen planus and psoriatic erythematous papules with silver, scaly plaques.
Time Frame: Three Rings Vulvoscopy, up to 45 minutes for each participant.
Population: "Three Rings Vulvoscopy" was performed in 328 patients, classified into four groups based on anamnestic data and clinical examination. Localization and specificity of the lesions were mapped into the "TRIV Form Data." Vulvar lesions in patients with vulvodynia were not relevant to the diagnosis of vulvodynia which was made by Friedrich's criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Vulva | Impaired Vulvar Skin | Vulvodynia | Vulvar Dermatosis
Number analyzed (Participants) | 82 | 82 | 82 | 82
Participants
  Non-specific Findings of the Outer Vulvar Ring | 0 | 4 | 15 | 58
  Non-specific Findings of the Middle Vulvar Ring | 26 | 71 | 79 | 68
  Non-specific Findings of the Inner Vulvar Ring | 32 | 79 | 81 | 70
  Erythema of the Outer Vulvar Ring | 0 | 3 | 12 | 27
  Erythema of the Middle Vulvar Ring | 2 | 41 | 62 | 45
  Erythema of the Inner Vulvar Ring | 11 | 61 | 76 | 59
  Excoriations of the Outer Vulvar Ring | 0 | 0 | 2 | 23
  Fissures of the Middle Vulvar Ring | 0 | 0 | 2 | 29
  Fissures of the Inner Vulvar Ring | 0 | 0 | 0 | 3
  Rhagades of the Outer Vulvar Ring | 0 | 1 | 0 | 32
  Smoothness of the Middle Vulvar Ring | 0 | 3 | 0 | 13
  Smoothness of the Inner Vulvar Ring | 12 | 23 | 41 | 28
  Ischemia of the Middle Vulvar Ring | 0 | 5 | 6 | 2
  Ischemia of the Inner Vulvar Ring | 6 | 36 | 40 | 27
  Punctuation of the Middle Vulvar Ring | 0 | 1 | 8 | 3
  Punctuation of the Inner Vulvar Ring | 0 | 36 | 45 | 20
  Papillae of the Inner Vulvar Ring | 9 | 21 | 21 | 2
  Specific Lesions of the Outer Vulvar Ring | 0 | 0 | 0 | 73
  Specific Lesions of the Middle Vulvar Ring | 0 | 0 | 0 | 66
  Specific Lesions of the Inner Vulvar Ring | 0 | 0 | 0 | 49
Statistical Analysis 1: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of non-specific lesions of the Outer Vulvar Ring in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of the Outer Vulvar Ring between patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 2: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of non-specific lesions of the Middle Vulvar Ring in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy". Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of the Middle Vulvar Ring between patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 3: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of non-specific lesions of the Inner Vulvar Ring in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of the Inner Vulvar Ring between patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 4: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of erythema of the Outer Vulvar Ring in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of erythema of the Outer Vulvar Ring between patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 5: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of erythema of the Middle Vulvar Ring in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of erythema of the Middle Vulvar Ring between patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 6: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of erythema of the Inner Vulvar Ring in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of erythema of the Inner Vulvar Ring between patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 7: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of excoriations of the Outer Vulvar Ring in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of excoriations of the Outer Vulvar Ring between patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 8: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of fissures of the Middle Vulvar Ring in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of fissures the Middle Vulvar Ring between patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 9: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of rhagades of the Outer Vulvar Ring in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of rhagades of the Outer Vulvar Ring between patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 10: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of smoothness of the Middle Vulvar Ring in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of vulvodynia; Test type: Superiority — Question: Is there a difference in the frequency of smoothness of the Middle Vulvar Ring between patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 11: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of smoothness of the Inner Vulvar Ring in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of smoothness of the Inner Vulvar Ring between patients within different groups?; p = 0.0000, Chi-squared
Statistical Analysis 12: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of ischemia of the Middle Vulvar Ring in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of ischemia of the Middle Vulvar Ring between patients from different groups?; p = 0.0632, Chi-squared
Statistical Analysis 13: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of ischemia of the Inner Vulvar Ring in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of ischemia of the Inner Vulvar Ring between patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 14: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of punctuation of the Middle Vulvar Ring in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of punctuation of the Middle Vulvar Ring between patients within different groups?; p = 0.0043, Chi-squared
Statistical Analysis 15: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of punctuation of the Inner Vulvar Ring in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Typ), evaluated with "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of punctuation of the Inner Vulvar Ring between patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 16: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of papillae of the Inner Vulvar Ring in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of papillae of the Inner Vulvar Ring between patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 17: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of non-specific lesions of the Outer versus non-specific lesions of the Middle Vulvar Ring in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of the Outer versus non-specific lesions of the Middle Vulvar Ring in patients with vulvar dermatosis?; p = 0.0697, t-test proportion
Statistical Analysis 18: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of non-specific lesions of the Outer versus non-specific lesions of the Inner Vulvar Ring in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of the Outer versus non-specific lesions of the Inner Vulvar Ring in patients with vulvar dermatosis?; p = 0.0319, t-test proportion
Statistical Analysis 19: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of non-specific lesions of Middle versus non-specific lesions of the Inner Vulvar Ring in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of Middle versus non-specific lesions of the Inner Vulvar Ring in patients with vulvar dermatosis?; p = 0.7273, t-test proportion
Statistical Analysis 20: Comparison: Vulvodynia; Parameter: The difference in the incidence of non-specific lesions of the Outer versus non-specific lesions of the Middle Vulvar Ring in patients with vulvodynia. The diagnosis of vulvodynia was based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection, Q-Tip) following Friedrich's criteria. Vulvoscopic lesions were not relevant to the diagnosis of vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of the Outer versus non-specific lesions of the Middle Vulvar Ring in patients with vulvodynia?; p = 0.0000, t-test proportion
Statistical Analysis 21: Comparison: Vulvodynia; Parameter: The difference in the incidence of non-specific lesions of the Outer versus non-specific lesions of the Inner Vulvar Ring in patients with vulvodynia. The diagnosis of vulvodynia was based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection, Q-Tip) following Friedrich's criteria. Vulvoscopic lesions were not relevant to the diagnosis of vulvodynia; Test type: Superiority — [test comment as in outcome 25, analysis 20]; p = 0.0000, t-test proportion
Statistical Analysis 22: Comparison: Vulvodynia; Parameter: The difference in the incidence of non-specific lesions of the Middle versus non-specific lesions of the Inner Vulvar Ring in patients with vulvodynia. The diagnosis of vulvodynia was based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection, Q-Tip) following Friedrich's criteria. Vulvoscopic lesions were not relevant to the diagnosis of vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of the Middle versus non-specific lesions of the Inner Vulvar Ring in patients with vulvodynia?; p = 0.2203, t-test proportion
Statistical Analysis 23: Comparison: Impaired Vulvar Skin; Parameter: The difference in the incidence of non-specific lesions of the Outer versus non-specific lesions of the Middle Vulvar Ring in patients with impaired vulvar skin; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of Outer versus non-specific lesions of the Middle Vulvar Ring in patients with impaired vulvar skin?; p = 0.0000, t-test proportion
Statistical Analysis 24: Comparison: Impaired Vulvar Skin; Parameter: The difference in the incidence of non-specific lesions of the Outer versus non-specific lesions of the Inner Vulvar Ring in patients with impaired vulvar skin; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of Outer versus non-specific lesions of the Inner Vulvar Ring in patients with impaired vulvar skin?; p = 0.0000, t-test proportion
Statistical Analysis 25: Comparison: Impaired Vulvar Skin; Parameter: The incidence of non-specific lesions of the Middle versus non-specific lesions of the Inner Vulvar Ring in patients with impaired vulvar skin; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of the Middle versus non-specific lesions of the Inner Vulvar Ring in patients with impaired vulvar skin?; p = 0.1456, t-test proportion
Statistical Analysis 26: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of specific lesions of the Outer versus specific lesions of the Middle Vulvar Ring in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of specific lesions of the Outer versus specific lesions of the Middle Vulvar Ring in patients with vulvar dermatosis?; p = 0.1133, t-test proportion
Statistical Analysis 27: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of specific lesions of the Outer versus specific lesions of the Inner Vulvar Ring in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of specific lesions of the Outer versus specific lesions of the Inner Vulvar Ring in patients with vulvar dermatosis?; p = 0.0000, t-test proportion
Statistical Analysis 28: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of specific lesions of the Middle versus specific lesions of the Inner Vulvar Ring in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of specific lesions of the Middle versus specific lesions of the Inner Vulvar Ring in patients with vulvar dermatosis?; p = 0.0058, t-test proportion

26. Secondary Outcome: Distribution of Non-Specific and Specific Lesions of the Outer Vulvar Ring According to the "Three Rings Vulvoscopy"
Description: The table shows the distribution of the non-specific and specific lesions of the vulva according to individual structures of the Outer Vulvar Ring according to the TRIV.
  The "OUTER Vulvar Ring" includes vulvar skin with the following structures: mons pubis, labia majora, and the perineum.
  "Non-Specific Lesions" include non-specific erythema, punctuations, papillae, paleness and smoothness, fissures or sores in the absence of infection and pre/malignancy in any part of the vulva.
  "Specific Lesions" (lesions specific for vulvar dermatosis) comprise eczematous inflammation with thickened, excoriated skin within chronic lichen simplex; hypopigmented or white lesions, fusion or resorption of the labia minora and clitoral hood, loss of vulvar architecture and sclerotic changes in lichen sclerosis; white reticular pattern to extensive erosion with agglutination or resorption of the labia within lichen planus and psoriatic erythematous papules with silver, scaly plaques.
Time Frame: Three Rings Vulvoscopy, up to 45 minutes for each participant.
Population: "Three Rings Vulvoscopy" was performed in 328 patients, classified into four groups based on anamnestic data and clinical examination. Localization and specificity of the lesions were mapped into the "TRIV Form Data". Vulvar lesions in patients with vulvodynia were not relevant for the diagnosis of vulvodynia which was made by Friedrich's criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Vulva | Impaired Vulvar Skin | Vulvodynia | Vulvar Dermatosis
Number analyzed (Participants) | 82 | 82 | 82 | 82
Participants
  Non-specific Lesions of Mons Pubis | 0 | 1 | 2 | 18
  Non-specific Lesions of Labia Majora | 0 | 1 | 7 | 38
  Non-specific Lesions of the Perineum | 0 | 4 | 15 | 51
  Erythema of Mons Pubis | 0 | 1 | 2 | 12
  Erythema of Labia Majora | 0 | 1 | 6 | 24
  Erythema of the Perineum | 0 | 3 | 11 | 20
  Excoriations of Mons Pubis | 0 | 0 | 0 | 9
  Excoriations of Labia Majora | 0 | 0 | 0 | 18
  Excoriations of the Perineum | 0 | 0 | 2 | 16
  Rhagades of Mons Pubis | 0 | 0 | 0 | 5
  Rhagades of Labia Majora | 0 | 0 | 0 | 12
  Rhagades of the Perineum | 0 | 1 | 0 | 28
  Specific Lesions of Mons Pubis | 0 | 0 | 0 | 30
  Specific Lesions of Labia Majora | 0 | 0 | 0 | 55
  Specific Lesions of the Perineum | 0 | 0 | 0 | 65
Statistical Analysis 1: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of non-specific lesions of Mons pubis in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant for the diagnosis of the vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of Mons Pubis among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 2: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of non-specific lesions of Labia Majora in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant for the diagnosis of the vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of Labia Majora among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 3: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of non-specific lesions of the Perineum in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant for the diagnosis of the vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of the Perineum among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 4: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of erythema of Mons Pubis in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant for the diagnosis of the vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of erythema of Mons Pubis among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 5: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of erythema of Labia Majora in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant for the diagnosis of the vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of erythema of Labia Majora among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 6: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of erythema of the Perineum in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant for the diagnosis of the vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of erythema of the Perineum among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 7: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of excoriations of Mons Pubis in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant for the diagnosis of the vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of excoriations of Mons Pubis among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 8: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of excoriations of Labia Majora in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant for the diagnosis of the vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of excoriations of Labia Majora among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 9: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of excoriations of the Perineum in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant for the diagnosis of the vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of excoriations of the Perineum among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 10: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of rhagades of Mons Pubis in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant for the diagnosis of the vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of rhagades of Mons Pubis among patients from different groups?; p = 0.0016, Chi-squared
Statistical Analysis 11: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of rhagades of Labia Majora in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant for the diagnosis of the vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of rhagades of Labia Majora among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 12: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of rhagades of the Perineum in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant for the diagnosis of the vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of rhagades of the Perineum among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 13: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of non-specific lesions of Mons Pubis versus non-specific lesions of Labia Majora in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of Mons Pubis versus non-specific lesions of Labia Majora in patients with vulvar dermatosis?; p = 0.0014, t-test proportion
Statistical Analysis 14: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of non-specific lesions of Mons Pubis versus non-specific lesions of the Perineum in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of Mons Pubis versus non-specific lesions of the Perineum in patients with vulvar dermatosis?; p = 0.0000, t-test proportion
Statistical Analysis 15: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of non-specific lesion of Labia Majora versus non-specific lesions of the Perineum in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of Labia Majora versus non-specific lesions of the Perineum in patients with vulvar dermatosis?; p = 0.0414, t-test proportion
Statistical Analysis 16: Comparison: Vulvodynia; Parameter: The difference in the incidence of non-specific lesions of Mons Pubis versus non-specific lesions of Labia Majora in patients with vulvodynia. The diagnosis of vulvodynia was based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection, Q-Tip) following Friedrich's criteria. Vulvoscopic lesions were not relevant to the diagnosis of vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of Mons Pubis versus non-specific lesions of Labia Majora in patients with vulvodynia?; p = 0.0898, t-test proportion
Statistical Analysis 17: Comparison: Vulvodynia; Parameter: The difference in the incidence of non-specific lesions of Mons Pubis versus non-specific lesions of the Perineum in patients with vulvodynia. The diagnosis of vulvodynia was based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection, Q-Tip) following Friedrich's criteria. Vulvoscopic lesions were not relevant to the diagnosis of vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of Mons Pubis versus non-specific lesions of the Perineum in patients with vulvodynia?; p = 0.0008, t-test proportion
Statistical Analysis 18: Comparison: Vulvodynia; Parameter: The difference in the incidence of non-specific lesions of Labia Majora versus non-specific lesions of the Perineum in patients with vulvodynia. The diagnosis of vulvodynia was based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection, Q-Tip) following Friedrich's criteria. Vulvoscopic lesions were not relevant to the diagnosis of vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of Labia Majora versus non-specific lesions of the Perineum in patients with vulvodynia?; p = 0.0587, t-test proportion
Statistical Analysis 19: Comparison: Impaired Vulvar Skin; Parameter: The difference in the incidence of non-specific lesions of Mons Pubis versus non-specific lesions of Labia Majora in patients with impaired vulvar skin; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of Mons Pubis versus non-specific lesions of Labia Majora in patients with impaired vulvar skin?; p = 1.0000, t-test proportion
Statistical Analysis 20: Comparison: Impaired Vulvar Skin; Parameter: The difference in the incidence of non-specific lesions of Mons Pubis versus non-specific lesions of the Perineum in patients with impaired vulvar skin; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of Mons Pubis versus non-specific lesions of the Perineum in patients with impaired vulvar skin?; p = 0.1352, t-test proportion
Statistical Analysis 21: Comparison: Impaired Vulvar Skin; Parameter: The difference in the incidence of non-specific lesion of Labia Majora versus non-specific lesions of the Perineum in patients with impaired vulvar skin; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of Labia Majora versus non-specific lesions of the Perineum in patients with impaired vulvar skin?; p = 0.1352, t-test proportion
Statistical Analysis 22: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of specific lesions of Mons Pubis versus specific lesions of Labia Majora in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of specific lesions of Mons Pubis versus specific lesions of Labia Majora in patients with vulvar dermatosis?; p = 0.0002, t-test proportion
Statistical Analysis 23: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of specific lesions of Mons Pubis versus specific lesions of the Perineum in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of specific lesions of Mons Pubis versus specific lesions of the Perineum in patients with vulvar dermatosis?; p = 0.0000, t-test proportion
Statistical Analysis 24: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of specific lesions of Labia Majora versus specific lesions of the Perineum in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of specific lesions of Labia Majora versus specific lesions of the Perineum in patients with vulvar dermatosis?; p = 0.0854, t-test proportion

27. Secondary Outcome: Distribution of Non-Specific and Specific Lesions of the Middle Vulvar Ring According to the "Three Rings Vulvoscopy"
Description: The table shows the distribution of non-specific and specific lesions of the vulva in relation to the individual structures of the Middle vulvar ring according to the "Three Rings Vulvoscopy." The "MIDDLE vulvar ring" includes the anterior commissure with the prepuce of the clitoris, interlabial sulci, labia minora, and the posterior commissure.
  "Non-Specific Lesions" include non-specific erythema, punctuations, papillae, paleness and smoothness, fissures or sores in the absence of infection and pre/malignancy in any part of the vulva.
  "Specific Lesions" comprise eczematous inflammation with thickened, excoriated skin within chronic lichen simplex; hypopigmented or white lesions, fusion or resorption of the labia minora and clitoral hood, loss of vulvar architecture and sclerotic changes in lichen sclerosis; white reticular pattern to extensive erosion with agglutination or resorption of the labia within lichen planus and psoriatic erythematous papules with silver, scaly plaques.
Time Frame: Three Rings Vulvoscopy, up to 45 minutes for each participant.
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Vulva | Impaired Vulvar Skin | Vulvodynia | Vulvar Dermatosis
Number analyzed (Participants) | 82 | 82 | 82 | 82
Participants
  Non-specific Lesions of the Anterior Commissure | 1 | 7 | 9 | 30
  Non-specific Lesions of Interlabial Sulci | 1 | 32 | 41 | 46
  Non-specific Lesions of Labia Minora | 10 | 25 | 48 | 42
  Non-specific Lesions of the Posterior Commissure | 23 | 56 | 76 | 56
  Erythema of the Anterior Commissure | 0 | 3 | 3 | 8
  Erythema of Interlabial Sulci | 0 | 28 | 35 | 25
  Erythema of Labia Minora | 10 | 9 | 25 | 21
  Erythema of the Posterior Commissure | 23 | 23 | 48 | 33
  Fissures of the Anterior Commissure | 0 | 0 | 0 | 6
  Fissures of Interlabial Sulci | 0 | 0 | 0 | 12
  Fissures of Labia Minora | 0 | 0 | 0 | 5
  Fissures of the Posterior Commissure | 0 | 0 | 2 | 20
  Smoothness of the Anterior Commissure | 0 | 0 | 0 | 9
  Smoothness of Interlabial Sulci | 0 | 1 | 0 | 11
  Smoothness of Labia Minora | 0 | 1 | 0 | 6
  Smoothness of the Posterior Commissure | 0 | 2 | 0 | 5
  Specific Lesions of the Anterior Commissure | 0 | 0 | 0 | 58
  Specific Lesions of Interlabial Sulci | 0 | 0 | 0 | 64
  Specific Lesions of Labia Minora | 0 | 0 | 0 | 60
  Specific Lesions of the Posterior Commissure | 0 | 0 | 0 | 61
Statistical Analysis 1: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of non-specific lesions of the Anterior Commissure in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of the Anterior Commissure among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 2: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of non-specific lesions of Interlabial Sulci in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of Interlabial Sulci among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 3: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of non-specific lesions of Labia Minora in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of Labia Minora among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 4: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of non-specific lesions of the Posterior Commissure in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy.". Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of the Posterior Commissure among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 5: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of erythema of the Anterior Commissure in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q- Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of erythema of the Anterior Commissure among patients from different groups?; p = 0.0199, Chi-squared
Statistical Analysis 6: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of erythema of Interlabial Sulci in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q- Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of erythema of Interlabial Sulci among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 7: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of erythema of Labia Minora in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q- Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of erythema of Labia Minora among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 8: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of erythema of the Posterior Commissure in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q- Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of erythema of the Posterior Commissure among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 9: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of fissures of Interlabial Sulci in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q- Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of fissures of Interlabial Sulci among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 10: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of fissures of the Posterior Commissure in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q- Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of fissures of the Posterior Commissure among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 11: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of smoothness of the Anterior Commissure in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of smoothness of the Anterior Commissure among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 12: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of smoothness of Interlabial Sulci in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q- Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of smoothness of Interlabial Sulci among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 13: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The frequency of smoothness of Labia Minora in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q- Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of vulvodynia; Test type: Superiority — Question: Is there a difference in the frequency of smoothness of Labia Minora among patients from different groups?; p = 0.0024, Chi-squared
Statistical Analysis 14: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of smoothness of the Posterior Commissure in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q- Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of smoothness of the Posterior Commissure among patients from different groups?; p = 0.0205, Chi-squared
Statistical Analysis 15: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of non-specific lesions of the Anterior Commissure versus non-specific lesions of Interlabial Sulci in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of the Anterior Commissure versus non-specific lesions of Interlabial Sulci in patients with vulvar dermatosis?; p = 0.0158, t-test proportion
Statistical Analysis 16: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of non-specific lesions of the Anterior Commissure versus non-specific lesions of the Posterior Commissure in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of the Anterior Commissure versus non-specific lesions of the Posterior Commissure in patients with vulvar dermatosis?; p = 0.0001, t-test proportion
Statistical Analysis 17: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of non-specific lesions of Labia Minora versus non-specific lesions of the Posterior Commissure in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of Labia Minora versus non-specific lesions of the Posterior Commissure in patients with vulvar dermatosis?; p = 0.0280, t-test proportion
Statistical Analysis 18: Comparison: Vulvodynia; Parameter: The difference in the incidence of non-specific lesions of the Anterior Commissure versus non-specific lesions of Interlabial Sulci in patients with vulvodynia. The diagnosis of vulvodynia was based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection, Q-Tip) following Friedrich's criteria. Vulvoscopic lesions were not relevant to the diagnosis of vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of the Anterior Commissure versus non-specific lesions of Interlabial Sulci in patients with vulvodynia?; p = 0.0000, t-test proportion
Statistical Analysis 19: Comparison: Vulvodynia; Parameter: The difference in the incidence of non-specific lesions of the Anterior Commissure versus non-specific lesions of Labia Minora in patients with vulvodynia. The diagnosis of vulvodynia was based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection, Q-Tip) following Friedrich's criteria. Vulvoscopic lesions were not relevant to the diagnosis of vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of the Anterior Commissure versus non-specific lesions of Labia Minora in patients with vulvodynia?; p = 0.0000, t-test proportion
Statistical Analysis 20: Comparison: Vulvodynia; Parameter: The difference in the incidence of non-specific lesions of the Anterior Commissure versus non-specific lesions of the Posterior Commissure in patients with vulvodynia. The diagnosis of vulvodynia was based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection, Q-Tip) following Friedrich's criteria. Vulvoscopic lesions were not relevant to the diagnosis of vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of the Anterior Commissure versus non-specific lesions of the Posterior Commissure in patients with vulvodynia?; p = 0.0000, t-test proportion
Statistical Analysis 21: Comparison: Vulvodynia; Parameter: The difference in the incidence of non-specific lesions of Interlabial Sulci versus non-specific lesions of the Posterior Commissure in patients with vulvodynia. The diagnosis of vulvodynia was based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection, Q-Tip) following Friedrich's criteria. Vulvoscopic lesions were not relevant to the diagnosis of vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of Interlabial Sulci versus non-specific lesions of the Posterior Commissure in patients with vulvodynia?; p = 0.0000, t-test proportion
Statistical Analysis 22: Comparison: Vulvodynia; Parameter: The difference in the incidence of non-specific lesions of Labia Minora versus non-specific lesions of the Posterior Commissure in patients with vulvodynia. The diagnosis of vulvodynia was based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection, Q-Tip) following Friedrich's criteria. Vulvoscopic lesions were not relevant to the diagnosis of vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of Labia Minora versus non-specific lesions of the Posterior Commissure in patients with vulvodynia?; p = 0.0000, t-test proportion
Statistical Analysis 23: Comparison: Impaired Vulvar Skin; Parameter: The difference in the incidence of non-specific lesions of the Anterior Commissure versus non-specific lesions of Interlabial Sulci in patients with impaired vulvar skin; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of the Anterior Commissure versus non-specific lesions of Interlabial Sulci in patients with impaired vulvar skin?; p = 0.0000, t-test proportion
Statistical Analysis 24: Comparison: Impaired Vulvar Skin; Parameter: The difference in the incidence of non-specific lesions of the Anterior Commissure versus non-specific lesions of Labia Minora in patients with impaired vulvar skin; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of the Anterior Commissure versus non-specific lesions of Labia Minora in patients with impaired vulvar skin?; p = 0.0006, t-test proportion
Statistical Analysis 25: Comparison: Impaired Vulvar Skin; Parameter: The difference in the incidence of non-specific lesions of the Anterior Commissure versus non-specific lesions of the Posterior Commissure in patients with impaired vulvar skin; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of the Anterior Commissure versus non-specific lesions of the Posterior Commissure in patients with impaired vulvar skin?; p = 0.0000, t-test proportion
Statistical Analysis 26: Comparison: Impaired Vulvar Skin; Parameter: The difference in the incidence of non-specific lesions of Interlabial Sulci versus non-specific lesions of the Posterior Commissure in patients with impaired vulvar skin; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of Interlabial Sulci versus non-specific lesions of the Posterior Commissure in patients with impaired vulvar skin?; p = 0.0003, t-test proportion
Statistical Analysis 27: Comparison: Impaired Vulvar Skin; Parameter: The difference in the incidence of non-specific lesions of Labia Minora versus non-specific lesions of the Posterior Commissure in patients with impaired vulvar skin; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of Labia Minora versus non-specific lesions of the Posterior Commissure in patients with impaired vulvar skin?; p = 0.0000, t-test proportion
Statistical Analysis 28: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of specific lesions of the Anterior Commissure versus specific lesions of Interlabial Sulci in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of specific lesion of the Anterior Commissure versus specific lesions of Interlabial Sulci in patients with vulvar dermatosis?; p = 0.3053, t-test proportion
Statistical Analysis 29: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of specific lesions of the Anterior Commissure versus specific lesions of Labia Minora in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of specific lesion of the Anterior Commissure versus specific lesions of Labia Minora in patients with vulvar dermatosis?; p = 0.7758, t-test proportion
Statistical Analysis 30: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of specific lesions of the Anterior Commissure versus specific lesions of the Posterior Commissure in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of specific lesion of the Anterior Commissure versus specific lesions of the Posterior Commissure in patients with vulvar dermatosis?; p = 0.6676, t-test proportion
Statistical Analysis 31: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of specific lesions of Interlabial Sulci versus specific lesions of Labia Minora in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of specific lesion of Interlabial Sulci versus specific lesions of Labia Minora in patients with vulvar dermatosis?; p = 0.4577, t-test proportion
Statistical Analysis 32: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of specific lesions of Interlabial Sulci versus specific lesions of the Posterior Commissure in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of specific lesion of Interlabial Sulci versus specific lesions of the Posterior Commissure in patients with vulvar dermatosis?; p = 0.1681, t-test proportion
Statistical Analysis 33: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of specific lesions of Labia Minora versus specific lesions of the Posterior Commissure in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of specific lesion of Labia Minora versus specific lesions of the Posterior Commissure in patients with vulvar dermatosis?; p = 0.8848, t-test proportion

28. Secondary Outcome: Distribution of Non-Specific and Specific Lesions of the Inner Vulvar Ring According to the "Three Rings Vulvoscopy"
Description: The table shows the distribution of non-specific and specific lesions of the vulva in relation to the individual structures of the Inner vulvar ring according to the "Three Rings Vulvoscopy." The "INNER vulvar ring" includes clitoris, Hart's line, urethral sulcus, urethral meatus, hymenal remnants, Bartholin's gland opening, and the vestibule.
  "Non-Specific Lesions" include non-specific erythema, punctuations, papillae, paleness and smoothness, fissures or sores in the absence of infection and pre/malignancy in any part of the vulva.
  "Specific Lesions" comprise eczematous inflammation with thickened, excoriated skin within chronic lichen simplex; hypopigmented or white lesions, fusion or resorption of the labia minora and clitoral hood, loss of vulvar architecture and sclerotic changes in lichen sclerosis; white reticular pattern to extensive erosion with agglutination or resorption of the labia within lichen planus and psoriatic erythematous papules with silver, scaly plaques.
Time Frame: Three Rings Vulvoscopy, up to 45 minutes for each participant.
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Vulva | Impaired Vulvar Skin | Vulvodynia | Vulvar Dermatosis
Number analyzed (Participants) | 82 | 82 | 82 | 82
Participants
  Non-specific Lesions of the clitoris | 8 | 43 | 76 | 34
  Non-specific Lesions of Hart's line | 21 | 68 | 81 | 55
  Non-specific Lesions of the Urethral Sulcus | 16 | 69 | 81 | 55
  Non-specific Lesions of the Urethral Meatus | 7 | 45 | 72 | 43
  Non-specific Lesions of Hymenal remnants | 6 | 37 | 69 | 30
  Non-specific Lesions of Bartholin's gland opening | 8 | 49 | 77 | 33
  Non-specific Lesions of the Vestibule | 22 | 59 | 80 | 61
  Erythema of the clitoris | 0 | 11 | 29 | 5
  Erythema of Hart's line | 11 | 52 | 69 | 43
  Erythema of the Urethral Sulcus | 0 | 26 | 43 | 16
  Erythema of the Urethral Meatus | 1 | 6 | 18 | 20
  Erythema of Hymenal remnants | 5 | 7 | 17 | 16
  Erythema of Bartholin's gland opening | 7 | 30 | 49 | 24
  Erythema of the Vestibule | 9 | 29 | 45 | 41
  Smoothness of the clitoris | 0 | 5 | 3 | 11
  Smootness of Hart's line | 1 | 1 | 1 | 5
  Smoothness of the Urethral Sulcus | 12 | 22 | 37 | 26
  Smoothness of the Urethral Meatus | 2 | 2 | 1 | 6
  Smoothness of Hymenal remnants | 1 | 1 | 0 | 5
  Smoothness of Bartholin's gland opening | 1 | 1 | 0 | 5
  Smoothness of the Vestibule | 3 | 3 | 4 | 6
  Ischemia of the clitoris | 0 | 11 | 14 | 8
  Ischemia of Hart's line | 1 | 1 | 4 | 1
  Ischemia of the Urethral Sulcus | 4 | 31 | 24 | 21
  Ischemia of the Urethral Meatus | 2 | 3 | 9 | 2
  Ischemia of Hymenal remnants | 0 | 0 | 4 | 2
  Ischemia of Bartholin's gland opening | 0 | 0 | 3 | 2
  Ischemia of the Vestibule | 6 | 7 | 14 | 8
  Punctuation of the clitoris | 0 | 0 | 0 | 0
  Punctuation of Hart's line | 0 | 36 | 43 | 12
  Punctuation of the Urethral Sulcus | 0 | 3 | 2 | 0
  Punctuation of the Urethral Meatus | 0 | 1 | 4 | 4
  Punctuation of Hymenal remnants | 0 | 2 | 5 | 3
  Punctuation of Bartholin's gland opening | 0 | 1 | 4 | 4
  Punctuation of the Vestibule | 0 | 8 | 10 | 8
  Papillae of Hart's line | 8 | 17 | 18 | 2
  Papillae of the Urethral Sulcus | 0 | 0 | 2 | 0
  Papillae of the Vestibule | 4 | 12 | 10 | 1
  Specific Lesions of the clitoris | 0 | 0 | 0 | 43
  Specific Lesions of Hart's line | 0 | 0 | 0 | 28
  Specific Lesions of the Urethral Sulcus | 0 | 0 | 0 | 36
  Specific Lesions of the Urethral Meatus | 0 | 0 | 0 | 29
  Specific Lesions of Hymenal remnants | 0 | 0 | 0 | 27
  Specific Lesions of Bartholin's gland opening | 0 | 0 | 0 | 25
  Specific Lesions of the Vestibule | 0 | 0 | 0 | 29
Statistical Analysis 1: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of non-specific lesions of the Clitoris in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant for the diagnosis of the vulvodynia; Test type: Equivalence — Question: Is there a difference in the incidence of non-specific lesions of the Clitoris among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 2: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of non-specific lesions of Hart's Line in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant for the diagnosis of the vulvodynia; Test type: Equivalence — Question: Is there a difference in the incidence of non-specific lesions of Hart's Line among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 3: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of non-specific lesions of the Urethral Sulcus in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of the vulvodynia; Test type: Equivalence — Question: Is there a difference in the incidence of non-specific lesions of the Urethral Sulcus among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 4: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of non-specific lesions of the Urethral meatus in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of the vulvodynia; Test type: Equivalence — Question: Is there a difference in the incidence of non-specific lesions of the Urethral Meatus among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 5: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of non-specific lesions of Hymenal Remnants in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of the vulvodynia; Test type: Equivalence — Question: Is there a difference in the incidence of non-specific lesions of Hymenal Remnants among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 6: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of non-specific lesions of Bartholin's Gland Opening in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of the vulvodynia; Test type: Equivalence — Question: Is there a difference in the incidence of non-specific lesions of Bartholin's Gland Opening among the patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 7: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of non-specific lesions of the Vestibule in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of the vulvodynia; Test type: Equivalence — Question: Is there a difference in the incidence of non-specific lesions of the Vestibule among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 8: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of erythema of the Clitoris in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of the vulvodynia; Test type: Equivalence — Question: Is there a difference in the incidence of erythema of the Clitoris among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 9: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of erythema of Hart's Line in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of the vulvodynia; Test type: Equivalence — Question: Is there a difference in the incidence of erythema of Hart's Line among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 10: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of erythema of the Urethral Sulcus in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of the vulvodynia; Test type: Equivalence — Question: Is there a difference in the incidence of erythema of the Urethral Sulcus among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 11: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of erythema of the Urethral Meatus in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of the vulvodynia; Test type: Equivalence — Question: Is there a difference in the incidence of erythema of the Urethral Meatus among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 12: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of erythema of Hymenal Remnants in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of the vulvodynia; Test type: Equivalence — Question: Is there a difference in the incidence of erythema of Hymenal Remnants among patients from different groups?; p = 0.0001, Chi-squared
Statistical Analysis 13: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of erythema of Bartholin's Gland Opening in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of the vulvodynia; Test type: Equivalence — Question: Is there a difference in the incidence of erythema of Bartholin's Gland Opening among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 14: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of erythema of the Vestibule in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of the vulvodynia; Test type: Equivalence — Question: Is there a difference in the incidence of erythema of the Vestibule among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 15: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of smoothness of the Clitoris in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of the vulvodynia; Test type: Equivalence — Question: Is there a difference in the incidence of smoothness of the Clitoris among patients from different groups?; p = 0.0023, Chi-squared
Statistical Analysis 16: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of smoothness of the Urethral Sulcus in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of the vulvodynia; Test type: Equivalence — Question: Is there a difference in the incidence of smoothness of the Urethral Sulcus among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 17: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of smoothness of Urethral Meatus in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of the vulvodynia; Test type: Equivalence — Question: Is there a difference in the incidence of smoothness of the Urethral Meatus among patients from different groups?; p = 0.0235, Chi-squared
Statistical Analysis 18: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of ischemia of the Clitoris in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of the vulvodynia; Test type: Equivalence — Question: Is there a difference in the incidence of ischemia of the Clitoris among patients from different groups?; p = 0.0021, Chi-squared
Statistical Analysis 19: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of ischemia of the Urethral Sulcus in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of the vulvodynia; Test type: Equivalence — Question: Is there a difference in the incidence of ischemia of the Urethral Sulcus among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 20: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of ischemia of the Urethral Meatus in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of the vulvodynia; Test type: Equivalence — Question: Is there a difference in the incidence of ischemia of the Urethral Meatus among patients from different groups?; p = 0.0038, Chi-squared
Statistical Analysis 21: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of ischemia of the Vestibule in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of the vulvodynia; Test type: Equivalence — Question: Is there a difference in the incidence of ischemia of the Vestibule among patients from different groups?; p = 0.0019, Chi-squared
Statistical Analysis 22: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of punctuation of Hart's Line in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of the vulvodynia; Test type: Equivalence — Question: Is there a difference in the incidence of punctuation of Hart's Line among patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 23: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of punctuation of the Vestibule in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy.". Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of the vulvodynia; Test type: Equivalence — Question: Is there a difference in the incidence of punctuation of the Vestibule among patients from different groups?; p = 0.0198, Chi-squared
Statistical Analysis 24: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of papillae of Hart's Line in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of the vulvodynia; Test type: Equivalence — Question: Is there a difference in the incidence of papillae of Hart's Line among patients from different groups?; p = 0.0004, Chi-squared
Statistical Analysis 25: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The incidence of papillae of the Vestibule in patients classified into four groups based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection and Q-Tip), which were examined by the "Three Rings Vulvoscopy." Vulvoscopic lesions in patients with vulvodynia were not relevant to the diagnosis of the vulvodynia; Test type: Equivalence — Question: Is there a difference in the incidence of papillae of the Vestibule among patients from different groups?; p = 0.0053, Chi-squared
Statistical Analysis 26: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of non-specific lesions of the Clitoris versus non-specific lesions of Hart's Line in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of the Clitoris versus non-specific lesions of Hart's Line in patients with vulvar dermatosis?; p = 0.0010, t-test proportion
Statistical Analysis 27: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of non-specific lesions of the Clitoris versus non-specific lesions of the Urethral Sulcus in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of the Clitoris versus non-specific lesions of the Urethral Sulcus in patients with vulvar dermatosis?; p = 0.0010, t-test proportion
Statistical Analysis 28: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of non-specific lesions of the Clitoris versus non-specific lesions of the Vestibule in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of the Clitoris versus non-specific lesions of the Vestibule in patients with vulvar dermatosis?; p = 0.0000, t-test proportion
Statistical Analysis 29: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of non-specific lesions of Hart's Line versus non-specific lesions of Hymenal Remnants in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of Hart's Line versus non-specific lesions of Hymenal Remnants in patients with vulvar dermatosis?; p = 0.0208, t-test proportion
Statistical Analysis 30: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of non-specific lesions of Hart's Line versus non-specific lesions of Bartholin's Gland Opening in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of Hart's Line versus non-specific lesions of Bartholin's Gland Opening in patients with vulvar dermatosis?; p = 0.0007, t-test proportion
Statistical Analysis 31: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of non-specific lesions of the Urethral Sulcus versus non-specific lesions of Hymenal Remnants in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of the Urethral Sulcus versus non-specific lesions of Hymenal Remnants in patients with vulvar dermatosis?; p = 0.0208, t-test proportion
Statistical Analysis 32: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of non-specific lesions of the Urethral Sulcus versus non-specific lesions of Bartholin's Gland Opening in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of the Urethral Sulcus versus non-specific lesions of Bartholin's Gland Opening in patients with vulvar dermatosis?; p = 0.0007, t-test proportion
Statistical Analysis 33: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of non-specific lesions of the Urethral Meatus versus non-specific lesions of the Vestibule in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of the Urethral Meatus versus non-specific lesions of the Vestibule in patients with vulvar dermatosis?; p = 0.0040, t-test proportion
Statistical Analysis 34: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of non-specific lesions of Hymenal Remnants versus non-specific lesions of the Vestibule in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of Hymenal Remnants versus non-specific lesions of the Vestibule in patients with vulvar dermatosis?; p = 0.0012, t-test proportion
Statistical Analysis 35: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of non-specific lesions of Bartholin's Gland Opening versus non-specific lesions of the Vestibule in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of Bartholin's Gland Opening versus non-specific lesions of the Vestibule in patients with vulvar dermatosis?; p = 0.0000, t-test proportion
Statistical Analysis 36: Comparison: Vulvodynia; Parameter: The difference in the incidence of non-specific lesions of Hart's Line versus non-specific lesions of the Urethral Meatus in patients with vulvodynia. The diagnosis of vulvodynia was based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection, Q-Tip) following Friedrich's criteria. Vulvoscopic lesions were not relevant to the diagnosis of vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of Hart's Line versus non-specific lesions of the Urethral Meatus in patients with vulvodynia?; p = 0.0048, t-test proportion
Statistical Analysis 37: Comparison: Vulvodynia; Parameter: The difference in the incidence of non-specific lesions of Hart's Line versus non-specific lesions of Hymenal Remnants in patients with vulvodynia. The diagnosis of vulvodynia was based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection, Q-Tip) following Friedrich's criteria. Vulvoscopic lesions were not relevant to the diagnosis of vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of Hart's Line versus non-specific lesions of Hymenal Remnants in patients with vulvodynia?; p = 0.0007, t-test proportion
Statistical Analysis 38: Comparison: Vulvodynia; Parameter: The difference in the incidence of non-specific lesions of the Urethral Sulcus versus non-specific lesions of the Urethral Meatus in patients with vulvodynia. The diagnosis of vulvodynia was based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection, Q-Tip) following Friedrich's criteria. Vulvoscopic lesions were not relevant to the diagnosis of vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of the Urethral Sulcus versus non-specific lesions of the Urethral Meatus in patients with vulvodynia?; p = 0.0048, t-test proportion
Statistical Analysis 39: Comparison: Vulvodynia; Parameter: The difference in the incidence of non-specific lesions of the Urethral Sulcus versus non-specific lesions of Hymenal Remnants in patients with vulvodynia. The diagnosis of vulvodynia was based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection, Q-Tip) following Friedrich's criteria. Vulvoscopic lesions were not relevant to the diagnosis of vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of the Urethral Sulcus versus non-specific lesions of Hymenal Remnants in patients with vulvodynia?; p = 0.0007, t-test proportion
Statistical Analysis 40: Comparison: Vulvodynia; Parameter: The difference in the incidence of non-specific lesions of the Urethral Meatus versus non-specific lesions of the Vestibule in patients with vulvodynia. The diagnosis of vulvodynia was based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection, Q-Tip) following Friedrich's criteria. Vulvoscopic lesions were not relevant to the diagnosis of vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of the Urethral Meatus versus non-specific lesions of the Vestibule in patients with vulvodynia?; p = 0.0131, t-test proportion
Statistical Analysis 41: Comparison: Vulvodynia; Parameter: The difference in the incidence of non-specific lesions of Hymenal Remnants versus non-specific lesions of Bartholin's Gland Opening in patients with vulvodynia. The diagnosis of vulvodynia was based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection, Q-Tip) following Friedrich's criteria. Vulvoscopic lesions were not relevant to the diagnosis of vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of Hymenal Remnants versus non-specific lesions of Bartholin's Gland Opening in patients with vulvodynia?; p = 0.0423, t-test proportion
Statistical Analysis 42: Comparison: Vulvodynia; Parameter: The difference in the incidence of non-specific lesions of Hymenal Remnants versus non-specific lesions of the Vestibule in patients with vulvodynia. The diagnosis of vulvodynia was based on anamnestic data (ISSVD Questionnaire) and clinical examination (Inspection, Q-Tip) following Friedrich's criteria. Vulvoscopic lesions were not relevant to the diagnosis of vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of Hymenal Remnants versus non-specific lesions of the Vestibule in patients with vulvodynia?; p = 0.0021, t-test proportion
Statistical Analysis 43: Comparison: Impaired Vulvar Skin; Parameter: The difference in the incidence of non-specific lesions of the Clitoris versus non-specific lesions of Hart's Line in patients with impaired vulvar skin; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of the Clitoris versus non-specific lesions of Hart's Line in patients with impaired vulvar skin?; p = 0.0000, t-test proportion
Statistical Analysis 44: Comparison: Impaired Vulvar Skin; Parameter: The difference in the incidence of non-specific lesions of the Clitoris versus non-specific lesions of the Urethral Sulcus in patients with impaired vulvar skin; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of the Clitoris versus non-specific lesions of the Urethral Sulcus in patients with impaired vulvar skin?; p = 0.0000, t-test proportion
Statistical Analysis 45: Comparison: Impaired Vulvar Skin; Parameter: The difference in the incidence of non-specific lesions of the Clitoris versus non-specific lesions of the Vestibule in patients with impaired vulvar skin; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of the Clitoris versus non-specific lesions of the Vestibule in patients with impaired vulvar skin?; p = 0.0091, t-test proportion
Statistical Analysis 46: Comparison: Impaired Vulvar Skin; Parameter: The difference in the incidence of non-specific lesions of Hart's Line versus non-specific lesions of the Urethral Meatus in patients with impaired vulvar skin; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of Hart's Line versus non-specific lesions of the Urethral Meatus in patients with impaired vulvar skin?; p = 0.0002, t-test proportion
Statistical Analysis 47: Comparison: Impaired Vulvar Skin; Parameter: The difference in the incidence of non-specific lesions of Hart's Line versus non-specific lesions of Hymenal Remnants in patients with impaired vulvar skin; Test type: Equivalence — Question: Is there a difference in the incidence of non-specific lesions of Hart's Line versus non-specific lesions of Hymenal Remnants in patients with impaired vulvar skin?; p = 0.0000, t-test proportion
Statistical Analysis 48: Comparison: Impaired Vulvar Skin; Parameter: The difference in the incidence of non-specific lesions of Hart's Line versus non-specific lesions of Bartholin's Gland Opening in patients with impaired vulvar skin; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of Hart's Line versus non-specific lesions of Bartholin's Gland Opening in patients with impaired vulvar skin?; p = 0.0013, t-test proportion
Statistical Analysis 49: Comparison: Impaired Vulvar Skin; Parameter: The difference in the incidence of non-specific lesions of the Urethral Sulcus versus non-specific lesions of the Urethral Meatus in patients with impaired vulvar skin; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of the Urethral Sulcus versus non-specific lesions of the Urethral Meatus in patients with impaired vulvar skin?; p = 0.0001, t-test proportion
Statistical Analysis 50: Comparison: Impaired Vulvar Skin; Parameter: The difference in the incidence of non-specific lesions of the Urethral Sulcus versus non-specific lesions of Hymenal Remnants in patients with impaired vulvar skin; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of the Urethral Sulcus versus non-specific lesions of Hymenal Remnants in patients with impaired vulvar skin?; p = 0.0000, t-test proportion
Statistical Analysis 51: Comparison: Impaired Vulvar Skin; Parameter: The difference in the incidence of non-specific lesions of the Urethral Sulcus versus non-specific lesions of Bartholin's Gland Opening in patients with impaired vulvar skin; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of the Urethral Sulcus versus non-specific lesions of Bartholin's Gland Opening in patients with impaired vulvar skin?; p = 0.0008, t-test proportion
Statistical Analysis 52: Comparison: Impaired Vulvar Skin; Parameter: The difference in the incidence of non-specific lesions of the Urethral Meatus versus non-specific lesions of the Vestibule in patients with impaired vulvar skin; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of the Urethral Meatus versus non-specific lesions of the Vestibule in patients with impaired vulvar skin?; p = 0.0251, t-test proportion
Statistical Analysis 53: Comparison: Impaired Vulvar Skin; Parameter: The difference in the incidence of non-specific lesions of Hymenal Remnants versus non-specific lesions of the Vestibule in patients with impaired vulvar skin; Test type: Superiority — Question: Is there a difference in the incidence of non-specific lesions of Hymenal Remnants versus non-specific lesions of the Vestibule in patients with impaired vulvar skin?; p = 0.0006, t-test proportion
Statistical Analysis 54: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of specific lesions of the Clitoris versus specific lesions of Hart's Line in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of specific lesions of the Clitoris versus specific lesions of Hart's Line in patients with vulvar dermatosis?; p = 0.0211, t-test proportion
Statistical Analysis 55: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of specific lesions of the Clitoris versus specific lesions of the Urethral Sulcus in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of specific lesions of the Clitoris versus specific lesions of the Urethral Sulcus in patients with vulvar dermatosis?; p = 0.3067, t-test proportion
Statistical Analysis 56: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of specific lesions of the Clitoris versus specific lesions of the Urethral Meatus in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of specific lesions of the Clitoris versus specific lesions of the Urethral Meatus in patients with vulvar dermatosis?; p = 0.0295, t-test proportion
Statistical Analysis 57: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of specific lesions of the Clitoris versus specific lesions of Hymenal Remnants in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of specific lesions of the Clitoris versus specific lesions of Hymenal Remnants in patients with vulvar dermatosis?; p = 0.0149, t-test proportion
Statistical Analysis 58: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of specific lesions of the Clitoris versus specific lesions of Bartholin's Gland Opening in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of specific lesions of the Clitoris versus specific lesions of Bartholin's Gland Opening in patients with vulvar dermatosis?; p = 0.0007, t-test proportion
Statistical Analysis 59: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of specific lesions of the Clitoris versus specific lesions of the Vestibule in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of specific lesions of the Clitoris versus specific lesions of the Vestibule in patients with vulvar dermatosis?; p = 0.0295, t-test proportion

29. Secondary Outcome: Aceto-Whitening Reaction (AWR) in Relation to the Three Vulvar Rings
Description: The table shows the presence, the quality, and the distribution of the aceto-whitening reaction after 5% acetic acid application (Aceto-Whitening Test), in relation to the three vulvar rings.
  The "OUTER Vulvar Ring" includes vulvar skin, the "MIDDLE Vulvar Ring" encompasses the modified mucosa, and the "INNER Vulvar Ring" is presented with glicogenized mucosa.
  Acetic acid is thought to cause swelling of the epithelial tissue through reversible coagulation or precipitation of the nuclear proteins and cytokeratins.
  Areas of pre-/malignant lesions turn densely white and opaque immediately after application of acetic acid, due to the presence of large numbers of dysplastic cells in the superficial layers of the epithelium.
  The acetowhite appearance is not unique to pre-/malignancy; it is also seen in other conditions with increased nuclear protein. The acetowhite reaction varies in intensity, within and between patients.
Time Frame: Aceto-Whitening Test, up to 10 minutes for each participant.
Population: The Aceto-Whitening test was performed in 328 patients, classified into four groups based on anamnestic data and clinical examination. Localization and type, as well as the velocity of the AWR, were mapped into the "TRIV Form Data." Aceto-Whitening of all structures of the Inner Vulvar Ring was named "Ring sign."
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Vulva | Impaired Vulvar Skin | Vulvodynia | Vulvar Dermatosis
Number analyzed (Participants) | 82 | 82 | 82 | 82
Participants
  Aceto-Whitening Presence | Positive AWR | 38 | 74 | 81 | 57
  Semitransparent AWR: Presence | 38 | 71 | 68 | 53
  Coarse AWR: Presence | 0 | 3 | 13 | 4
  Fast AWR (<30 sec) | 1 | 7 | 12 | 9
  Slow AWR (>60 sec) | 24 | 24 | 21 | 23
  Provoked Erythema | 0 | 2 | 9 | 0
  Sharply bordered AWR | 6 | 23 | 40 | 21
  AWR of Outer Vulvar Ring | 0 | 4 | 12 | 37
  AWR of Middle Vulvar Ring | 23 | 61 | 75 | 48
  AWR of Inner Vulvar Ring | 27 | 64 | 79 | 32
  Ring Sign | 6 | 31 | 67 | 9
Statistical Analysis 1: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of aceto-whitening between patients from different groups, with positive AWR; Test type: Equivalence — Question: Is there a difference in the incidence of aceto-whitening between patients from different groups, with positive AWR?; p = 0.0000, Chi-squared
Statistical Analysis 2: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of coarse AWR between patients from different groups and positive AWR; Test type: Equivalence — Question: Is there a difference in the incidence of coarse AWR between patients from different groups and positive AWR?; p = 0.0071, Chi-squared
Statistical Analysis 3: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of slow AWR occurrence between patients from different groups and positive AWR; Test type: Equivalence — Question: Is there a difference in the incidence of slow AWR between patients from different groups and positive AWR?; p = 0.0010, Chi-squared
Statistical Analysis 4: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of provoked erythema among patients from different groups and positive AWR; Test type: Equivalence — Question: Is there a difference in the incidence of provoked erythema among patients from different groups and positive AWR?; p = 0.0036, Chi-squared
Statistical Analysis 5: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of sharply bordered AWR between patients from different groups and positive AWR; Test type: Equivalence — Question: Is there a difference in the incidence of sharply bordered AWR between patients from different groups and positive AWR?; p = 0.0032, Chi-squared
Statistical Analysis 6: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of aceto-whitening of Outer Vulvar Ring between the patients from different groups and positive AWR; Test type: Equivalence — Question: Is there a difference in the incidence of aceto-whitening of Outer Vulvar Ring between the patients from different groups and positive AWR?; p = 0.0000, Chi-squared
Statistical Analysis 7: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of aceto-whitening of Middle Vulvar Ring between the patients from different groups and positive AWR; Test type: Equivalence — Question: Is there a difference in the incidence of aceto-whitening of Middle Vulvar Ring between the patients from different groups and positive AWR?; p = 0.0000, Chi-squared
Statistical Analysis 8: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of aceto-whitening of Inner Vulvar Ring between the patients from different groups and positive AWR; Test type: Equivalence — Question: Is there a difference in the incidence of aceto-whitening of Inner Vulvar Ring between the patients from different groups and positive AWR?; p = 0.0000, Chi-squared
Statistical Analysis 9: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of "Ring sign", aceto-whitening of all structures of the Inner Vulvar Ring, between the patients from different groups and positive AWR; Test type: Equivalence — Question: Is there a difference in the incidence of "Ring sign" between the patients from different groups and positive AWR?; p = 0.0000, Chi-squared
Statistical Analysis 10: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of aceto-whitening of Outer versus Middle Vulvar Ring in patients with vulvar dermatosis and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Outer versus Middle Vulvar Ring in patients with vulvar dermatosis and positive AWR?; p = 0.0856, t-test proportion
Statistical Analysis 11: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of aceto-whitening of Outer versus Inner Vulvar Ring in patients with vulvar dermatosis and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Outer versus Inner Vulvar Ring in patients with vulvar dermatosis and positive AWR?; p = 0.4290, t-test proportion
Statistical Analysis 12: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of aceto-whitening of Middle versus Inner Vulvar Ring in patients with vulvar dermatosis and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Middle versus Inner Vulvar Ring in patients with vulvar dermatosis and positive AWR?; p = 0.0124, t-test proportion
Statistical Analysis 13: Comparison: Vulvodynia; Parameter: The difference in the incidence of aceto-whitening of Outer versus Middle Vulvar Ring in patients with vulvodynia and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Outer versus Middle Vulvar Ring in patients with vulvodynia and positive AWR?; p = 0.0000, t-test proportion
Statistical Analysis 14: Comparison: Vulvodynia; Parameter: The difference in the incidence of aceto-whitening of Outer versus Inner Vulvar Ring in patients with vulvodynia and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Outer versus Inner Vulvar Ring in patients with vulvodynia and positive AWR?; p = 0.0000, t-test proportion
Statistical Analysis 15: Comparison: Vulvodynia; Parameter: The difference in the incidence of aceto-whitening of Middle versus Inner Vulvar Ring in patients with vulvodynia and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Middle versus Inner Vulvar Ring in patients with vulvodynia and positive AWR?; p = 0.1918, t-test proportion
Statistical Analysis 16: Comparison: Impaired Vulvar Skin; Parameter: The difference in the incidence of aceto-whitening of Outer versus Middle Vulvar Ring in patients with impaired vulvar skin and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Outer versus Middle Vulvar Ring in patients with impaired vulvar skin and positive AWR?; p = 0.0000, t-test proportion
Statistical Analysis 17: Comparison: Impaired Vulvar Skin; Parameter: The difference in the incidence of aceto-whitening of Outer versus Inner Vulvar Ring in patients with impaired vulvar skin and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Outer versus Inner Vulvar Ring in patients with impaired vulvar skin and positive AWR?; p = 0.0000, t-test proportion
Statistical Analysis 18: Comparison: Impaired Vulvar Skin; Parameter: The difference in the incidence of aceto-whitening of Middle versus Inner Vulvar Ring in patients with impaired vulvar skin and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Middle versus Inner Vulvar Ring in patients with impaired vulvar skin and positive AWR?; p = 0.5822, t-test proportion
Statistical Analysis 19: Comparison: Normal Vulva; Parameter: The difference in the incidence of aceto-whitening of Outer versus Middle Vulvar Ring in patients with normal vulva and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Outer versus Middle Vulvar Ring in patients with normal vulva and positive AWR?; p = 0.0000, t-test proportion
Statistical Analysis 20: Comparison: Normal Vulva; Parameter: The difference in the incidence of aceto-whitening of Outer versus Inner Vulvar Ring in patients with normal vulva and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Outer versus Inner Vulvar Ring in patients with normal vulva and positive AWR?; p = 0.0000, t-test proportion
Statistical Analysis 21: Comparison: Normal Vulva; Parameter: The difference in the incidence of aceto-whitening of Middle versus Inner Vulvar Ring in patients with normal vulva and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Middle versus Inner Vulvar Ring in patients with normal vulva and positive AWR?; p = 0.4975, t-test proportion

30. Secondary Outcome: Velocity of the Aceto-Whitening Reaction (Mean ± SD)
Description: The table shows the velocity (Mean ± SD) of the aceto-whitening occurrence after 5% acetic acid application (AWR - aceto-whitening reaction) in patients with positive AWR classified into four groups based on anamnestic data and clinical examination.
  Acetic acid is thought to cause swelling of the epithelial tissue through reversible coagulation or precipitation of the nuclear proteins and cytokeratins.
  Areas of pre-/malignant lesions turn densely white and opaque immediately after application of acetic acid, due to their higher concentration of abnormal nuclear protein and the presence of large numbers of dysplastic cells in the superficial layers of the epithelium.
  The acetowhite appearance is not unique to pre-/malignancy; it is also seen in other conditions with increased nuclear protein like immature squamous metaplasia, regeneration, inflammation, HPV-infection, hyperkeratosis, etc. The acetowhite reaction varies in intensity, within and between patients.
Time Frame: Aceto-Whitening Test, up to 10 minutes for each participant.
Population: The velocity of the AWR was measured with a stopwatch and noted into the "TRIV Form Data" only in the patients with a positive test.
Measure: Mean (Standard Deviation); unit: second
Arm/Group | Normal Vulva | Impaired Vulvar Skin | Vulvodynia | Vulvar Dermatosis
Number analyzed (Participants) | 37 | 74 | 81 | 57
second | 69.2 (24.3) | 54.9 (21.5) | 51.6 (21.2) | 65.9 (34.7)
Statistical Analysis 1: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the velocity of the aceto-whitening occurrence (positive AWR) among patients from different groups, in which the AWR was positive; Test type: Equivalence — Question: Is there a difference in the velocity of the aceto-whitening occurrence among patients from different groups, in which the AWR was positive?; p = 0.0003, ANOVA

31. Secondary Outcome: Velocity of Aceto-Whitening Reaction (Median | Range)
Description: The table shows the velocity (Median | Range) of the aceto-whitening occurrence after 5% acetic acid application (AWR - aceto-whitening reaction) in patients with positive AWR classified into four groups based on anamnestic data and clinical examination.
  Acetic acid is thought to cause swelling of the epithelial tissue through reversible coagulation or precipitation of the nuclear proteins and cytokeratins.
  Areas of pre-/malignant lesions turn densely white and opaque immediately after application of acetic acid, due to their higher concentration of abnormal nuclear protein and the presence of large numbers of dysplastic cells in the superficial layers of the epithelium.
  The acetowhite appearance is not unique to pre-/malignancy; it is also seen in other conditions with increased nuclear protein like immature squamous metaplasia, regeneration, inflammation, HPV-infection, hyperkeratosis, etc. The acetowhite reaction varies in intensity, within and between patients.
Time Frame: Aceto-Whitening Test, up to 10 minutes for each participant.
Population: as for outcome 30
Measure: Median (Full Range); unit: second
Arm/Group | Normal Vulva | Impaired Vulvar Skin | Vulvodynia | Vulvar Dermatosis
Number analyzed (Participants) | 37 | 74 | 81 | 57
second | 64.5 [30 to 120] | 51.5 [21 to 131] | 49 [16 to 120] | 58 [18 to 184]
Statistical Analysis 1: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the velocity of the aceto-whitening occurrence among patients with positive AWR from different groups; Test type: Equivalence — Question: Is there a difference in the velocity of the aceto-whitening occurrence among patients with positive AWR from different groups?; p = 0.0004, Kruskal-Wallis
Statistical Analysis 2: Comparison: Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the velocity of the aceto-whitening occurrence between patients with vulvar dermatosis and vulvodynia, with positive AWR; Test type: Superiority — Question: Is there a difference in the velocity of the aceto-whitening occurrence between patients with vulvar dermatosis and vulvodynia, with positive AWR?; p = 0.0231, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Normal Vulva vs Impaired Vulvar Skin; Parameter: The difference in the velocity of the aceto-whitening occurrence between the patients with normal vulva and impaired vulvar skin, with positive AWR; Test type: Superiority — Question: Is there a difference in the velocity of the aceto-whitening occurrence between the patients with normal vulva and impaired vulvar skin, with positive AWR?; p = 0.0006, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Normal Vulva vs Vulvodynia; Parameter: The difference in the velocity of the aceto-whitening occurrence between patients with normal vulva and vulvodynia, with positive AWR; Test type: Superiority — Question: Is there a difference in the velocity of the aceto-whitening occurrence between patients with normal vulva and vulvodynia, with positive AWR?; p = 0.0000, Wilcoxon (Mann-Whitney)

32. Secondary Outcome: Distribution of Aceto-Whitening Reaction in Relation to the Structures of the Outer Vulvar Ring
Description: The table shows the distribution of aceto-whitening occurrence (AWR) after 5% acetic acid application in relation to the structures of the Outer Vulvar Ring.
  The "OUTER Vulvar Ring" is presented with the following structures: Mons Pubis, Labia Majora, and the Perineum.
  Acetic acid is thought to cause swelling of the epithelial tissue through reversible coagulation or precipitation of the nuclear proteins and cytokeratins.
  Areas of pre-/malignant lesions turn densely white and opaque immediately after application of acetic acid, due to the presence of large numbers of dysplastic cells in the superficial layers of the epithelium.
  The acetowhite appearance is not unique to pre-/malignancy; it is also seen in other conditions with increased nuclear protein. The acetowhite reaction varies in intensity, within and between patients.
Time Frame: Aceto-Whitening Test, up to 10 minutes for each participant.
Population: We performed the aceto-whitening test with 5% acetic acid application in 328 patients, classified into four groups based on anamnestic data and clinical examination. Localization and type, as well as the velocity of the AWR, were mapped into the "TRIV Form Data".
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Vulva | Impaired Vulvar Skin | Vulvodynia | Vulvar Dermatosis
Number analyzed (Participants) | 82 | 82 | 82 | 82
Participants
  AWR of Mons Pubis | 0 | 0 | 0 | 8
  AWR of Labia Majora | 0 | 0 | 4 | 20
  AWR of the Perineum | 0 | 4 | 10 | 31
Statistical Analysis 1: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of aceto-whitening of Mons Pubis among patients from different groups, with positive AWR; Test type: Equivalence — Question: Is there a difference in the incidence of aceto-whitening of Mons Pubis among patients from different groups, with positive AWR?; p = 0.0000, Chi-squared
Statistical Analysis 2: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of aceto-whitening of Labia Majora among patients from different groups, with positive AWR; Test type: Equivalence — Question: Is there a difference in the incidence of aceto-whitening of Labia Majora among patients from different groups, with positive AWR?; p = 0.0000, Chi-squared
Statistical Analysis 3: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of aceto-whitening of the Perineum among patients from different groups, with positive AWR; Test type: Equivalence — Question: Is there a difference in the incidence of aceto-whitening of the Perineum among patients from different groups, with positive AWR?; p = 0.0000, Chi-squared
Statistical Analysis 4: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of aceto-whitening of Mons Pubis versus Labia Majora in patients with vulvar dermatosis and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Mons Pubis versus Labia Majora in patients with vulvar dermatosis and positive AWR?; p = 0.0128, t-test proportion
Statistical Analysis 5: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of aceto-whitening of Mons Pubis versus Perineum in patients with vulvar dermatosis and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Mons Pubis versus Perineum in patients with vulvar dermatosis and positive AWR?; p = 0.0000, t-test proportion
Statistical Analysis 6: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of aceto-whitening of Labia Majora versus Perineum in patients with vulvar dermatosis and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Labia Majora versus Perineum in patients with vulvar dermatosis and positive AWR?; p = 0.0635, t-test proportion
Statistical Analysis 7: Comparison: Vulvodynia; Parameter: The difference in the incidence of aceto-whitening of Mons Pubis versus Labia Majora in patients with vulvodynia and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Mons Pubis versus Labia Majora in patients with vulvodynia and positive AWR?; p = 0.0429, t-test proportion
Statistical Analysis 8: Comparison: Vulvodynia; Parameter: The difference in the incidence of aceto-whitening of Mons Pubis versus Perineum in patients with vulvodynia and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Mons Pubis versus Perineum in patients with vulvodynia and positive AWR?; p = 0.0011, t-test proportion
Statistical Analysis 9: Comparison: Vulvodynia; Parameter: The difference in the incidence of aceto-whitening of Labia Majora versus Perineum in patients with vulvodynia and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Labia Majora versus Perineum in patients with vulvodynia and positive AWR?; p = 0.0936, t-test proportion
Statistical Analysis 10: Comparison: Impaired Vulvar Skin; Parameter: The difference in the incidence of aceto-whitening of Mons Pubis versus Labia Majora in patients with impaired vulvar skin and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Mons Pubis versus Labia Majora in patients with impaired vulvar skin and positive AWR?; p = 1.0000, t-test proportion
Statistical Analysis 11: Comparison: Impaired Vulvar Skin; Parameter: The difference in the incidence of aceto-whitening of Mons Pubis versus Perineum in patients with impaired vulvar skin and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Mons Pubis versus Perineum in patients with impaired vulvar skin and positive AWR?; p = 0.0429, t-test proportion
Statistical Analysis 12: Comparison: Impaired Vulvar Skin; Parameter: The difference in the incidence of aceto-whitening of Labia Majora versus Perineum in patients with impaired vulvar skin and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Labia Majora versus Perineum in patients with impaired vulvar skin and positive AWR?; p = 0.0429, t-test proportion

33. Secondary Outcome: Distribution of Aceto-Whitening Reaction in Relation to the Structures of the Middle Vulvar Ring
Description: The distribution of aceto-whitening occurrence after 5% acetic acid application (AWR - aceto-whitening reaction) in relation to the structures of the Middle Vulvar Ring.
  The "MIDDLE vulvar ring" encompasses the following structures: the anterior commissure with the prepuce of the clitoris, interlabial sulci, labia minora, and the posterior commissure.
Time Frame: Aceto-Whitening Test, up to 10 minutes for each participant.
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Vulva | Impaired Vulvar Skin | Vulvodynia | Vulvar Dermatosis
Number analyzed (Participants) | 82 | 82 | 82 | 82
Participants
  AWR of the Anterior Commissure | 1 | 2 | 4 | 15
  AWR of Interlabial Sulci | 1 | 16 | 22 | 27
  AWR of Labia Minora | 6 | 20 | 43 | 27
  AWR of the Posterior Commissure | 23 | 53 | 72 | 40
Statistical Analysis 1: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of aceto-whitening of the Anterior Commissure among patients from different groups, with positive AWR; Test type: Equivalence — Question: Is there a difference in the incidence of aceto-whitening of the Anterior Commissure among patients from different groups, with positive AWR?; p = 0.0000, Chi-squared
Statistical Analysis 2: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of aceto-whitening of the Interlabial Sulci among patients from different groups, with positive AWR; Test type: Equivalence — Question: Is there a difference in the incidence of aceto-whitening of the Interlabial Sulci among patients from different groups, with positive AWR?; p = 0.0000, Chi-squared
Statistical Analysis 3: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of aceto-whitening of the Labia Minora among patients from different groups, with positive AWR; Test type: Equivalence — Question: Is there a difference in the incidence of aceto-whitening of the Labia Minora among patients from different groups, with positive AWR?; p = 0.0000, Chi-squared
Statistical Analysis 4: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of aceto-whitening of the Posterior Commissure among patients from different groups, with positive AWR; Test type: Equivalence — Question: Is there a difference in the incidence of aceto-whitening of the Posterior Commissure among patients from different groups, with positive AWR?; p = 0.0000, Chi-squared
Statistical Analysis 5: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of aceto-whitening of the Anterior Commissure versus Interlabial Sulci in patients with vulvar dermatosis and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of the Anterior Commissure versus Interlabial Sulci in patients with vulvar dermatosis and positive AWR?; p = 0.0318, t-test proportion
Statistical Analysis 6: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of aceto-whitening of the Anterior Commissure versus Labia Minora in patients with vulvar dermatosis and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of the Anterior Commissure versus Labia Minora in patients with vulvar dermatosis and positive AWR?; p = 0.0318, t-test proportion
Statistical Analysis 7: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of aceto-whitening of the Anterior Commissure versus Posterior Commissure in patients with vulvar dermatosis and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of the Anterior Commissure versus Posterior Commissure in patients with vulvar dermatosis and positive AWR?; p = 0.0000, t-test proportion
Statistical Analysis 8: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of aceto-whitening of the Interlabial Sulci versus Labia Minora in patients with vulvar dermatosis and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of the Interlabial Sulci versus Labia Minora in patients with vulvar dermatosis and positive AWR?; p = 1.0000, t-test proportion
Statistical Analysis 9: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of aceto-whitening of the Interlabial Sulci versus Posterior Commissure in patients with vulvar dermatosis and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of the Interlabial Sulci versus Posterior Commissure in patients with vulvar dermatosis and positive AWR?; p = 0.0389, t-test proportion
Statistical Analysis 10: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of aceto-whitening of the Labia Minora versus Posterior Commissure in patients with vulvar dermatosis and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of the Labia Minora versus Posterior Commissure in patients with vulvar dermatosis and positive AWR?; p = 0.0389, t-test proportion
Statistical Analysis 11: Comparison: Vulvodynia; Parameter: The difference in the incidence of aceto-whitening of the Anterior Commissure versus Interlabial Sulci in patients with vulvodynia and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of the Anterior Commissure versus Interlabial Sulci in patients with vulvodynia and positive AWR?; p = 0.00001, t-test proportion
Statistical Analysis 12: Comparison: Vulvodynia; Parameter: The difference in the incidence of aceto-whitening of the Anterior Commissure versus Labia Minora in patients with vulvodynia and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of the Anterior Commissure versus Labia Minora in patients with vulvodynia and positive AWR?; p = 0.0000, t-test proportion
Statistical Analysis 13: Comparison: Vulvodynia; Parameter: The difference in the incidence of aceto-whitening of the Anterior Commissure versus Posterior Commissure in patients with vulvodynia and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of the Anterior Commissure versus Posterior Commissure in patients with vulvodynia and positive AWR?; p = 0.0000, t-test proportion
Statistical Analysis 14: Comparison: Vulvodynia; Parameter: The difference in the incidence of aceto-whitening of Interlabial Sulci versus Labia Minora in patients with vulvodynia and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Interlabial Sulci versus Labia Minora in patients with vulvodynia and positive AWR?; p = 0.0008, t-test proportion
Statistical Analysis 15: Comparison: Vulvodynia; Parameter: The difference in the incidence of aceto-whitening of Interlabial Sulci versus Posterior Commissure in patients with vulvodynia and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Interlabial Sulci versus Posterior Commissure in patients with vulvodynia and positive AWR?; p = 0.0000, t-test proportion
Statistical Analysis 16: Comparison: Vulvodynia; Parameter: The difference in the incidence of aceto-whitening of Labia Minora versus Posterior Commissure in patients with vulvodynia and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Labia Minora versus Posterior Commissure in patients with vulvodynia and positive AWR?; p = 0.0000, t-test proportion
Statistical Analysis 17: Comparison: Impaired Vulvar Skin; Parameter: The difference in the incidence of aceto-whitening of the Anterior Commissure versus Interlabial Sulci in patients with impaired vulvar skin and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of the Anterior Commissure versus Interlabial Sulci in patients with impaired vulvar skin and positive AWR?; p = 0.0005, t-test proportion
Statistical Analysis 18: Comparison: Impaired Vulvar Skin; Parameter: The difference in the incidence of aceto-whitening of the Anterior Commissure versus Labia Minora in patients with impaired vulvar skin and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of the Anterior Commissure versus Labia Minora in patients with impaired vulvar skin and positive AWR?; p = 0.0000, t-test proportion
Statistical Analysis 19: Comparison: Impaired Vulvar Skin; Parameter: The difference in the incidence of aceto-whitening of the Anterior Commissure versus Posterior Commissure in patients with impaired vulvar skin and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of the Anterior Commissure versus Posterior Commissure in patients with impaired vulvar skin and positive AWR?; p = 0.0000, t-test proportion
Statistical Analysis 20: Comparison: Impaired Vulvar Skin; Parameter: The difference in the incidence of aceto-whitening of the Interlabial Sulci versus Labia Minora in patients with impaired vulvar skin and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of the Interlabial Sulci versus Labia Minora in patients with impaired vulvar skin and positive AWR?; p = 0.4505, t-test proportion
Statistical Analysis 21: Comparison: Impaired Vulvar Skin; Parameter: The difference in the incidence of aceto-whitening of Interlabial Sulci versus Posterior Commissure in patients with impaired vulvar skin and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Interlabial Sulci versus Posterior Commissure in patients with impaired vulvar skin and positive AWR?; p = 0.0000, t-test proportion
Statistical Analysis 22: Comparison: Impaired Vulvar Skin; Parameter: The difference in the incidence of aceto-whitening of the Labia Minora versus Posterior Commissure in patients with impaired vulvar skin and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of the Labia Minora versus Posterior Commissure in patients with impaired vulvar skin and positive AWR?; p = 0.0000, t-test proportion
Statistical Analysis 23: Comparison: Normal Vulva; Parameter: The difference in the incidence of aceto-whitening of the Anterior Commissure versus Interlabial Sulci in patients with normal vulva and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of the Anterior Commissure versus Interlabial Sulci in patients with normal vulva and positive AWR?; p = 1.0000, t-test proportion
Statistical Analysis 24: Comparison: Normal Vulva; Parameter: The difference in the incidence of aceto-whitening of the Anterior Commissure versus Labia Minora in patients with normal vulva and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of the Anterior Commissure versus Labia Minora in patients with normal vulva and positive AWR?; p = 0.0534, t-test proportion
Statistical Analysis 25: Comparison: Normal Vulva; Parameter: The difference in the incidence of aceto-whitening of the Anterior Commissure versus Posterior Commissure in patients with normal vulva and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of the Anterior Commissure versus Posterior Commissure in patients with normal vulva and positive AWR?; p = 0.0000, t-test proportion
Statistical Analysis 26: Comparison: Normal Vulva; Parameter: The difference in the incidence of aceto-whitening of the Interlabial Sulci versus Labia Minora in patients with normal vulva and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of the Interlabial Sulci versus Labia Minora in patients with normal vulva and positive AWR?; p = 0.0534, t-test proportion
Statistical Analysis 27: Comparison: Normal Vulva; Parameter: The difference in the incidence of aceto-whitening of the Interlabial Sulci versus Posterior Commissure in patients with normal vulva and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of the Interlabial Sulci versus Posterior Commissure in patients with normal vulva and positive AWR?; p = 0.0000, t-test proportion
Statistical Analysis 28: Comparison: Normal Vulva; Parameter: The difference in the incidence of aceto-whitening of the Labia Minora versus Posterior Commissure in patients with normal vulva and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of the Labia Minora versus Posterior Commissure in patients with normal vulva and positive AWR?; p = 0.0005, t-test proportion

34. Secondary Outcome: Distribution of Aceto-Whitening Reaction in Relation to the Structures of the Inner Vulvar Ring
Description: The table shows the distribution of aceto-whitening reaction (AWR) after 5% acetic acid application (AWR - aceto-whitening reaction) in relation to the structures of the Inner Vulvar Ring.
  The "INNER Vulvar Ring" is presented with the following structures: the clitoris, Hart's line, the urethral sulcus, the urethral meatus, hymenal remnants, Bartholin's gland opening, and the vestibule.
  Acetic acid is thought to cause swelling of the epithelial tissue through reversible coagulation or precipitation of the nuclear proteins and cytokeratins.
  Areas of pre-/malignant lesions turn densely white and opaque immediately after application of acetic acid, due to the presence of large numbers of dysplastic cells in the superficial layers of the epithelium.
  The acetowhite appearance is not unique to pre-/malignancy; it is also seen in other conditions with increased nuclear protein. The acetowhite reaction varies in intensity, within and between patients.
Time Frame: Aceto-Whitening Test, up to 10 minutes for each participant.
Population: We performed the aceto-whitening test with 5% acetic acid application in 328 patients, classified into four groups based on anamnestic data and clinical examination. Localization and type, as well as the velocity of the AWR, were mapped into the "TRIV Form Data". Aceto-Whitening of all structures of the Inner vulvar ring was named "Ring sign".
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Vulva | Impaired Vulvar Skin | Vulvodynia | Vulvar Dermatosis
Number analyzed (Participants) | 82 | 82 | 82 | 82
Participants
  AWR of the Clitoris | 8 | 35 | 73 | 20
  AWR of Hart's Line | 14 | 50 | 79 | 19
  AWR of the Urethral Sulcus | 16 | 49 | 73 | 21
  AWR of the Urethral Meatus | 6 | 38 | 70 | 14
  AWR of Hymenal Remnants | 6 | 33 | 69 | 14
  AWR of Bartholin's Gland Opening | 8 | 42 | 75 | 12
  AWR of the Vestibule | 21 | 49 | 76 | 23
Statistical Analysis 1: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of aceto-whitening of the Clitoris among patients from different groups, with positive AWR; Test type: Equivalence — Question: Is there a difference in the incidence of aceto-whitening of the Clitoris among patients from different groups, with positive AWR?; p = 0.0000, Chi-squared
Statistical Analysis 2: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of aceto-whitening of Hart's Line among patients from different groups, with positive AWR; Test type: Equivalence — Question: Is there a difference in the incidence of aceto-whitening of Hart's Line among patients from different groups, with positive AWR?; p = 0.0000, Chi-squared
Statistical Analysis 3: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of aceto-whitening of the Urethral Sulcus among patients from different groups, with positive AWR; Test type: Equivalence — Question: Is there a difference in the incidence of aceto-whitening of the Urethral Sulcus among patients from different groups, with positive AWR?; p = 0.0000, Chi-squared
Statistical Analysis 4: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of aceto-whitening of the Urethral Meatus among patients from different groups, with positive AWR; Test type: Equivalence — Question: Is there a difference in the incidence of aceto-whitening of the Urethral Meatus among patients from different groups, with positive AWR?; p = 0.0000, Chi-squared
Statistical Analysis 5: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of aceto-whitening of Hymenal Remnants among patients from different groups, with positive AWR; Test type: Equivalence — Question: Is there a difference in the incidence of aceto-whitening of Hymenal Remnants among patients from different groups, with positive AWR?; p = 0.0000, Chi-squared
Statistical Analysis 6: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of aceto-whitening of Bartholin's Gland Opening among patients from different groups, with positive AWR; Test type: Equivalence — Question: Is there a difference in the incidence of aceto-whitening of Bartholin's Gland Opening among patients from different groups, with positive AWR?; p = 0.0000, Chi-squared
Statistical Analysis 7: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of aceto-whitening of the Vestibule among patients from different groups, with positive AWR; Test type: Equivalence — Question: Is there a difference in the incidence of aceto-whitening of the Vestibule among patients from different groups, with positive AWR?; p = 0.0000, Chi-squared
Statistical Analysis 8: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of aceto-whitening of the Clitoris versus Hart's line in patients with vulvar dermatosis and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of the Clitoris versus Hart's line in patients with vulvar dermatosis and positive AWR?; p = 0.8545, t-test proportion
Statistical Analysis 9: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of aceto-whitening of the Clitoris versus Urethral Sulcus in patients with vulvar dermatosis and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of the Clitoris versus Urethral Sulcus in patients with vulvar dermatosis and positive AWR?; p = 0.8569, t-test proportion
Statistical Analysis 10: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of aceto-whitening of the Clitoris versus Urethral Meatus in patients with vulvar dermatosis and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of the Clitoris versus Urethral Meatus in patients with vulvar dermatosis and positive AWR?; p = 0.2478, t-test proportion
Statistical Analysis 11: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of aceto-whitening of the Clitoris versus Hymenal Remnants in patients with vulvar dermatosis and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of the Clitoris versus Hymenal Remnants in patients with vulvar dermatosis and positive AWR?; p = 0.2478, t-test proportion
Statistical Analysis 12: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of aceto-whitening of the Clitoris versus Bartholin's Gland Opening in patients with vulvar dermatosis and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of the Clitoris versus Bartholin's Gland Opening in patients with vulvar dermatosis and positive AWR?; p = 0.1627, t-test proportion
Statistical Analysis 13: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of aceto-whitening of the Clitoris versus Vestibule in patients with vulvar dermatosis and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of the Clitoris versus Vestibule in patients with vulvar dermatosis and positive AWR?; p = 0.5943, t-test proportion
Statistical Analysis 14: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of aceto-whitening of Hart's Line versus Urethral Sulcus in patients with vulvar dermatosis and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Hart's Line versus Urethral Sulcus in patients with vulvar dermatosis and positive AWR?; p = 0.7161, t-test proportion
Statistical Analysis 15: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of aceto-whitening of Hart's Line versus Urethral Meatus in patients with vulvar dermatosis and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Hart's Line versus Urethral Meatus in patients with vulvar dermatosis and positive AWR?; p = 0.3301, t-test proportion
Statistical Analysis 16: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of aceto-whitening of Hart's Line versus Hymenal Remnants in patients with vulvar dermatosis and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Hart's Line versus Hymenal Remnants in patients with vulvar dermatosis and positive AWR?; p = 0.3301, t-test proportion
Statistical Analysis 17: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of aceto-whitening of Hart's Line versus Bartholin's Gland Opening in patients with vulvar dermatosis and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Hart's Line versus Bartholin's Gland Opening in patients with vulvar dermatosis and positive AWR?; p = 0.1627, t-test proportion
Statistical Analysis 18: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of aceto-whitening of Hart's Line versus Vestibule in patients with vulvar dermatosis and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Hart's Line versus Vestibule in patients with vulvar dermatosis and positive AWR?; p = 0.4742, t-test proportion
Statistical Analysis 19: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of aceto-whitening of Urethral Sulcus versus Urethral Meatus in patients with vulvar dermatosis and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Urethral Sulcus versus Urethral Meatus in patients with vulvar dermatosis and positive AWR?; p = 0.1822, t-test proportion
Statistical Analysis 20: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of aceto-whitening of Urethral Sulcus versus Hymenal Remnants in patients with vulvar dermatosis and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Urethral Sulcus versus Hymenal Remnants in patients with vulvar dermatosis and positive AWR?; p = 0.1822, t-test proportion
Statistical Analysis 21: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of aceto-whitening of Hymenal Remnants versus Vestibule in patients with vulvar dermatosis and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Hymenal Remnants versus Vestibule in patients with vulvar dermatosis and positive AWR?; p = 0.0927, t-test proportion
Statistical Analysis 22: Comparison: Vulvar Dermatosis; Parameter: The difference in the incidence of aceto-whitening of Bartholin's Gland Opening versus Vestibule in patients with vulvar dermatosis and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Bartholin's Gland Opening versus Vestibule in patients with vulvar dermatosis and positive AWR?; p = 0.0360, t-test proportion
Statistical Analysis 23: Comparison: Vulvodynia; Parameter: The difference in the incidence of aceto-whitening of the Clitoris versus Hart's Line in patients with vulvodynia and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of the Clitoris versus Hart's Line in patients with vulvodynia and positive AWR?; p = 0.0720, t-test proportion
Statistical Analysis 24: Comparison: Vulvodynia; Parameter: The difference in the incidence of aceto-whitening of the Clitoris versus Urethral Sulcus in patients with vulvodynia and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of the Clitoris versus Urethral Sulcus in patients with vulvodynia and positive AWR?; p = 1.0000, t-test proportion
Statistical Analysis 25: Comparison: Vulvodynia; Parameter: The difference in the incidence of aceto-whitening of the Clitoris versus Urethral Meatus in patients with vulvodynia and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of the Clitoris versus Urethral Meatus in patients with vulvodynia and positive AWR?; p = 0.4833, t-test proportion
Statistical Analysis 26: Comparison: Vulvodynia; Parameter: The difference in the incidence of aceto-whitening of the Clitoris versus Hymenal Remnants in patients with vulvodynia and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of the Clitoris versus Hymenal Remnants in patients with vulvodynia and positive AWR?; p = 0.3594, t-test proportion
Statistical Analysis 27: Comparison: Vulvodynia; Parameter: The difference in the incidence of aceto-whitening of the Clitoris versus Bartholin's Gland Opening in patients with vulvodynia and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of the Clitoris versus Bartholin's Gland Opening in patients with vulvodynia and positive AWR?; p = 0.5987, t-test proportion
Statistical Analysis 28: Comparison: Vulvodynia; Parameter: The difference in the incidence of aceto-whitening of the Clitoris versus Vestibule in patients with vulvodynia and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of the Clitoris versus Vestibule in patients with vulvodynia and positive AWR?; p = 0.4164, t-test proportion
Statistical Analysis 29: Comparison: Vulvodynia; Parameter: The difference in the incidence of aceto-whitening of Hart's Line versus Urethral Sulcus in patients with vulvodynia and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Hart's Line versus Urethral Sulcus in patients with vulvodynia and positive AWR?; p = 0.0720, t-test proportion
Statistical Analysis 30: Comparison: Vulvodynia; Parameter: The difference in the incidence of aceto-whitening of Hart's Line versus Urethral Meatus in patients with vulvodynia and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Hart's Line versus Urethral Meatus in patients with vulvodynia and positive AWR?; p = 0.0148, t-test proportion
Statistical Analysis 31: Comparison: Vulvodynia; Parameter: The difference in the incidence of aceto-whitening of Hart's Line versus Hymenal Remnants in patients with vulvodynia and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Hart's Line versus Hymenal Remnants in patients with vulvodynia and positive AWR?; p = 0.0085, t-test proportion
Statistical Analysis 32: Comparison: Vulvodynia; Parameter: The difference in the incidence of aceto-whitening of Hart's Line versus Bartholin's Gland Opening in patients with vulvodynia and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Hart's Line versus Bartholin's Gland Opening in patients with vulvodynia and positive AWR?; p = 0.1918, t-test proportion
Statistical Analysis 33: Comparison: Vulvodynia; Parameter: The difference in the incidence of aceto-whitening of Hart's line versus Vestibule in patients with vulvodynia and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Hart's line versus Vestibule in patients with vulvodynia and positive AWR?; p = 0.3037, t-test proportion
Statistical Analysis 34: Comparison: Vulvodynia; Parameter: The difference in the incidence of aceto-whitening of the Urethral Sulcus versus Urethral Meatus in patients with vulvodynia and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of the Urethral Sulcus versus Urethral Meatus in patients with vulvodynia and positive AWR?; p = 0.4833, t-test proportion
Statistical Analysis 35: Comparison: Vulvodynia; Parameter: The difference in the incidence of aceto-whitening of the Urethral Sulcus versus Hymenal Remnants in patients with vulvodynia and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of the Urethral Sulcus versus Hymenal Remnants in patients with vulvodynia and positive AWR?; p = 0.3594, t-test proportion
Statistical Analysis 36: Comparison: Vulvodynia; Parameter: The difference in the incidence of aceto-whitening of the Hymenal Remnants versus Vestibule in patients with vulvodynia and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of the Hymenal Remnants versus Vestibule in patients with vulvodynia and positive AWR?; p = 0.0877, t-test proportion
Statistical Analysis 37: Comparison: Vulvodynia; Parameter: The difference in the incidence of aceto-whitening of Bartholin's Gland Opening versus Vestibule in patients with vulvodynia and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Bartholin's Gland Opening versus Vestibule in patients with vulvodynia and positive AWR?; p = 0.7726, t-test proportion
Statistical Analysis 38: Comparison: Impaired Vulvar Skin; Parameter: The difference in the incidence of aceto-whitening of the Clitoris versus Hart's Line in patients with impaired vulvar skin and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of the Clitoris versus Hart's Line in patients with impaired vulvar skin and positive AWR?; p = 0.0191, t-test proportion
Statistical Analysis 39: Comparison: Impaired Vulvar Skin; Parameter: The difference in the incidence of aceto-whitening of the Clitoris versus Urethral Sulcus in patients with impaired vulvar skin and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of the Clitoris versus Urethral Sulcus in patients with impaired vulvar skin and positive AWR?; p = 0.0287, t-test proportion
Statistical Analysis 40: Comparison: Impaired Vulvar Skin; Parameter: The difference in the incidence of aceto-whitening of the Clitoris versus Urethral Meatus in patients with impaired vulvar skin and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of the Clitoris versus Urethral Meatus in patients with impaired vulvar skin and positive AWR?; p = 0.6374, t-test proportion
Statistical Analysis 41: Comparison: Impaired Vulvar Skin; Parameter: The difference in the incidence of aceto-whitening of the Clitoris versus Hymenal Remnants in patients with impaired vulvar skin and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of the Clitoris versus Hymenal Remnants in patients with impaired vulvar skin and positive AWR?; p = 0.7512, t-test proportion
Statistical Analysis 42: Comparison: Impaired Vulvar Skin; Parameter: The difference in the incidence of aceto-whitening of the Clitoris versus Bartholin's Gland Opening in patients with impaired vulvar skin and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of the Clitoris versus Bartholin's Gland Opening in patients with impaired vulvar skin and positive AWR?; p = 0.2734, t-test proportion
Statistical Analysis 43: Comparison: Impaired Vulvar Skin; Parameter: The difference in the incidence of aceto-whitening of the Clitoris versus Vestibule in patients with impaired vulvar skin and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of the Clitoris versus Vestibule in patients with impaired vulvar skin and positive AWR?; p = 0.0287, t-test proportion
Statistical Analysis 44: Comparison: Impaired Vulvar Skin; Parameter: The difference in the incidence of aceto-whitening of Hart's Line versus Urethral Sulcus in patients with impaired vulvar skin and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Hart's Line versus Urethral Sulcus in patients with impaired vulvar skin and positive AWR?; p = 0.8732, t-test proportion
Statistical Analysis 45: Comparison: Impaired Vulvar Skin; Parameter: The difference in the incidence of aceto-whitening of Hart's Line versus Urethral Meatus in patients with impaired vulvar skin and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Hart's Line versus Urethral Meatus in patients with impaired vulvar skin and positive AWR?; p = 0.0602, t-test proportion
Statistical Analysis 46: Comparison: Impaired Vulvar Skin; Parameter: The difference in the incidence of aceto-whitening of Hart's Line versus Hymenal Remnants in patients with impaired vulvar skin and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Hart's Line versus Hymenal Remnants in patients with impaired vulvar skin and positive AWR?; p = 0.0079, t-test proportion
Statistical Analysis 47: Comparison: Impaired Vulvar Skin; Parameter: The difference in the incidence of aceto-whitening of Hart's Line versus Bartholin's Gland Opening in patients with impaired vulvar skin and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Hart's Line versus Bartholin's Gland Opening in patients with impaired vulvar skin and positive AWR?; p = 0.2081, t-test proportion
Statistical Analysis 48: Comparison: Impaired Vulvar Skin; Parameter: The difference in the incidence of aceto-whitening of Hart's Line versus Vestibule in patients with impaired vulvar skin and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Hart's Line versus Vestibule in patients with impaired vulvar skin and positive AWR?; p = 0.8732, t-test proportion
Statistical Analysis 49: Comparison: Impaired Vulvar Skin; Parameter: The difference in the incidence of aceto-whitening of the Urethral Sulcus versus Urethral Meatus in patients with impaired vulvar skin and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of the Urethral Sulcus versus Urethral Meatus in patients with impaired vulvar skin and positive AWR?; p = 0.0852, t-test proportion
Statistical Analysis 50: Comparison: Impaired Vulvar Skin; Parameter: The difference in the incidence of aceto-whitening of the Urethral Sulcus versus Hymenal Remnants in patients with impaired vulvar skin and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of the Urethral Sulcus versus Hymenal Remnants in patients with impaired vulvar skin and positive AWR?; p = 0.0125, t-test proportion
Statistical Analysis 51: Comparison: Impaired Vulvar Skin; Parameter: The difference in the incidence of aceto-whitening of Hymenal Remnants versus Vestibule in patients with impaired vulvar skin and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Hymenal Remnants versus Vestibule in patients with impaired vulvar skin and positive AWR?; p = 0.0125, t-test proportion
Statistical Analysis 52: Comparison: Impaired Vulvar Skin; Parameter: The difference in the incidence of aceto-whitening of Bartholin's Gland Opening versus Vestibule in patients with impaired vulvar skin and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Bartholin's Gland Opening versus Vestibule in patients with impaired vulvar skin and positive AWR?; p = 0.2714, t-test proportion
Statistical Analysis 53: Comparison: Normal Vulva; Parameter: The difference in the incidence of aceto-whitening of the Clitoris versus Hart's Line in patients with normal vulva and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of the Clitoris versus Hart's Line in patients with normal vulva and positive AWR?; p = 0.1692, t-test proportion
Statistical Analysis 54: Comparison: Normal Vulva; Parameter: The difference in the incidence of aceto-whitening of the Clitoris versus Urethral Sulcus in patients with normal vulva and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of the Clitoris versus Urethral Sulcus in patients with normal vulva and positive AWR?; p = 0.0772, t-test proportion
Statistical Analysis 55: Comparison: Normal Vulva; Parameter: The difference in the incidence of aceto-whitening of the Clitoris versus Urethral Meatus in patients with normal vulva and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of the Clitoris versus Urethral Meatus in patients with normal vulva and positive AWR?; p = 0.5762, t-test proportion
Statistical Analysis 56: Comparison: Normal Vulva; Parameter: The difference in the incidence of aceto-whitening of the Clitoris versus Hymenal Remnants in patients with normal vulva and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of the Clitoris versus Hymenal Remnants in patients with normal vulva and positive AWR?; p = 0.5762, t-test proportion
Statistical Analysis 57: Comparison: Normal Vulva; Parameter: The difference in the incidence of aceto-whitening of the Clitoris versus Bartholin's Gland Opening in patients with normal vulva and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of the Clitoris versus Bartholin's Gland Opening in patients with normal vulva and positive AWR?; p = 1.0000, t-test proportion
Statistical Analysis 58: Comparison: Normal Vulva; Parameter: The difference in the incidence of aceto-whitening of the Clitoris versus Vestibule in patients with normal vulva and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of the Clitoris versus Vestibule in patients with normal vulva and positive AWR?; p = 0.0078, t-test proportion
Statistical Analysis 59: Comparison: Normal Vulva; Parameter: The difference in the incidence of aceto-whitening of Hart's Line versus Urethral Sulcus in patients with normal vulva and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Hart's Line versus Urethral Sulcus in patients with normal vulva and positive AWR?; p = 0.6862, t-test proportion
Statistical Analysis 60: Comparison: Normal Vulva; Parameter: The difference in the incidence of aceto-whitening of Hart's Line versus Urethral Meatus in patients with normal vulva and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Hart's Line versus Urethral Meatus in patients with normal vulva and positive AWR?; p = 0.0563, t-test proportion
Statistical Analysis 61: Comparison: Normal Vulva; Parameter: The difference in the incidence of aceto-whitening of Hart's Line versus Hymenal Remnants in patients with normal vulva and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Hart's Line versus Hymenal Remnants in patients with normal vulva and positive AWR?; p = 0.0563, t-test proportion
Statistical Analysis 62: Comparison: Normal Vulva; Parameter: The difference in the incidence of aceto-whitening of Hart's Line versus Bartholin's Gland Opening in patients with normal vulva and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Hart's Line versus Bartholin's Gland Opening in patients with normal vulva and positive AWR?; p = 0.1692, t-test proportion
Statistical Analysis 63: Comparison: Normal Vulva; Parameter: The difference in the incidence of aceto-whitening of Hart's Line versus Vestibule in patients with normal vulva and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Hart's Line versus Vestibule in patients with normal vulva and positive AWR?; p = 0.1822, t
Statistical Analysis 64: Comparison: Normal Vulva; Parameter: The difference in the incidence of aceto-whitening of Urethral Sulcus versus Urethral Meatus in patients with normal vulva and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Urethral Sulcus versus Urethral Meatus in patients with normal vulva and positive AWR?; p = 0.0220, t-test proportion
Statistical Analysis 65: Comparison: Normal Vulva; Parameter: The difference in the incidence of aceto-whitening of Urethral Sulcus versus Hymenal Remnants in patients with normal vulva and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Urethral Sulcus versus Hymenal Remnants in patients with normal vulva and positive AWR?; p = 0.0220, t-test proportion
Statistical Analysis 66: Comparison: Normal Vulva; Parameter: The difference in the incidence of aceto-whitening of Hymenal Remnants versus Vestibule in patients with normal vulva and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Hymenal Remnants versus Vestibule in patients with normal vulva and positive AWR?; p = 0.0220, t-test proportion
Statistical Analysis 67: Comparison: Normal Vulva; Parameter: The difference in the incidence of aceto-whitening of Bartholin's Gland Opening versus Vestibule in patients with normal vulva and positive AWR; Test type: Superiority — Question: Is there a difference in the incidence of aceto-whitening of Bartholin's Gland Opening versus Vestibule in patients with normal vulva and positive AWR?; p = 0.0078, t-test proportion

35. Secondary Outcome: Histopathological Characteristics of Vulvar Specimens in Patients With And Without Vulvar Discomfort
Description: The table shows the distribution of histopathological findings of vulvar epidermis among patients with and without vulvar discomfort, classified into four groups based on anamnestic data, clinical examination and "Three Rings Vulvoscopy." Histopathological characteristics of vulvar epidermis included hyperkeratosis, parakeratosis, acanthosis, and epidermal atrophy. In the vulvar dermis, there were evaluated presence of inflammatory infiltrates (monocytes, lymphocytes, mastocytes), collagen fibers, hyalinization, hyperpigmentation, elongated dermal papillae, blood vessels, sebaceous glands, and nerve fibers.
Time Frame: Histopathological Examination, up to 30 minutes for each vulvar sample.
Population: We performed a biopsy of the vulva in 164 symptomatic patients during the routine clinical care to histopathologically confirm or exclude a skin disorder. Vulvar specimens from 164 asymptomatic patients were granted from the women undergoing planned labiaplasty.
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Vulva | Impaired Vulvar Skin | Vulvodynia | Vulvar Dermatosis
Number analyzed (Participants) | 82 | 82 | 82 | 82
Participants
  Hyperkeratosis | 0 | 6 | 3 | 62
  Parakeratosis | 3 | 5 | 7 | 30
  Acanthosis | 3 | 1 | 1 | 16
  Epidermal Atrophy | 0 | 0 | 0 | 25
  Inflammatory Infiltrates | 42 | 52 | 65 | 73
  Mononuclear Infiltrates | 33 | 46 | 61 | 63
  Lymphocytes | 9 | 3 | 3 | 13
  Mastocytes | 2 | 0 | 6 | 0
  Collagen Fibers | 7 | 1 | 9 | 44
  Hyalinization | 2 | 0 | 0 | 25
  Hyperpigmentation | 7 | 2 | 5 | 0
  Elongated Dermal Papillae | 5 | 7 | 0 | 1
  Blood Vessels | 31 | 30 | 53 | 5
  Sebaceous Glands | 39 | 48 | 61 | 1
  Nerve Fibers | 28 | 27 | 68 | 0
Statistical Analysis 1: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of the histopathological finding of hyperkeratosis in vulvar specimens of patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of hyperkeratosis in vulvar specimens of patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 2: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of the histopathological finding of parakeratosis in vulvar specimens of patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of parakeratosis in vulvar specimens of patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 3: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of the histopathological finding of acanthosis in vulvar specimens of patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of acanthosis in vulvar specimens of patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 4: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of the histopathological finding of epidermal atrophy in vulvar specimens of patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of epidermal atrophy in vulvar specimens of patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 5: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of the histopathological finding of inflammatory infiltrates in vulvar specimens of patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of inflammatory infiltrates in vulvar specimens of patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 6: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of the histopathological finding of mononuclear inflammatory infiltrates in vulvar specimens of patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of mononuclear inflammatory infiltrates in vulvar specimens of patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 7: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of the histopathological finding of lymphocytes (infiltrates) in vulvar specimens of patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of lymphocytes in vulvar specimens of patients from different groups?; p = 0.0105, Chi-squared
Statistical Analysis 8: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of the histopathological finding of mastocytes in vulvar specimens of patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of mastocytes in vulvar specimens of patients from different groups?; p = 0.0064, Chi-squared
Statistical Analysis 9: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of the histopathological finding of collagen fibers in vulvar specimens of patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of collagen fibers in vulvar specimens of patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 10: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of the histopathological finding of hyalinization in vulvar specimens of patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of hyalinization in vulvar specimens of patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 11: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of the histopathological finding of hyperpigmentation in vulvar specimens of patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of hyperpigmentation in vulvar specimens of patients from different groups?; p = 0.0342, Chi-squared
Statistical Analysis 12: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of the histopathological finding of elongated dermal papillae in vulvar specimens of patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of elongated dermal papillae in vulvar specimens of patients from different groups?; p = 0.0148, Chi-squared
Statistical Analysis 13: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of the histopathological finding of blood vessels in vulvar specimens of patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of blood vessels in vulvar specimens of patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 14: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of the histopathological finding of sebaceous glands in vulvar specimens of patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of sebaceous glands in vulvar specimens of patients from different groups?; p = 0.0000, Chi-squared
Statistical Analysis 15: Comparison: Normal Vulva vs Impaired Vulvar Skin vs Vulvodynia vs Vulvar Dermatosis; Parameter: The difference in the incidence of the histopathological finding of nerve fibers in vulvar specimens of patients from different groups; Test type: Equivalence — Question: Is there a difference in the incidence of nerve fibers in vulvar specimens of patients from different groups?; p = 0.0000, Chi-squared

36. Secondary Outcome: Histopathological Features of the Vulvar Epidermis and Vulvar Discomfort in Patients With Vulvar Dermatosis
Description: The table shows the relationship between histopathological features of the vulvar epidermis (normal versus abnormal) and single vulvar symptoms from the categories of the dull ("slow") and sharp ("fast") pain of the vulva in 82 patients with vulvar dermatosis.
  The dull pain comprises sensations of burning, stinging, soreness, irritation,itching, inflammation and aching.
  The fast pain includes sensations like sticking and stabbing, paper-cut or knife-like pain.
Time Frame: Histopathological Examination, up to 30 minutes for each vulvar sample.
Population: We performed a biopsy of the vulva in 82 symptomatic patients with vulvar dermatosis diagnosed anamnestically and by clinical examination during the routine clinical care, to confirm the diagnosis on histopathology.
Measure: Count of Participants; unit: Participants
Groups:
- Vulvar Dermatosis With Normal Epidermis: Histopathological Finding of Normal Epidermis among the various vulvar complaints in patients with vulvar dermatosis.
- Vulvar Dermatosis With Abnormal Epidermis: Histopathological Finding of Abnormal Epidermis among the various vulvar complaints in patients with vulvar dermatosis.
Arm/Group | Vulvar Dermatosis With Normal Epidermis | Vulvar Dermatosis With Abnormal Epidermis
Number analyzed (Participants) | 29 | 53
Participants
  Dull / Slow Pain | 29 | 53
  Burning | 6 | 16
  Stinging | 24 | 41
  Soreness | 13 | 24
  Irritation | 12 | 23
  Itching | 28 | 51
  Inflammation | 13 | 25
  Aching | 8 | 13
  Sharp / Fast Pain | 3 | 9
  Knife-Like Pain | 0 | 5
  Paper-Cuts Pain | 1 | 2
  Stabbing | 2 | 4
  Sticking | 3 | 6
Statistical Analysis 1: Comparison: Vulvar Dermatosis With Normal Epidermis vs Vulvar Dermatosis With Abnormal Epidermis; Parameter: The difference in the incidence of vulvar complaints depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of vulvar complaints depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvar dermatosis?; p = 0.0000, Chi-squared
Statistical Analysis 2: Comparison: Vulvar Dermatosis With Normal Epidermis vs Vulvar Dermatosis With Abnormal Epidermis; Parameter: The difference in the incidence of symptoms of the dull (slow) pain of the vulva (burning, stinging, soreness, irritation, itching, inflammation, aching) depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of symptoms of the dull pain of the vulva on the histopathology of the epidermis (normal versus abnormal) in patients with vulvar dermatosis?; p = 1.0000, Chi-squared
Statistical Analysis 3: Comparison: Vulvar Dermatosis With Normal Epidermis vs Vulvar Dermatosis With Abnormal Epidermis; Parameter: The incidence of vulvar burning depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of vulvar burning depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvar dermatosis?; p = 0.3533, Chi-squared
Statistical Analysis 4: Comparison: Vulvar Dermatosis With Normal Epidermis vs Vulvar Dermatosis With Abnormal Epidermis; Parameter: The incidence of vulvar stinging depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of vulvar stinging depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvar dermatosis?; p = 0.5641, Chi-squared
Statistical Analysis 5: Comparison: Vulvar Dermatosis With Normal Epidermis vs Vulvar Dermatosis With Abnormal Epidermis; Parameter: The incidence of vulvar soreness depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of vulvar soreness depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvar dermatosis?; p = 0.9684, Chi-squared
Statistical Analysis 6: Comparison: Vulvar Dermatosis With Normal Epidermis vs Vulvar Dermatosis With Abnormal Epidermis; Parameter: The incidence of vulvar irritation depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of vulvar irritation depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvar dermatosis?; p = 0.8599, Chi-squared
Statistical Analysis 7: Comparison: Vulvar Dermatosis With Normal Epidermis vs Vulvar Dermatosis With Abnormal Epidermis; Parameter: The incidence of vulvar itching depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of vulvar itching depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvar dermatosis?; p = 0.9402, Chi-squared
Statistical Analysis 8: Comparison: Vulvar Dermatosis With Normal Epidermis vs Vulvar Dermatosis With Abnormal Epidermis; Parameter: The incidence of the feeling of vulvar inflammation depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of the feeling of vulvar inflammation depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvar dermatosis?; p = 0.8389, Chi-squared
Statistical Analysis 9: Comparison: Vulvar Dermatosis With Normal Epidermis vs Vulvar Dermatosis With Abnormal Epidermis; Parameter: The incidence of vulvar aching depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of vulvar aching depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvar dermatosis?; p = 0.7617, Chi-squared
Statistical Analysis 10: Comparison: Vulvar Dermatosis With Normal Epidermis vs Vulvar Dermatosis With Abnormal Epidermis; Parameter: The difference in the incidence of the sharp (fast) pain of the vulva (knife-like pain, paper-cuts pain, stabbing, sticking) depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of the sharp pain of the vulva depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvar dermatosis?; p = 0.4613, Chi-squared
Statistical Analysis 11: Comparison: Vulvar Dermatosis With Normal Epidermis vs Vulvar Dermatosis With Abnormal Epidermis; Parameter: The incidence of the vulvar knife-like pain depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of vulvar knife-like pain depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvar dermatosis?; p = 0.0331, Chi-squared, Corrected
Statistical Analysis 12: Comparison: Vulvar Dermatosis With Normal Epidermis vs Vulvar Dermatosis With Abnormal Epidermis; Parameter: The incidence of the vulvar paper-cuts pain depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of vulvar paper-cuts pain depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvar dermatosis?; p = 0.9402, Chi-squared
Statistical Analysis 13: Comparison: Vulvar Dermatosis With Normal Epidermis vs Vulvar Dermatosis With Abnormal Epidermis; Parameter: The incidence of vulvar pain like stabbing depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of vulvar pain like stabbing depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvar dermatosis?; p = 0.9139, Chi-squared
Statistical Analysis 14: Comparison: Vulvar Dermatosis With Normal Epidermis vs Vulvar Dermatosis With Abnormal Epidermis; Parameter: The incidence of the vulvar pain like sticking depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvar dermatosis; Test type: Superiority — Question: Is there a difference in the incidence of vulvar pain like sticking depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvar dermatosis?; p = 0.8925, Chi-squared

37. Secondary Outcome: Histopathological Features of the Vulvar Epidermis and Vulvar Complaints in Patients With Vulvodynia
Description: The table shows the relationship between histopathological features of the vulvar epidermis (normal versus abnormal), and single vulvar symptoms from the categories of the dull ("slow") and sharp ("fast") pain of the vulva in 82 patients with vulvodynia diagnosed anamnestically and clinically following Friedrich's criteria.
  The "dull" pain comprises sensations of burning, stinging, soreness, irritation, itching, inflammation and aching. The "fast" pain includes sensations like sticking and stabbing, paper-cut or knife-like pain.
Time Frame: Histopathological Examination, up to 30 minutes for each vulvar sample.
Population: We performed a biopsy of the vulva in 82 symptomatic patients with vulvodynia diagnosed anamnestically and by clinical examination following Friedrich's criteria during the routine clinical care, to exclude other skin diseases on histopathology.
Measure: Count of Participants; unit: Participants
Groups:
- Vulvodynia With Normal Epidermis: Histopathological Finding of Normal Epidermis among the various vulvar complaints in patients with vulvodynia.
- Vulvodynia With Abnormal Epidermis: Histopathological Finding of Abnormal Epidermis among the various vulvar complaints in patients with vulvodynia.
Arm/Group | Vulvodynia With Normal Epidermis | Vulvodynia With Abnormal Epidermis
Number analyzed (Participants) | 71 | 11
Participants
  Dull / Slow Pain | 70 | 11
  Burning | 30 | 7
  Stinging | 57 | 9
  Soreness | 48 | 6
  Irritation | 39 | 9
  Itching | 54 | 9
  Inflammation | 41 | 8
  Aching | 38 | 7
  Sharp / Fast Pain | 22 | 9
  Knife-Like Pain | 7 | 6
  Paper-Cuts Pain | 6 | 4
  Stabbing | 12 | 5
  Sticking | 15 | 3
Statistical Analysis 1: Comparison: Vulvodynia With Normal Epidermis vs Vulvodynia With Abnormal Epidermis; Parameter: The difference in the incidence of vulvar complaints depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of vulvar complaints depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvodynia?; p = 0.0000, Chi-squared
Statistical Analysis 2: Comparison: Vulvodynia With Normal Epidermis vs Vulvodynia With Abnormal Epidermis; Parameter: The difference in the incidence of symptoms of the dull (slow) pain depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of symptoms of the dull pain depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvodynia?; p = 0.6921, Chi-squared
Statistical Analysis 3: Comparison: Vulvodynia With Normal Epidermis vs Vulvodynia With Abnormal Epidermis; Parameter: The incidence of vulvar burning depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of vulvar burning on the histopathology of the epidermis (normal versus abnormal) in patients with vulvodynia?; p = 0.1848, Chi-squared
Statistical Analysis 4: Comparison: Vulvodynia With Normal Epidermis vs Vulvodynia With Abnormal Epidermis; Parameter: The incidence of vulvar stinging depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of vulvar stinging depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvodynia?; p = 0.9048, Chi-squared
Statistical Analysis 5: Comparison: Vulvodynia With Normal Epidermis vs Vulvodynia With Abnormal Epidermis; Parameter: The incidence of vulvar soreness depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of vulvar soreness depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvodynia?; p = 0.3953, Chi-squared
Statistical Analysis 6: Comparison: Vulvodynia With Normal Epidermis vs Vulvodynia With Abnormal Epidermis; Parameter: The incidence of vulvar irritation depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of vulvar irritation depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvodynia?; p = 0.0921, Chi-squared
Statistical Analysis 7: Comparison: Vulvodynia With Normal Epidermis vs Vulvodynia With Abnormal Epidermis; Parameter: The incidence of vulvar itching depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of vulvar itching depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvodynia?; p = 0.6734, Chi-squared
Statistical Analysis 8: Comparison: Vulvodynia With Normal Epidermis vs Vulvodynia With Abnormal Epidermis; Parameter: The incidence of the feeling of vulvar inflammation depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of the feeling of vulvar inflammation depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvodynia?; p = 0.3458, Chi-squared
Statistical Analysis 9: Comparison: Vulvodynia With Normal Epidermis vs Vulvodynia With Abnormal Epidermis; Parameter: The incidence of vulvar aching depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of vulvar aching depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvodynia?; p = 0.5304, Chi-squared
Statistical Analysis 10: Comparison: Vulvodynia With Normal Epidermis vs Vulvodynia With Abnormal Epidermis; Parameter: The difference in the incidence of symptoms of the sharp (fast) pain depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of symptoms of the sharp pain depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvodynia?; p = 0.0012, Chi-squared
Statistical Analysis 11: Comparison: Vulvodynia With Normal Epidermis vs Vulvodynia With Abnormal Epidermis; Parameter: The incidence of vulvar knife-like pain depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of vulvar knife-like pain depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvodynia?; p = 0.0002, Chi-squared
Statistical Analysis 12: Comparison: Vulvodynia With Normal Epidermis vs Vulvodynia With Abnormal Epidermis; Parameter: The incidence of vulvar paper-cuts pain depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of vulvar paper-cuts pain depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvodynia?; p = 0.0218, Chi-squared, Corrected
Statistical Analysis 13: Comparison: Vulvodynia With Normal Epidermis vs Vulvodynia With Abnormal Epidermis; Parameter: The incidence of vulvar pain like stabbing depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of vulvar pain like stabbing depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvodynia?; p = 0.0297, Chi-squared
Statistical Analysis 14: Comparison: Vulvodynia With Normal Epidermis vs Vulvodynia With Abnormal Epidermis; Parameter: The incidence of vulvar pain like sticking depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvodynia; Test type: Superiority — Question: Is there a difference in the incidence of vulvar pain like sticking depending on the histopathology of the epidermis (normal versus abnormal) in patients with vulvodynia?; p = 0.6468, Chi-squared

38. Secondary Outcome: Histopathological Features of Vulvar Dermis in Patients With Vulvar Dermatosis Depending On The Duration of Vulvar Discomfort
Description: The table shows the relationship between histopathological features of the vulvar dermis depending on the duration of vulvar discomfort (less or more than 24 months) in 82 consecutive patients with vulvar dermatosis.
  Histopathological characteristics of vulvar dermis included inflammatory infiltrates (mononuclear, lymphocytes, mastocytes), collagen fibers, hyalinization, hyperpigmentation, elongated dermal papillae, blood vessels, sebaceous glands, and nerve fibers.
Time Frame: Histopathological Examination, up to 30 minutes for each vulvar sample.
Population: as for outcome 36
Measure: Count of Participants; unit: Participants
Groups:
- Vulvar Dermatosis 1: Patients with duration of symptoms of the vulvar dermatosis less than 24 months.
- Vulvar Dermatosis 2: Patients with duration of symptoms of the vulvar dermatosis more than 24 months.
Arm/Group | Vulvar Dermatosis 1 | Vulvar Dermatosis 2
Number analyzed (Participants) | 24 | 58
Participants
  Inflammatory Infiltrates | 23 | 50
  Mononuclear Inflammatory Infiltrates | 19 | 44
  Lymphocytes | 5 | 8
  Mastocytes | 0 | 0
  Collagen Fibers | 11 | 33
  Hyalinization | 7 | 18
  Hyperpigmentation | 0 | 0
  Elongated Dermal Papillae | 0 | 1
  Blood Vessels | 1 | 4
  Sebaceous Glands | 0 | 1
  Nerve Fibers | 0 | 0
Statistical Analysis 1: Comparison: Vulvar Dermatosis 1 vs Vulvar Dermatosis 2; Parameter: The difference in the incidence of the histopathological finding of inflammatory infiltrates in vulvar specimens from patients with vulvar dermatosis depending on the duration of vulvar discomfort; Test type: Superiority — Question: Is there a difference in the incidence of the finding of inflammatory infiltrates in vulvar specimens from patients with vulvar dermatosis depending on the duration of vulvar discomfort for less or more than 24 months?; p = 0.2045, Chi-squared
Statistical Analysis 2: Comparison: Vulvar Dermatosis 1 vs Vulvar Dermatosis 2; Parameter: The difference in the incidence of the histopathological finding of mononuclear inflammatory infiltrates in vulvar specimens from patients with vulvar dermatosis depending on the duration of vulvar discomfort; Test type: Superiority — Question: Is there a difference in the incidence of the finding of mononuclear inflammatory infiltrates in vulvar specimens from patients with vulvar dermatosis depending on the duration of vulvar discomfort for less or more than 24 months?; p = 0.7469, Chi-squared
Statistical Analysis 3: Comparison: Vulvar Dermatosis 1 vs Vulvar Dermatosis 2; Parameter: The difference in the incidence of the histopathological finding of lymphocytes in vulvar specimens from patients with vulvar dermatosis depending on the duration of vulvar discomfort; Test type: Superiority — Question: Is there a difference in the incidence of the finding of lymphocytes in vulvar specimens from patients with vulvar dermatosis depending on the duration of vulvar discomfort for less or more than 24 months?; p = 0.4271, Chi-squared
Statistical Analysis 4: Comparison: Vulvar Dermatosis 1 vs Vulvar Dermatosis 2; Parameter: The difference in the incidence of the histopathological finding of collagen fibers in vulvar specimens from patients with vulvar dermatosis depending on the duration of vulvar discomfort; Test type: Superiority — Question: Is there a difference in the incidence of the finding of collagen fibers in vulvar specimens from patients with vulvar dermatosis depending on the duration of vulvar discomfort for less or more than 24 months?; p = 0.3607, Chi-squared
Statistical Analysis 5: Comparison: Vulvar Dermatosis 1 vs Vulvar Dermatosis 2; Parameter: The difference in the incidence of the histopathological finding of hyalinization in vulvar specimens from patients with vulvar dermatosis depending on the duration of vulvar discomfort; Test type: Superiority — Question: Is there a difference in the incidence of the finding of hyalinization in vulvar specimens from patients with vulvar dermatosis depending on the duration of vulvar discomfort for less or more than 24 months?; p = 0.8672, Chi-squared

39. Secondary Outcome: Histopathological Features of the Vulvar Dermis in Patients With Vulvodynia Depending on The Duration of Vulvar Discomfort
Description: The table shows the relationship between histopathological features of the vulvar dermis depending on the duration of vulvar discomfort (less or more than 24 months) in 82 patients with vulvodynia, diagnosed anamnestically and clinically following Friedrich's criteria.
  Histopathological characteristics of vulvar dermis included inflammatory infiltrates (mononuclear, lymphocytes, mastocytes), collagen fibers, hyalinization, hyperpigmentation, elongated dermal papillae, blood vessels, sebaceous glands, and nerve fibers.
Time Frame: Histopathological Examination, up to 30 minutes for each vulvar sample.
Population: We performed a biopsy of the vulva in 82 symptomatic patients with vulvodynia diagnosed anamnestically and by clinical examination following Friedrich's criteria during the routine clinical care, to exclude other skin diseases.
Measure: Count of Participants; unit: Participants
Groups:
- Vulvodynia 1: Patients with duration of symptoms of the vulvodynia less than 24 months.
- Vulvodynia 2: Patients with duration of symptoms of vulvodynia more than 24 months.
Arm/Group | Vulvodynia 1 | Vulvodynia 2
Number analyzed (Participants) | 29 | 53
Participants
  Inflammatory Infiltrates | 18 | 47
  Mononuclear Inflammatory Infiltrates | 16 | 45
  Lymphocytes | 1 | 2
  Mastocytes | 4 | 2
  Collagen Fibers | 1 | 8
  Hyalinization | 0 | 0
  Hyperpigmentation | 1 | 4
  Elongated Dermal Papillae | 0 | 0
  Blood Vessels | 14 | 39
  Sebaceous Glands | 22 | 39
  Nerve Fibers | 21 | 47
Statistical Analysis 1: Comparison: Vulvodynia 1 vs Vulvodynia 2; Parameter: The difference in the incidence of the histopathological finding of inflammatory infiltrates in vulvar specimens from patients with vulvodynia depending on the duration of vulvar discomfort; Test type: Superiority — Question: Is there a difference in the incidence of the finding of inflammatory infiltrates in vulvar specimens from patients with vulvodynia depending on the duration of vulvar discomfort for less or more than 24 months?; p = 0.0045, Chi-squared
Statistical Analysis 2: Comparison: Vulvodynia 1 vs Vulvodynia 2; Parameter: The difference in the incidence of the histopathological finding of mononuclear inflammatory infiltrates in vulvar specimens from patients with vulvodynia depending on the duration of vulvar discomfort; Test type: Superiority — Question: Is there a difference in the incidence of the finding of mononuclear inflammatory infiltrates in vulvar specimens from patients with vulvodynia depending on the duration of vulvar discomfort for less or more than 24 months?; p = 0.0032, Chi-squared
Statistical Analysis 3: Comparison: Vulvodynia 1 vs Vulvodynia 2; Parameter: The difference in the incidence of the histopathological finding of collagen fibers in vulvar specimens from patients with vulvodynia depending on the duration of vulvar discomfort; Test type: Superiority — Question: Is there a difference in the incidence of the finding of collagen fibers in vulvar specimens from patients with vulvodynia depending on the duration of vulvar discomfort for less or more than 24 months?; p = 0.1067, Chi-squared
Statistical Analysis 4: Comparison: Vulvodynia 1 vs Vulvodynia 2; Parameter: The difference in the incidence of the histopathological finding of hyalinization in vulvar specimens from patients with vulvodynia depending on the duration of vulvar discomfort; Test type: Superiority — Question: Is there a difference in the incidence of inflammatory cells in vulvar specimens from patients with vulvodynia depending on the duration of vulvar discomfort for less or more than 24 months?; p = 0.8672, Chi-squared
Statistical Analysis 5: Comparison: Vulvodynia 1 vs Vulvodynia 2; Parameter: The difference in the incidence of the histopathological finding of blood vessels in vulvar specimens from patients with vulvodynia depending on the duration of vulvar discomfort; Test type: Superiority — Question: Is there a difference in the incidence of blood vessels in vulvar specimens from patients with vulvodynia depending on the duration of vulvar discomfort for less or more than 24 months?; p = 0.0219, Chi-squared
Statistical Analysis 6: Comparison: Vulvodynia 1 vs Vulvodynia 2; Parameter: The difference in the incidence of the histopathological finding of sebaceous glands in vulvar specimens from patients with vulvodynia depending on the duration of vulvar discomfort; Test type: Superiority — Question: Is there a difference in the incidence of sebaceous glands in vulvar specimens from patients with vulvodynia depending on the duration of vulvar discomfort for less or more than 24 months?; p = 0.8213, Chi-squared
Statistical Analysis 7: Comparison: Vulvodynia 1 vs Vulvodynia 2; Parameter: The difference in the incidence of the histopathological finding of nerve fibers in vulvar specimens from patients with vulvodynia depending on the duration of vulvar discomfort; Test type: Superiority — Question: Is there a difference in the incidence of the finding of nerve fibers in vulvar specimens from patients with vulvodynia depending on the duration of vulvar discomfort for less or more than 24 months?; p = 0.0613, Chi-squared

ADVERSE EVENTS:
Time Frame: We collected the adverse event data from hospital admission up to 2 years after TRIV for each participant.
Description: Agency for Medicinal Products And Medical Devices of Croatia (HALMED), Ministry of Health of Republic Croatia
Groups:
- Normal Vulva: Patients without vulvar discomfort and any vulvar lesion undergoing planned labioplasty, before surgery.
- Impaired Vulvar Skin: Patients without vulvar symptoms with some non-specific lesions of the vulva found by clinical examination, undergoing planned labioplasty, before surgery.
- Vulvodynia: Patients with vulvar discomfort, who clinically fulfilled Friedrich's criteria. Non-specific lesions found with TRIV were not relevant to the diagnosis of vulvodynia.
- Vulvar Dermatosis: Patients with vulvar discomfort and vulvar lesions specific for dermatosis found by clinical examination.
Arm/Group | Normal Vulva | Impaired Vulvar Skin | Vulvodynia | Vulvar Dermatosis
All-Cause Mortality (participants affected / at risk) | 0/82 | 0/82 | 0/82 | 0/82
Serious Adverse Events (participants affected / at risk) | 0/82 | 0/82 | 0/82 | 0/82
Other Adverse Events (participants affected / at risk) | 0/82 | 0/82 | 0/82 | 0/82

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No